

#### **Clinical Trial Protocol**

| | <b>Document Number:</b> | c03357704-04 |
|---|---|---|
| EudraCT No.: | 2014-005102-38 | |
| BI Trial No.: | 1311.4 | |
| BI Investigational Product: | BI 655066/ ABBV-066 (risankizum | ab) |
| Title: | BI 655066 / ABBV-066 (risankizum<br>Multicenter randomized double-blin<br>Moderate to severe chronic plaque p<br>efficacy and safety with randomized<br>(IMMhance) | d study in patients with osoriasis evaluating the |
| Brief Title: | BI 655066 / ABBV-066 (risankizum chronic plaque psoriasis with randor treatment. | |
| Clinical Phase: | III | |
| Trial Clinical<br>Monitor: | Boehringer Ingelheim Pharmaceutic<br>900 Ridgebury Road<br>Ridgefield CT USA 06877 | als |
| Coordinating<br>Investigator: | | |
| Status: | Revised Protocol (based on Global A | Amendment #3) |
| Version and Date: | 4.0 | Date: 11-Oct-2016 |
| | Proprietary confidential information | |

Proprietary confidential information.

© 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

**Trial Protocol** 


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **CLINICAL TRIAL PROTOCOL SYNOPSIS**

| Name of company:<br>Boehringer Ingelheim | | | |
|---|---|---|---|
| Name of finished product | t: | | |
| Not Applicable | | | |
| Name of active ingredien | t: | | |
| BI 655066/ ABBV-06 | 6 (risankizumab) | | |
| Protocol date: | Trial number: | | Revision date: |
| 22-Oct-2015 | 1311.4 | | 11-Oct-2016 |
| Title of trial: | Multicenter random Moderate to severe | V-066 (risankizumab) versus pmized double-blind study in pecHronic plAque psoriasis evy with randomized withdrawa | atients with aluatiNg the |
| Coordinating<br>Investigator: | | | |
| Trial site(s): | Multicentre Trial o | conducted in approximately 10 | ) countries |
| Clinical phase: | III | | |
| Objective(s): | efficacy of BI 655<br>with moderate to s<br>efficacy evaluation | tives of this trial are to assess 066 150 mg in comparison to severe chronic plaque psoriasis at 16 weeks. Following drug sponse as well as the response cluated. | placebo in patients<br>s with the primary<br>g withdrawal, the |
| | | iasis patients with concomitant<br>ptoms of psoriatic arthritis will<br>nt during the trial. | |
| Methodology: | double-blind, place<br>at a ratio of 4:1 to<br>Randomisation wi | tory, multinational, multicente<br>ebo controlled study. Patients<br>either BI 655066 150 mg or to<br>Il be stratified with to respect<br>r exposure to TNF antagonists | will be randomized o placebo. weight (≤ 100 kg vs. |

| Name of company:<br>Boehringer Ingelheim | | | |
|---|---|---|---|
| Name of finished produc | t: | | |
| Name of active ingredien<br>BI 655066/ ABBV-06 | | | |
| Protocol date: | Trial number: | | Revision date: |
| 22-Oct-2015 | 1311.4 | | 11-Oct-2016 |
| No. of patients: | (Randomisation), tweeks thereafter wateratment, patients Patients will be off (OLE) trial, if they | the second dose at Week 4, and with the last dose at Week 88. will continue in the 16 week fered to roll over into an open of have completed the study and E trial at the End of Observation. | d then every 12 After the end of follow up period. label extension d meet the inclusion |
| total entered: | Approximately 50 | 0 patients | |
| each treatment: | 400 BI 655066, 10 | 00 placebo | |
| Diagnosis: | Moderate to severe | ere chronic plaque psoriasis | |
| Main criteria for inclusion: | <ul> <li>Have a diagnor psoriatic arthri administration</li> <li>Have stable money without psoriation</li> <li>Have at a stable money and the stable money and the stable money are a stable money and the stable money and the stable money are a stable money are a stable money and the stable money are a stable money and the stable money are a stable money and the stable money are a stable money and the stable money are a stable money and the stable money are a stable money are a stable money and the stable money are a stable money and the stable money are a stable money and the stable money are a stable money and the stable money are a stable money are a stable money and the stab</li></ul> | oderate to severe chronic plaq<br>tic arthritis at both Screening a | with or without re the first ue psoriasis with or and Baseline (BSA) ≥ 10% and and (PASI) score ≥ ssment (sPGA) score |

| Name of company:<br>Boehringer Ingelheim | | | |
|---|---|---|---|
| Name of finished produc | t: | | |
| Name of active ingredien<br>BI 655066/ ABBV-06 | | | |
| Protocol date: | Trial number: | | Revision date: |
| 22-Oct-2015 | 1311.4 | | 11-Oct-2016 |
| Test product(s): | BI 655066 | | <u> </u> |
| dose: | | s, 75mg each) at week 0, 4 an | d every 12 weeks |
| mode of administration: | s.c. | | |
| Comparator products: | Placebo | | |
| dose: | Not applicable | | |
| mode of administration: | s.c. | | |
| Duration of treatment: | 88 weeks | | |
| Endpoints | (PASI 90) Achievement 1) at Week Key Secondary En Achievement (PASI 75) at Achievement (PASI 100) Achievement Achievement score of 0 at Achievement 1) at Week Other Secondary En | ent of ≥ 90% reduction from b<br>at Week 16<br>ent of an sPGA score of clear ent<br>adpoints:<br>ent of 75% reduction from bas<br>at Week 16<br>ent of 100% reduction from bas<br>at Week 16<br>ent of an sPGA score of clear<br>ent of a Dermatology Life Qual<br>or 1 at Week 16<br>ent of an sPGA score of clear<br>ent of an sPGA score of clear | or almost clear (0 or seline PASI score aseline PASI score (0) at Week 16 ality Index (DLQI) |

| | | I | |
|---|---|---|---|
| Name of company: | | | |
| Boehringer Ingelheim | | | |
| Name of finished prod | luct: | | |
| Name of active ingred<br>BI 655066/ ABBV- | ient:<br>·066 (risankizumab) | | |
| Protocol date: | Trial number: | | Revision date: |
| 22-Oct-2015 | 1311.4 | | 11-Oct-2016 |
| | Note that all key a | ent of PASI 100 at Week 52<br>nd other secondary endpoints<br>tients re-randomised at Week | |
| Safety criteria: | Physical examinations, vital signs, 12 lead electrocardiogram (ECG), laboratory testing, adverse events, local tolerability | | |
| Statistical methods: | Co-primary analysticlear or almost cle are binary variable proportion responding will be estimated a difference estimate (≤ 100 kg versus ≥1) with we secondary analysis | sis: The achievement of PASI ar at Week 16 are the co-primes with values of 0 or 1. The ding between the BI 655066 and tested using the Cochran-lestratified by the randomisation 100 kg) and prior exposure to eights proposed by Greenland stream the stratified by the randomisation of the proposed by Greenland and the stratified by Greenland strategies are the same methods for the proposed strategies are the same methods for the same methods for the same methods for the same methods for the sam | 90 and sPGA of ary endpoints and ifference in arm and placebo arm Mantel-Haenszel risk on factors of weight TNF antagonists (0 & Robins. |
| | All hypotheses wil tests with a type I | Il be tested in a hierarchical or error of 0.05. | der using two-sided |

11-Oct- 2016

Bochringer Ingelheim BI Trial No.: 1311.0004 c03357704-04


## FLOW CHART 1

| Trial Period | Screening | | | | | | | | | T | Treatment | 'nt | | | | | | | | | Fol | Follow-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | 1 | 2 | က | 4 | w | 9 | 7 | ∞ | 6 | 01 | 11 | | 13 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21<br>EOT | Follow-u<br>#1 <sup>12</sup> | Follow-up #2<br>(EOO) |
| Week | | | 4 | <b>%</b> | 12 | 16 | 20 | 24 | 28 | 32 3 | 36 4 | 40 4 | 44 48 | 52 | 28 | 64 | 70 | 92 | 82 | 88 | 94<br>EOT+<br>6wks | 104<br>EOT+<br>16wks |
| Day | -42 to -7 | 1 | 28 | 99 | 84 | 112 | 140 | | | | | | | | Ĥ | Ĥ | Ť | H | H | | | 728 |
| Visit window (days) | N/A | | #3 | ±7 | ±7 | ±3 | ±7 | ±7 | ±7 = | ∓7 ∓ | ±7 = | ±7 ± | ±7 ±7 | 1 ±7 | ±2 | ±7 | ±2 | ±2 | ±7 | ±2 | ±7 | ±7 |
| Informed consent | X | | | | | | | | | $\vdash$ | H | H | H | H | Ц | Ц | | | Ц | | | |
| Demographics | X | | | | | | | | | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | | | | | | | | |
| Smoking, alcohol history | X | | | | | | | | | | | H | | | Ц | | | | Ц | | | |
| Psoriatic arthritis Medical<br>History <sup>19</sup> | X | | | | | | | | | | | | | | | | | | | | | |
| Inclusion-/exclusion<br>criteria | X | X | | | | | | | | | | | | | | | | | | | | |
| % BSA involvement | X | X | | | | | | | | | | | | | | | | | | | | |
| Psoriasis therapy history | X | | | | | | | | | | | | | | | | | | | | | |
| Height | X | | | | | | | | | | | | | | | Щ | | | | | | |
| Weight, waist circumference <sup>9</sup> | × | | | | | | | | × | | | | | × | | | | × | | | | × |
| CASPAR for PsA <sup>8</sup> | X | | | | | | | | | | | | | | | | | | | | | |
| Vitals | X | $X^{13}$ | $X^{13}$ | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Physical examination <sup>4</sup> | Xc | Xt | Xt | Xt | Xt | Xt | Xt | Хc | | Χt | Xt | -1 | Xt Xt | | Xt | _ | Xt | Xc | Χţ | | Xt | Xc |
| 12 lead-ECG | X | × | X | | | X | | | X | 1 | - 1 | X | | X | | X | | X | | × | | X |
| Safety laboratory testing <sup>14</sup> | × | × | × | | | × | | | × | | ′ 1 | X | | X | | X | | × | | × | | X |
| Adverse events | X | × | X | X | × | X | X | × | | × | × | | X | X | | X | X | X | × | × | X | X |
| Concomitant therapy | X | X | X | X | × | X | X | × | × | × | × | X | X | | × | × | × | × | × | × | X | X |
| Infection Testing 23 | X | | | | | | | | | | | _ | | X | | _ | | | _ | | | X |
| Pregnancy testing | Xs | Χn | χn | | | χn | 1 | | Χn | + | ~ | χn | | Χn | 4 | Χn | | Χn | _ | Χn | | Xu |
| Optional DNA Banking" | | × | | | | | | 1 | 1 | $\dashv$ | 1 | $\dashv$ | | - | | 4 | | | | _ | | |
| Randomisation via IRT | 3 | × | ; | | 1 | ; | 1 | $\dagger$ | | $\dashv$ | - | + | $\dashv$ | | + | + | - | 4 | 7 | 4 | | , |
| Contact IRT | X | X | X | | 1 | X | | | + | X X | X | 1 | Х Х | + | X | 4 | X | 4 | X | 4 | | X |
| Administer trial drug <sup>24</sup> | | × | × | | | × | | | _ | 1 | 1 | | | + | | × | | × | _ | × | | |
| Local tolerability assessment | | | × | × | × | × | × | × | × | <u>~</u><br>× | <u>~</u><br>× | <u>~ </u> | ×<br>× | × | × | × | × | × | × | × | | |
| Blood sampling for PK | | <b>X</b> <sup>7</sup> | <b>X</b> <sup>7</sup> | | × | <b>X</b> <sup>7</sup> | | | <b>X</b> ' | × | ^ | <b>X</b> <sup>7</sup> | | X, | × | X, | × | <b>X</b> | | <b>X</b> | | × |
| ADA assessment sampling | | $\mathbf{X}^{\prime}$ | $\mathbf{X}'$ | | | $\mathbf{X}^{7}$ | | | $\mathbf{X}^{\prime}$ | | Υ | $X^7$ | | X, | | $\mathbf{X}^{\prime}$ | | $\mathbf{X}^{\prime}$ | | $\mathbf{X}^{\prime}$ | | X |
| Biomarker sampling <sup>10</sup> , | | X | X | | | X | | | X | | . 1 | X | | X | | X | | X | | X | | X |
| PASI, sPGA | X | X | X | X | X | X | X | X | Н | X . | X | X | X | X | X | X | X | X | X | X | X | X |
| NAPSI, PSSI, PPASI | | X | | | | X | | | X | | | | _ | _ | | _ | | | | | | |
| DLQI 3 | | X | | | X | X | | | | | | | | | | | | | | | | |
| HAQ-DI, Pain VAS/ PtGA | | X | | | | X | | | X | | | | | X | | | | X | | | | × |
| V ZOS | | | 1 | 1 | | | 1 | 1 | $\left\{ \right.$ | -[ | - | $\frac{1}{2}$ | $\left\{ \right.$ | _ | - | - | - | | - | - | | |

**Boehringer Ingelheim** 

BI Trial No.: 1311.0004

c03357704-04

Trial Protocol


11-Oct- 2016

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Visit 1 2 3 Week 4 4 Day -42 to -7 1 28 Visit window (days) N/A ±3 | | | | | | | Trea | Treatment | | | | | | | | | Fol | Follow-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| k<br>-42 to -7 1 28<br>window (days) N/A ±3 | 4 | 2 | 2 9 | 8 | 6 | 10 | 111 | 12 | 13 | 14 | 15 | 91 | 17 | 18 1 | 19 20 | 0<br>EOT | Follow-up<br>I #1 <sup>12</sup> | Follow-up #2<br>(EOO) |
| -42 to -7 1 28 xindow (days) N/A ±3 | 8 | 12 1 | 16 20 | 0 24 | . 28 | 32 | 36 | 40 | 44 | 48 | 52 | 58 | 64 | 70 7 | 76 82 | 88 2 | 94<br>EOT+<br>6wks | 104<br>EOT+<br>16wks |
| N/A ±3 | 99 | 84 1 | 112 140 | 168 | 961 8 | 224 | 252 | 280 | 308 | 336 | 364 | 700 | 448 4 | 490 53 | 532 574 | 4 616 | 959 | 728 |
| | 7= | ±7 ± | ±3 ±7 | ZŦ | £1 | 47 | 7± | 1-7 | £1 | 1-7 | +7 | ±7 | F LŦ | ±7 ± | T± 7± | 7 ±7 | ±7 | ±7 |
| TJC/SJC, DAS28 <sup>16</sup> X | | 200 | X | | X | 2 3 | | | | | X | _ | _ | | X | | | X |
| sPGA assessment of relapse <sup>22</sup> | a : | | | ca s | | $X^{17}$ | $X^{IJ}$ | $_{L}X$ | XIX | X <sub>1</sub> , | X <sub>1</sub> , | XIX | $\mathbf{x}_{u}$ | X <sub>u</sub> X | 8IX 8IX | 18 X <sup>21</sup> | | St |
| Termination of trial drug <sup>15</sup> | | | | | | | | | | | | | _ | | | X | | |
| Trial completion | | - | | × | _ | | | 8-8 | | | 8 8 | | _ | S (0 | | _ | 8 | X |
| Open label extension | | Н | H | Н | Ц | | | | | П | П | H | Н | H | Н | Н | | $X_{\varrho}$ |
| Vital Status <sup>20</sup> | 0 0 | _ | 5 C | 0 | _ | o_ o | | 2-2 | 5 S | | 0 2 | | J. J | o o | - | <u>.</u> . | | X |

## Flow Chart 1 Footnotes

- Pregnancy Testing: Xs =serum testing; Xu= onsite urine testing; Serum pregnancy is done at screening and as a reflex when urine testing is
  - Voluntary DNA banking sample will be stored after informed consent is given. This may be a separate informed consent or part of the main informed consent in accordance with local ethical and regulatory requirements. Refer to Section 5.5 2
- PRO= Patient Reported Outcomes are performed electronically at clinic visits and completed by patients in a quiet place prior to any other visit procedure. The order will be as follows (see also <u>Appendix 10.6</u> and <u>Appendix 10.7</u>): 3
- HAQ-DI [for psoriatic arthritis patients at selected sites]
- Pain VAS [for psoriatic arthritis patients at selected sites] 0
- Patient Global Assessment (PtGA) VAS [for psoriatic arthritis patients at selected sites]
  - Physical exams: T = targeted, C = complete. Refer to Section 5.3.1 for details.
- Randomisation via IRT at Visit 2. Re-randomisation via IRT at Week 28 for Responders (sPGA =0 or 1). See Section 6.2.2
- who have not discontinued drug prematurely and who also meet the eligibility criteria will be offered to roll over into an open label extension Patients who have completed the study (which is defined as patients completing the EOO visit within the specified window per the flow charts.) (OLE) trial. Refer to Clinical Trial Protocol (CTP) Section 6.2.3 for additional information on the OLE trial. 6. 5
  - Blood samples for PK and Anti-drug antibodies (ADA) should be taken within 60 minutes before the subcutaneous injection (pre-dose).
- At Visit 1 at selected study sites, patients with a positive history of PsA or suspected to have PsA will be further evaluated for PsA diagnosis based on CASPAR (CIASsification of Psoriatic Arthritis) criteria (R15-1001) See Appendix 10.6 . ×
- For detailed instruction how to measure waist circumference see Section 5.3.1.1 of the protocol

11-Oct- 2016


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Trial Protocol

- Biomarker sampling should be done prior to administration of study drug at dosing visits. See Section 5.5 and lab manual for procedure
- For those patients continuing in the double-blind portion of the trial an additional IRT call will be needed when patients in the randomized withdrawal part of trial reach sPGA≥3 at a non-dosing visit starting at Week 32. See also footnote # 17 and #18. 1
- Follow-up Visit #1 is not required for patients discontinuing treatment early. After completing the EOT visit, these patients go right to EOO visit end of treatment + 16 weeks). See Section 6 12
- Vital signs will be assessed prior to treatment as well as approximately 5 and 60 minutes post dose (after last injection) at the first 2 dosing visits 13.
- Blood samples should be taken after patient has fasted for at least 8 hours prior (except screening visit). If not fasted mark on laboratory requisition 4.
- Visits. Termination of trial medication eCRF should be completed and end of study registered as a non-completer in IRT. Refer to Section 6.2.3 Patients that terminate trial medication early should remain in the trial and complete all remaining Treatment Period visits and, FU1 and FU2 or details and further instruction if patient cannot or will not continue in the trial. 15.
- Fender and swollen joint counts (TJC/SJC) and Disease Activity Score (DAS28) will be done at selected sites for confirmed psoriatic arthritis oatients (See Appendix 10.6) 16.
- The patient will be switched to Flow Chart 2 if relapse occurs between Week 32 through Week 70 (inclusive). The R1 visit from the Flowchart 2 must be conducted instead of the current scheduled or unscheduled visit. See also Flow Chart 2 and Sections 3.1 and 6.2.2. 17.
  - The patient will be switched to Flow Chart 3 if they relapse after week 70 through to week 82 (inclusive). The R1 visit from Flowchart 3 must be conducted instead of the current scheduled or unscheduled visit. See also Flow Chart 3 and Sections 3.1 and 6.2.2. ∞
    - History for psoriatic arthritis is done on all patients at all sites
    - For patients who discontinue early, vital status should be collected every 12 months after discontinuation up to the original planned EOO. 19. 20.
- Patients relapsing after Week 82 through Week 88 will immediately follow EOT procedures per Flow Chart 1 (see also Section 3.1 and 6.2.2) 21.
- For patients re-randomized at Week 28 continuing in the double blind treatment portion of the study, assessment of relapse is defined as having an  $sPGA \ge 3$ . If the sPGA is  $\ge 3$ , the result is entered into IRT and IRT will immediately dispense open label BI 655066.
  - Infection Testing: Note that at the Screening Visit (or prior to randomization) only TB testing is required. See Section 5.3.3:1 for a complete list of 23.
- Patients should be closely monitored for signs and symptoms of hypersensitivity reactions for approximately 2 hours after the last injection at Visit 2 and for approximately one hour after the last injection at all other visits where drug is administered. Hypersensitivity reactions should be treated according to medical standards. 2.

11-Oct- 2016

BI Trial No.: 1311.0004 c03357704-04 **Boehringer Ingelheim** 


**Trial Protocol** 

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# FOR RELAPSED AND RE-TREATED PATIENTS FROM WEEK 32 THROUGH WEEK 70 FLOW CHART 2

| | | | Re-Treatment | | | Follo | Follow-up |
|---|---|---|---|---|---|---|---|
| Relapse Visit | R1 | R2 | R3 | R4 | R5<br>(EOT) | Follow-up #1 | Follow-up #2<br>EOO |
| Weeks of Re-Treatment | | 4 | œ | 12 | 16 | EOT+<br>6wks | EOT+<br>16wks |
| Day of Re-Treatment | 1 | 28 | 99 | 84 | 112 | 154 | 224 |
| Visit window (days) | | ∓3 | <b>L</b> ∓ | ±7 | ±7 | 7= | ±7 |
| Weight, waist circumference <sup>4</sup> | × | | | | | | X |
| Vitals | × | X | X | × | × | X | X |
| Physical examination <sup>2</sup> | Xc | Xt | Xt | Xt | Xc | Xt | Xc |
| 12 lead-ECG | X | X | | | X | | X |
| Safety laboratory testing <sup>5</sup> | X | X | | | X | | X |
| Adverse events | X | X | X | X | X | X | X |
| Concomitant therapy | X | X | X | X | X | X | X |
| Infection Testing | $X^{11}$ | | | | | | X |
| Pregnancy testing <sup>1</sup> | Xu | $\mathfrak{n}_X$ | | | Xu | | Xu |
| Contact IRT | X | X | | | X | | X |
| Local tolerability | × | X | X | X | X | | |
| Blood sampling for PK | 'X | X, | | | 'X | | × |
| ADA assessment sampling | ίχ. | Χ' | | | X, | | × |
| Biomarker sampling <sup>8</sup> | × | × | | | × | | × |
| PASI, sPGA | X | X | X | X | X | X | X |
| HAQ-DI, Pain VAS/PtGA<br>VAS <sup>3</sup> | X | | | | × | | X |
| TJC/SJC, DAS289 | × | | | | × | | × |
| Administer trial drug <sup>12</sup> | X | X(load) | | | X | | |
| Termination of trial drug | | | | | X | | |
| Trial completion | | | | | | | X |
| Open label extension <sup>6</sup> | | | | | | | X |
| Vital status <sup>10</sup> | | | | | | | X |

BI Trial No.: 1311.0004 **Boehringer Ingelheim** c03357704-04

11-Oct- 2016


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Trial Protocol

## Flow Chart 2 Footnotes

- Pregnancy Testing: Xu= onsite urine testing. Serum pregnancy done as a reflex if urine test is positive.
  - Physical exams: T = targeted, C = complete. Refer to Section 5.3.1 for details
- PRO= Patient Reported Outcomes are performed electronically at clinic visits and completed by patients in a quiet place prior to any other visit procedure. The order will be as follows ( see also Appendix 10.6 and Appendix 10.7):
  - a) HAQ-DI [for psoriatic arthritis patients at selected sites]
- Pain VAS [for psoriatic arthritis patients at selected sites] þ)
- c) Patient Global Assessment (PtGA) VAS [for psoriatic arthritis patients at selected sites]
- For detailed instruction how to measure waist circumference see Section 5.3.1.1 of the protocol
- Blood samples should be taken after patient has fasted for at least 8 hours prior (except screening visit). If not fasted mark on laboratory requisition.
- Patients who have completed the study (which is defined as patients completing the EOO visit within the specified window per the flow charts, who have not discontinued drug prematurely and who also meet the eligibility criteria) will be offered to roll over into an open label extension (OLE) trial. Refer to CTP Section 6.2.3 for additional information on the OLE trial.
  - Blood samples for PK and Anti-drug antibodies (ADA) should be taken within 60 minutes before the subcutaneous injection (pre-dose) **.**. ∞ •
- Biomarker sampling should be done prior to administration of study drug at dosing visits. See Section 5.5 and lab manual for procedure
- Tender and swollen joint counts (TJC/SJC) and Disease Activity Score (DAS28) will be done at selected sites for confirmed psoriatic arthritis patients (See Appendix 10.6)
- For relapsed and retreated patients following Flow Chart #2 and who discontinue early, Vital Status should be collected after discontinuation up to the new planned EOO per Flow Chart #2.
- 11. Infection Testing at R1 visit only for patients relapsing on or before Visit 15 (Week 52)
- 12. Patients should be closely monitored for signs and symptoms of hypersensitivity reactions for approximately 2 hours after the last injection at Visit 2 and for approximately 1 hour after the last injection at all other visits where drug is administered. Hypersensitivity reactions should be treated according to medical standards.

Boehringer Ingelheim

BI Trial No.: 1311.0004 c03357704-04

Trial Protocol


11-Oct- 2016

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

FLOW CHART 3 FOR RELAPSE AND RE-TREATED PATIENTS AFTER WEEK 70 THROUGH WEEK 82

| | Re-tre | Re-treatment | Foll | Follow-up |
|---|---|---|---|---|
| Relapse Visit | R1 | R2<br>(EOT) | Follow-up #1 | Follow-up #2<br>EOO |
| Weeks of Re-Treatment | | 4 | EOT+ | EOT+ |
| Day of Re-Treatment | 1 | 28 | OWKS | LOWKS |
| Visit window (days) | l | #3 | 7= | 7= |
| Weight, waist circumference <sup>4</sup> | × | | | × |
| Vitals | X | X | × | × |
| Physical examination <sup>2</sup> | Хс | Xc | Xt | Xc |
| 12 lead-ECG | × | × | | × |
| Safety laboratory testing <sup>5</sup> | X | × | | × |
| Adverse events | × | × | X | × |
| Concomitant therapy | × | × | X | × |
| Infection Testing | | | | X |
| Pregnancy testing <sup>1</sup> | nX | nX | | Xu |
| Contact IRT | X | X | | X |
| Local tolerability | X | X | | |
| assessment | | | | |
| Blood sampling for PK | $\mathbf{X}_{'}$ | $\mathbf{X}^7$ | | X |
| ADA assessment sampling | $\mathbf{X}_{2}$ | $\mathbf{X}^7$ | | X |
| Biomarker sampling <sup>8</sup> | X | X | | X |
| PASI, sPGA | X | X | X | X |
| HAQ-DI, Pain VAS/ PtGA<br>VAS <sup>3</sup> | X | X | | X |
| TJC/SJC, DAS289 | × | × | | X |
| Administer trial drug <sup>11</sup> | X | X(load) | | |
| Termination of trial drug | | X | | |
| Trial completion | | | | X |
| Open label extension <sup>6</sup> | | | | X |
| Vital status <sup>10</sup> | | | | X |

Note: Patients relapsing after Week 82 will immediately follow EOT procedures, and then return for Follow-up #1 and Follow-up #2. A loading dose will not be administered.

BI Trial No.: 1311.0004 **Boehringer Ingelheim** c03357704-04

11-Oct- 2016


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Trial Protocol

# Flow Chart 3 Footnotes

- Pregnancy Testing: Xu= onsite urine testing. Serum pregnancy done as a reflex if urine test is positive.
  - Physical exams: T = targeted, C = complete. Refer to Section 5.3.1 for details
- PRO= Patient Reported Outcomes are performed electronically at clinic visits and completed by patients in a quiet place prior to any other visit procedure. The order will be as follows (see also <u>Appendix 10.6</u> and <u>Appendix 10.7</u>):
  - a) HAQ-DI [for psoriatic arthritis patients at selected sites] b) Pain VAS [for psoriatic arthritis patients at selected sites]
- Pain VAS [for psoriatic arthritis patients at selected sites]
- Patient Global Assessment (PtGA) VAS [for psoriatic arthritis patients at selected sites]
- For detailed instruction how to measure waist circumference see Section 5.3.1.1 of the protocol
- Patients who have completed the study (which is defined as patients completing the EOO visit within the specified window per the flow charts) who Blood samples should be taken after patient has fasted for at least 8 hours prior (except screening visit). If not fasted mark on laboratory requisition. have not discontinued drug prematurely and who also meet the eligibility criteria will be offered to roll over into an open label extension (OLE)
- Blood samples for PK and Anti-drug antibodies (ADA) should be taken within 60 minutes before the subcutaneous injection (pre-dose)

trial. Refer to CTP Section 6.2.3 for additional information on the OLE trial.

- Biomarker sampling should be done prior to administration of study drug at dosing visits. See Section 5.5 and lab manual for procedure ۲. % و.
- Tender and swollen joint counts (TJC/SJC) and Disease Activity Score (DAS28) will be done at selected sites for confirmed psoriatic arthritis patients (See Appendix 10.6)
- For relapsed and re-treated patients following Flow Chart #3 who discontinue early, Vital Status should be collected after discontinuation up to the new planned EOO per Flow Chart #3.
- Patients should be closely monitored for signs and symptoms of hypersensitivity reactions for approximately 2 hours after the last injection at Visit 2 and for approximately 1 hour after the last injection at all other visits where drug is administered. Hypersensitivity reactions should be treated according to medical standards. 11:

#### **TABLE OF CONTENTS**

| TITLE P | PAGE | 1 |
|---|---|---|
| CLINIC | AL TRIAL PROTOCOL SYNOPSIS | 2 |
| FLOW ( | CHART 1 | 6 |
| FLOW ( | CHART 2 FOR RELAPSED AND RE-TREATED PATIENTS FROM 32 THROUGH WEEK 70 | |
| FLOW ( | CHART 3 FOR RELAPSE AND RE-TREATED PATIENTS AFTER V THROUGH WEEK 82 | |
| TABLE | OF CONTENTS | 13 |
| ABBREV | VIATIONS | 17 |
| 1. | INTRODUCTION | 20 |
| 1.1<br>1.2 | MEDICAL BACKGROUNDDRUG PROFILE | |
| 2. | RATIONALE, OBJECTIVES, AND BENEFIT - RISK ASSESSMEN | JT 22 |
| 2.1<br>2.2<br>2.3 | RATIONALE FOR PERFORMING THE TRIAL TRIAL OBJECTIVES BENEFIT - RISK ASSESSMENT | 22 |
| 3. | DESCRIPTION OF DESIGN AND TRIAL POPULATION | |
| 3.1<br>3.1.1<br>3.1.2<br>3.1.3<br>3.2 | OVERALL TRIAL DESIGN AND PLAN Administrative structure of the trial Data Monitoring Committee (DMC) MACE Adjudication Committee DISCUSSION OF TRIAL DESIGN, INCLUDING THE CHOICE OF | 25<br>26<br>27 |
| 3.3<br>3.3.1<br>3.3.2<br>3.3.3.<br>3.3.4<br>3.3.4.1<br>3.3.4.2 | CONTROL GROUP(S) SELECTION OF TRIAL POPULATION Main diagnosis for trial entry Inclusion criteria Exclusion criteria Removal of patients from therapy or assessments Removal of individual patients Discontinuation of the trial by the sponsor | 27<br>28<br>28<br>29 |
| <b>4.</b> | TREATMENTS | |
| 4.1<br>4.1.1<br>4.1.2 | TREATMENTS TO BE ADMINISTERED Identity of BI investigational product and reference product Method of assigning patients to treatment groups | 32<br>32<br>33 |
| <b>4.1.3 4.1.4 4.1.5 4.1.5.1</b> | Selection of doses in the trial Drug assignment and administration of doses for each patient Blinding and procedures for unblinding Blinding | 34<br>36 |
| 4.1.5.2<br><b>4.1.6</b><br><b>4.1.7</b> | Unblinding and breaking the code Packaging, labelling, and re-supply Storage conditions | 37 |

Trial Protocol 

| Proprieta <b>4.1.8</b> | ry confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies |
|---|---|
| | Drug accountability |
| 4.2 | |
| 421 | TREATMENT |
| 4.2.1 | Rescue medication, emergency procedures, and additional treatment(s) 38 |
| 4.2.2 | Restrictions |
| 4.2.2.1 | Restrictions regarding concomitant treatment |
| 4.2.2.2 | Restrictions on diet and life style |
| 4.2.2.3 | Restrictions regarding women of childbearing potential |
| 4.3 | TREATMENT COMPLIANCE |
| 5. | VARIABLES AND THEIR ASSESSMENT41 |
| 5.1 | TRIAL ENDPOINTS41 |
| 5.1.1 | Primary Endpoint(s)41 |
| 5.1.2 | Secondary Endpoints41 |
| 5.1.3. | Further Endpoints41 |
| 5.2 | ASSESSMENT OF EFFICACY42 |
| 5.3 | ASSESSMENT OF SAFETY42 |
| 5.3.1 | Physical examination43 |
| 5.3.2 | Vital Signs |
| 5.3.3 | Safety laboratory parameters |
| 5.3.4 | Electrocardiogram |
| 5.3.5 | Other safety parameters |
| 5.3.5.1 | Local Tolerability 47 |
| 5.3.6 | Assessment of adverse events 47 |
| 5.3.6.1 | Definitions of AEs |
| 5.3.7 | Adverse event collection and reporting |
| 5.4 | DRUG CONCENTRATION MEASUREMENTS AND |
| | PHARMACOKINETICS |
| 5.4.1 | Assessment of Pharmacokinetics |
| 5.4.2 | Methods of sample collection |
| 5.4.2.1 | Plasma sampling for pharmacokinetic analysis |
| 5.4.2.2 | Plasma sampling for ADA |
| 5.4.3 | Analytical determinations |
| 5.4.4 | Pharmacokinetic-Pharmacodynamic Relationship |
| 5.5 | ASSESSMENT OF EXPLORATORY BIOMARKERS |
| 5.5.1 | Assessment of soluble protein biomarkers in blood |
| 5.5.1.1 | |
| 5.5.1.1 | Methods of sample collection |
| 5.5.1.2<br>5.5.2 | |
| 5.5.2.1. | DNA Banking |
| | * |
| 5.5.2.2. | Analytical determinations 53 |
| 5.5.3 | Biomarker sample banking |
| 5.6 | OTHER ASSESSMENTS |
| 5.7 | APPROPRIATENESS OF MEASUREMENTS53 |
| 6.0 | INVESTIGATIONAL PLAN |
| 6.1 | VISIT SCHEDULE54 |
| 6.2 | DETAILS OF TRIAL PROCEDURES AT SELECTED VISITS54 |
| 6.2.1 | Screening period |
| 6.2.2 | Treatment period55 |

Trial Protocol 

| Propriet <b>6.2.3</b> | ary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies Follow up Period and Trial Completion |
|---|---|
| 7.0 | STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE58 |
| 7.1 | STATISTICAL DESIGN - MODEL58 |
| 7.2 | NULL AND ALTERNATIVE HYPOTHESES |
| 7.3 | PLANNED ANALYSES 59 |
| 7.3.1 | Primary endpoint analyses |
| 7.3.1 | Secondary endpoint analyses |
| 7.3.3 | Further endpoint analyses 61 |
| 7.3.4 | Safety analyses |
| 7.3.5 | Pharmacokinetic analyses 62 |
| 7.3.6 | Pharmacodynamic analysis |
| 7.3.7 | Biomarker analyses |
| 7.3.7 | INTERIM ANALYSES 63 |
| 7.4<br>7.5 | HANDLING OF MISSING DATA |
| 7.6 | RANDOMISATION |
| 7.0<br>7.7 | DETERMINATION OF SAMPLE SIZE 64 |
| 8.0 | INFORMED CONSENT, DATA PROTECTION, TRIAL RECORDS66 |
| 8.1 | TRIAL APPROVAL, PATIENT INFORMATION, AND INFORMED CONSENT |
| 8.2 | DATA QUALITY ASSURANCE |
| 8.3 | RECORDS 67 |
| 8.3.1 | Source documents 67 |
| 8.3.2 | Direct access to source data and documents |
| 8.3.3 | Storage period of records (Applicable to Japan only) |
| 8.4 | LISTEDNESS AND EXPEDITED REPORTING OF ADVERSE EVENTS68 |
| 8.4.1 | Listedness AND EATEDITED REFORTING OF ADVERSE EVENTS08 Listedness 68 |
| 8.4.2 | Expedited reporting to health authorities and IEC / IRB |
| 8.5 | STATEMENT OF CONFIDENTIALITY |
| 8.6 | END OF TRIAL 68 |
| 8.7 | PROTOCOL VIOLATIONS 68 |
| 8.8 | COMPENSATION AVAILABLE TO THE PATIENT IN THE EVENT OF |
| 0.0 | TRIAL RELATED INJURY |
| 9.0 | REFERENCES |
| 9.1 | PUBLISHED REFERENCES |
| 9.2 | UNPUBLISHED REFERENCES |
| 10 | APPENDICES73 |
| 10.1 | PASI DEFINITIONS AND USE73 |
| 10.1 | STATIC PHYSICIAN GLOBAL ASSESSMENT (SPGA) |
| 10.2 | NAPSI – NAIL PSORIASIS SEVERITY INDEX |
| 10.3 | PPASI – PALMOPLANTAR PSORIASIS SEVERITY INDEX77 |
| 10.4 | PSORIASIS SCALP SEVERITY INDEX (PSSI) |
| 10.5 | DIAGNOSIS AND ASSESSMENTS FOR PATIENTS WITH PSORIATIC |
| 10.0 | ARTHRITIS (AT SELECTED SITES ONLY)79 |
| 10.6.1 | Disease Activity Score in 28 Joints (DAS 28) |
| 10.0.1 | HEALTH OUTCOMES/QUALITY OF LIFE |
| 10.7 | Dermatology Life Quality Index |
| 10.7.1 | Health Assessment Ouestionnaire Disability Index (HAO-DI) |
| 13/0/04 | - 115/0110 (550550111011 570551101111011 C 1715/011111 V 111110 X 1117(7-1711 |

| Boehringer Ingelheim | | | 11 Oct 2016 |
|---|---|---|---|
| BI Trial N | No.: 1311.0004 | | |
| c03357704 | 4-04 | Trial Protocol | |
| Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies | | | |
| 10.7.3 | Pain VAS | ••••• | 86 |
| 10.7.4 | Patient global assess | sment VAS | 86 |
| 11. | DESCRIPTION OF | GLOBAL AMENDMENTS | S87 |

Boehringer Ingelheim 11 Oct 2016

BI Trial No.: 1311.0004

c03357704-04 Trial Protocol 

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **ABBREVIATIONS**

ADA Anti-drug antibodies AE Adverse Event

AESI Adverse events of special interest

ALT Alanine transferase AP Alkaline Phosphatase

aPTT Activated Partial Thromboplastin Time

AST Aspartate transferase
AUC Area under the Curve
BI Boehringer Ingelheim
BSA Body Surface Area
BUN Blood Urea Nitrogen
CA Competent Authority

CASPAR Classification criteria for Psoriatic Arthritis

CK Creatine Kinase

CK-MB Creatine Kinase Muscle Brain

Cmax maximal Concentration
CML Local Clinical Monitor
CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

CRP C-Reactive Protein
CTP Clinical Trial Protocol
CTR Clinical Trial Report
DAS Disease Activity Score

DEDP Drug Exposure During Pregnancy

DILI Drug induced liver injury

DLQI Dermatology Life Quality Index
DMC Data Monitoring Committee
DNA Deoxyribonucleic acid
ECG Electrocardiogram

eCOA Electronic Clinical Outcomes Assessment

eCRF Electronic Case Report Form
eGFR Estimated glomerular filtration rate
ELISA Enzyme Linked Immunosorbent Assay

EOO End of Observation EOT End of Treatment

EudraCT European Clinical Trials Database

FAS Full Analysis Set FC Flow Chart

GCP Good Clinical Practice

GGT Gamma-Glutamyl Transferase

GRAPPA The Group for Research and Assessment of Psoriasis and Psoriatic

Arthritis

HAQ-DI Health Assessment Questionnaire Disability Index

Hb Hemoglobin Hct Hematocrit

HDL High density lipoprotein

HIV Human immunodeficiency virus

lheim 11 Oct 2016

c03357704-04 Trial Protocol 

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

HIPAA Health insurance portability and accountability act HOMA-IR Homeostatis model assessment of insulin resistance

IB Investigator's Brochure IC Inhibitory Concentration

ICH International conference on harmonisation

IEC Independent Ethics Committee

IgG Immunoglobulin G

INR International normalized ratio

IL Interleukin

IQR Interquartile Range

IRB Institutional Review Board IRT Interactive Response Technology

ISF Investigator Site File

i.v. Intravenous

LDL Low density lipoprotein

LOCF Last observation carried forward

mAb Monoclonal Antibody

MACE Major adverse cardiovascular events

MedDRA Medical Dictionary for Drug Regulatory Activities

MMRM Mixed effect Model Repeat Measurement

Nab Neutralizing Antibody NAPSI Nail Psoriasis Severity Index

NGAL Neutrophil gelatinase associated lipocalin-2

NOAEL No Observed Adverse Effect Level

NRI No Response Imputation OLE Open label extension

OPU Operative unit

PASI Psoriasis Area and Severity Index

PD Pharmacodynamics PK Pharmacokinetics

PoCC Proof of Clinical Concept

PPASI Palmoplantar Psoriasis Severity Index

PPD Purified Protein Derivative

PPS Per Protocol Set

PRO Patient Reported Outcomes

PsA Psoriatic Arthritis

PSI Psoriasis Symptom Inventory PSSI Psoriasis Scalp Severity Index PtGA Patient Global Assessment

RBC Red Blood Cells

RCTC Rheumatology Common Toxicity Criteria

RDC Remote Data Capture

REP Residual effect period, after the last dose of medication with measureable

drug levels or pharmacodynamic effects still likely to be present

RRS-PPS Re-Randomized Per Protocol Set

SAE Serious Adverse Event

SAF Safety Set

SD Standard deviation

SOP Standard Operating Procedures

s.c. subcutaneous

Boehringer Ingelheim BI Trial No.: 1311.0004 11 Oct 2016

c03357704-04 Trial Protocol 

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

sPGA Static Physician Global Assessment

SUSAR Suspected Unexpected Serious Adverse Reaction

TB Tuberculosis

TJC/SJC Tender or swollen joint count

TMF Trial Master File

TNF Tumor Necrosis Factor

TSAP Trial Statistical Analysis Plan
TSH Thyroid Stimulating Hormone

ULN Upper limit of normal VAS Visual Analog Scale

VEGF Vascular endothelial growth factor

WBC White Blood cells

**Trial Protocol** 


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 1. INTRODUCTION

#### 1.1 MEDICAL BACKGROUND

Psoriasis is a chronic inflammatory disease with well-demarcated erythematous plaques with adherent silvery scales (R11-1257). It is the most prevalent immune-mediated skin disease, affecting 2% of the world population (R08-1089). Twenty-five percent of patients have moderate to severe disease with considerable negative impact on psychosocial and economic status (R11-1259). It is increasingly recognized that psoriasis is more than a superficial disease, with 30% of patients having joint involvement and a high correlation between psoriasis and obesity, diabetes, depression, metabolic syndrome, and cardiovascular risk (R15-1393).

While many psoriasis patients with mild disease are managed with topical therapies, those with severe and/or refractory disease may require phototherapy and/or systemic therapy. Oral systemic agents provide modest efficacy, but increasingly patients are treated with more effective biologic agents, such as TNF-alpha inhibitors (etanercept, adalimumab) and the p40 IL-12/23 inhibitor (ustekinumab) (R14-5159). While the clinical efficacy of ustekinumab indicates a role for both IL-12 and IL-23 in the pathogenesis of psoriasis (R11-1547), more recent data suggest that IL-23 is disproportionately involved in the maintenance of chronic psoriasis (R11-1547). IL-23 is thought to act in the pathophysiology of psoriasis via induction and maintenance of Th17 cells as well as other IL-23 responsive cells. This is supported by recent clinical data indicating that monoclonal antibodies that block IL-17A, the cytokine produced by the Th17 cells, have high efficacy in psoriasis.

There is still clinical need for increased efficacy as the most effective anti-TNF and IL12/23 agents provide only 75% improvement in psoriasis in about 60-70% of patients, and these responses tend to be lost over time. While the anti-IL-17A agents provide better efficacy, they require monthly injections; thus, their long-term utility is still undetermined. BI 655066 is a humanized monoclonal antibody with high affinity for the p19 component of human IL-23 that specifically neutralizes IL-23. Proof of clinical concept (PoCC) for BI 655066 was demonstrated in a single dose phase I trial in 39 patients with moderate to severe plaque psoriasis, where 87% of patients achieved at least 75% reduction in Psoriasis Area and Severity Index (PASI 75) with no safety concerns (c02434648-01).

A 48-week Phase II dose ranging trial of BI 655066 vs. ustekinumab indicates a 37% greater improvement for BI 655066 (90 mg and 180 mg, pooled data) when compared to ustekinumab in the proportion of patients achieving 90% reduction in PASI (PASI 90) at Week 12. We propose the current trial to establish the safety and efficacy of BI 655066 in larger numbers of patients over a longer duration of treatment.

#### 1.2 DRUG PROFILE

BI 655066 is a fully humanized monoclonal antibody (mAb) of the IgG1 subclass directed towards IL-23p19. The antibody has been engineered to reduce Fc $\gamma$  receptor and complement binding and potential charge heterogeneity. BI 655066 binds with high affinity to human IL-23 and inhibits IL-23 stimulated IL-17 production at IC 50 concentrations below 10 pM, as compared with 167 pM for ustekinumab in the same system. BI 655066 does not affect IL-12 at a maximum tested concentration (33 nM) and it does not inhibit IL-12 stimulated IFN- $\gamma$  production.

Boehringer Ingelheim BI Trial No.: 1311.0004 c03357704-04

11 Oct 2016

57704-04 Trial Protocol 

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The toxicology data suggest BI 655066 can be safely administered to humans, as supported by chronic administration to monkeys for up to 26 weeks. The monkey was identified as the most relevant toxicology species with a NOAEL of 50 mg/kg/dose, corresponding to an exposure (combined sex) of 677  $\mu$ g/mL for the Cmax and 86,250  $\mu$ g\*h/mL for AUC0-168, respectively.

BI 655066 has been studied in approximately 200 patients with psoriasis without any unexpected adverse events or safety issue. Based on the efficacy and safety findings in the completed and ongoing studies, the risk benefit profile of BI 655066 is appropriate for initiation of Phase III studies. In Study 1311.1 (c02434648-01), a Phase I single rising dose trial in 39 patients with chronic plaque psoriasis, administration of BI 655066 either intravenously (i.v.) or subcutaneously (s.c.) was well tolerated. Over the 24 weeks following a single i.v. or s.c. administration of BI 655066, 65% (20/31) of patients experienced an AE compared with 88% (7/8) of patients receiving placebo. The most frequently reported AEs were mild to moderate upper respiratory tract infections, mild nasopharyngitis and mild to moderate headache. The severity of AEs did not appear related to the dose of BI 655066. Injection site reactions were reported in 2/18) patients receiving BI 655066 i.v., in 1/6 patients receiving placebo i.v. and in none of the patients receiving BI 655066 or placebo s.c.

In patients receiving BI 655066 either i.v. (n=18) or s.c. (n=13), 87% achieved at least 75% reduction in Psoriasis Severity and Area Index (PASI 75) by Week 12, compared to none in the placebo group. Twenty four weeks after a single administration of BI 655066, 71% of patients maintained at least a PASI 75; nearly half (48%) had 90% reduction in PASI (PASI 90) and 29% had complete resolution of lesions (PASI 100). A protocol amendment allowed an optional extension of follow-up beyond Week 24 for patients in the s.c. dose cohort; six of thirteen originally enrolled patients maintained a PASI 100 improvement for 41–66 weeks after treatment.

After a single i.v. administration, BI 655066 geometric mean  $AUC_{0-inf}$  ranged from 2.93–1650 day\* $\mu$ g/mL and  $C_{max}$  from 0.311–110  $\mu$ g/mL, with exposure increasing in a dose-proportional manner. Group mean clearance and terminal phase volume of distribution were 0.33 L/day and 10.8 L, respectively PK parameter variability, expressed as gCV (%) was <50%. After a single s.c. administration of BI 655066, maximal exposures were reached between 5-13 days and subcutaneous bioavailability was 73% (expressed as the ratio of geometric mean dose normalised  $AUC_{0-inf}$  after s.c. and i.v. administration).

For a more detailed description of the drug profile refer to the current Investigator's Brochure (IB) (c01569420-06) which is included in the Investigator Site File (ISF).

c03357704-04


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 2. RATIONALE, OBJECTIVES, AND BENEFIT - RISK ASSESSMENT

#### 2.1 RATIONALE FOR PERFORMING THE TRIAL

Psoriasis is a chronic inflammatory disease affecting 2% of the world population with significant impact on patient quality of life with significant systemic disease (R08-1089). IL-23 plays a key role in the pathophysiology of psoriasis through induction and maintenance of Th17 type cells that secrete inflammatory cytokines. BI 655066 is a humanized monoclonal antibody that specifically neutralizes the IL-23 axis. Proof of clinical concept (PoCC) for BI 655066 was demonstrated in a single dose phase I trial in 39 patients with moderate to severe plaque psoriasis where 87% of patients achieved at least 75% reduction in Psoriasis Area and Severity Index (PASI 75) with no safety concerns (c02434648-01).

This trial is being performed to assess the safety and efficacy of BI 655066 to support a registration for the treatment of moderate to severe plaque psoriasis in adult patients.

#### 2.2 TRIAL OBJECTIVES

The primary objectives of this trial are to assess the safety and efficacy of BI 655066 150 mg in comparison to placebo in patients with moderate to severe chronic plaque psoriasis. The primary efficacy evaluation will be performed at 16 weeks. In addition, the maintenance of response following drug withdrawal will be assessed after Week 28 through Week 104. Subsequent to drug withdrawal, patients who experience relapse will be retreated with BI 655066 to assess response after retreatment.

In addition, this trial will assess PK and the emergence of anti-drug antibodies (ADA) and their effect on efficacy and safety. Moreover, it will be explored how the use of BI 655066 may influence gene and protein expression levels and disease specific protein markers.

In a subset of psoriasis patients with concomitant psoriatic arthritis, the signs and symptoms of psoriatic arthritis will be evaluated to assess improvement during the trial.

Lastly, the influence of study treatment on some metabolic risk factors will be evaluated.

#### 2.3 BENEFIT - RISK ASSESSMENT

Participation in this study may help to generate future benefit for larger groups of patients with psoriasis if BI 655066 proves to be successful in treating this disease. BI 655066 has been studied in approximately 200 patients with moderate to severe plaque psoriasis. In these studies, the majority of patients receiving BI 655066 achieved 90% improvement of their disease. The most common adverse events reported in these trials were mild symptoms of the upper respiratory tract, including nasal stuffiness, sore throat, influenza, and headache. These events were not considered to be related to drug treatment. Local reactions following subcutaneous administration of BI 655066 were uncommon, and limited to mild redness, swelling or induration at the injection site. No serious drug related adverse events were reported.

As with many immune modulating agents, BI 655066 may impair immune function resulting in a risk of infection. This will be monitored by collection of all AEs during the treatment and

#### **Trial Protocol**


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

observation periods. Patients with clinically important active infection will not be included in the study.

IL-23 inhibition is not known to increase the risk of TB infection or impair the response to TB infection in animal models (R15-5488; R15-5495). Thus, low risk patients with positive Quantiferon testing do not need to be treated with anti-tuberculosis therapy prior to receiving BI-655066, but should be carefully monitored for any sign of TB reactivation. Absence of TB reactivation, despite not receiving anti-tuberculosis prophylaxis will provide important information in humans as to whether TB testing is required prior to treatment with BI 655066 (R15-5497).

There is not enough information at this time to rule out a risk of cancer with BI 655066, but this risk is considered small with this type of compound because long-term experience with the anti-IL-12/23 mAb ustekinumab has not been associated with significant cancer risk. Patients will be monitored for signs and symptoms of malignancy at each visit.

Increases in major adverse cardiovascular events (MACE) including myocardial infarction, cerebrovascular accident, and cardiovascular death, reported initially with anti-IL-12/23 agents, such as ustekinumab, have not been observed in longer term studies. While the likelihood of increased MACE is small, all cardiovascular events (serious or non-serious) observed in this study will be adjudicated by an independent MACE Adjudication Committee.

A patient will have a 20% (1 in 5) chance in being randomized to the placebo arm. Patients assigned to placebo will have a low rate of response. These patients will be crossed over to active BI 655066 treatment at Week 16 of study participation. The knowledge gained from the placebo treatment group in a relatively short period of time can be used to control for bias and effect size. The delay in starting treatment does not diminish the potential benefit of treatment or introduce any risk. Patients will be monitored with study visits every 4 weeks through the end of the placebo period at Week 16.

Although rare, a potential for drug-induced liver injury is under constant surveillance by sponsors and regulators. Therefore, this trial requires timely detection, evaluation, and follow-up of laboratory alterations in selected liver laboratory parameters to ensure patients' safety, see Section 5.3.6.1.

In conclusion, the benefit-risk profile is considered appropriate for this stage of clinical development. In order to recognize any safety signals as early as possible, an independent DMC will monitor all studies where patients are receiving BI 655066.

c03357704-04


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 3. DESCRIPTION OF DESIGN AND TRIAL POPULATION

#### 3.1 OVERALL TRIAL DESIGN AND PLAN

This is a confirmatory, multinational, multicenter, randomized, double-blind, placebo controlled, study that includes up to a 42 day screening period, an 88 week treatment period and a 16- week follow-up period. The primary objectives of this trial are to assess the safety and efficacy of BI 655066 in comparison to placebo in patients with moderate to severe chronic plaque psoriasis. The primary efficacy will be evaluated at 16 weeks. In addition, the maintenance of response following drug withdrawal in patients who respond to treatment prior to Week 28 will be assessed after Week 28 through Week 104. Subsequent to drug withdrawal, patients who experience relapse will be retreated with BI 655066 to assess response after retreatment.

In total, approximately 500 patients with moderate to severe chronic plaque psoriasis will be randomised and receive study treatment in this trial. A sufficient number of patients will be screened to meet this randomized goal. Patients are considered enrolled in the study once they have signed the informed consent.

Patients suitable after screening will be eligible to participate in this study and will be randomized at a ratio of 4:1 to one of two treatment arms as shown in <u>Figure 3.1:1</u>. Arm 1 refers to those patients originally randomized to BI 655066 and Arm 2 refers to those patients originally randomized to placebo. Randomisation will be stratified as listed in <u>Section 7.6</u>.

All patients will receive the first dose of study medication on day 1 (Randomisation), the second dose at Week 4, and then every 12 weeks thereafter with the last dose at Week 88. After the end of treatment, patients will continue in the 16- week follow- up period. At the Week 16 visit (primary endpoint), all patients randomized to Arm 2 (placebo) will start receiving 150 mg BI 655066 active treatment every 12 weeks and continue until the end of the treatment period. In order to maintain the blind, this will be performed in a blinded fashion at Week 16.

At the Week 28 visit, all patients will be assessed for responsiveness. Patients not meeting the protocol defined response criteria (sPGA is  $\geq$  2) (Week 28 non-responders), will receive open label BI 655066 150 mg from Week 28 until the end of the treatment period (Week 88), regardless of originally randomized treatment arm. Patients who meet the protocol defined responder criteria (sPGA of 0 or 1) (Week 28 responders), will continue to receive blinded drug. In Arm 1, patients will be re-randomized; in Arm 2, they will continue to receive blinded BI655066 treatment as described in Section 7.6.

Starting with Week 32, Week 28 responders will have their sPGA assessed for protocol defined relapse (sPGA of  $\geq$  3). Once a patient reaches a sPGA of  $\geq$  3, they will be switched to open label BI 655066. If this relapse occurs anytime between Week 32 through Week 70, the patients will follow Flow Chart #2 and be re-treated for 16 weeks. If this relapse occurs after Week 70 through Week 82, the patient will follow Flow Chart #3 and be re-treated for 28 days. If the relapse occurs after Week 82 through Week 88 the patient will immediately have the EOT procedures performed, including the final dose of study medication and continue into the 16-week Follow-Up Period. This process will be managed by IRT.

Patients will be offered to roll over into an open label extension (OLE) trial, if they have completed the study and meet the inclusion criteria for the OLE trial at the End of Observation (EOO) visit. See Section 6.2.2 and Section 6.2.3.

Patients who discontinue from the trial will **not** have the possibility to participate in the OLE study.

There will not be an interim analysis from a statistical standpoint however a primary endpoint analysis will be conducted after the last patient has been in the study for 52 weeks (or discontinued). See Section 7.4.

Individual patient participation is concluded when the patient has completed the last planned visit. The "last-patient-last-visit-primary-endpoint" is the last scheduled primary endpoint visit (Week 16) completed by the last patient. The end of the trial is defined as "last patient out", i.e. last scheduled visit completed by last patient.

Part A is defined as the induction and response period from initial randomisation through Week 28. Part B is defined as the withdrawal and re-treatment period from Week 28 through Week 88.



Figure 3.1:1 Trial Design

#### 3.1.1 Administrative structure of the trial

The trial is sponsored by AbbVie in the USA and Boehringer Ingelheim (BI) for all other non-USA participating countries.

Boehringer Ingelheim BI Trial No.: 1311.0004 c03357704-04

11 Oct 2016

57704-04 Trial Protocol 

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Boehringer Ingelheim has appointed a Trial Clinical Monitor, responsible for coordinating all required activities, in order to

- manage the trial in accordance with applicable regulations and internal SOPs;
- direct the clinical trial team in the preparation, conduct, and reporting of the trial;
- order the materials as needed for the trial; and
- ensure appropriate training and information of local clinical monitors (CML), Clinical Research Associates (CRAs), and Investigators of participating countries.

Data Management will be done by BI according to BI SOPs and the Statistical Evaluation will be done by AbbVie according to their SOPs.

Tasks and functions assigned in order to organise, manage, and evaluate the trial will be defined according to BI SOPs. A list of responsible persons and relevant local information can be found in the ISF.

The organisation of the trial in the participating countries will be performed by the respective local BI-organisation (Operative Unit (OPU) or by a Contract Research Organisation (CRO) which the responsibilities and tasks will have been agreed and a written contract filed before initiation of the clinical trial. In each OPU participating in this study, a CML will be appointed responsible for coordinating the activities required in order to manage the trial in accordance with applicable regulations and internal SOPs in the countries covered by the respective BI OPU.

A Coordinating Investigator will be responsible to coordinate investigators at different centres participating in this multicentre trial. Tasks and responsibilities will be defined in a contract. Relevant documentation on the participating (Principal) Investigators and other important participants, including their curricula vitae, will be filed in ISF.

Details of the trial supplies including responsible institutions are given in Section 4 of this protocol.

The ISF will be maintained at the sites as required by local regulation and BI-SOPs. A copy of the essential ISF documents will also be kept as an electronic TMF document according to BI SOPs.

A central laboratory service and vendors for ECG, eCOA and an IRT (Interactive Response Technology) will be used in this trial. Details will be provided in the applicable manuals available in the ISF.

#### 3.1.2 Data Monitoring Committee (DMC)

A data monitoring committee (DMC), independent of the Sponsor will be established to assess the progress of the clinical trial, including unblinded safety assessments at specified intervals, and to recommend to the Sponsor whether to continue, modify, or stop the trial.

Any efficacy data provided to the DMC will only be used for DMC's obligation to assess the full benefit-to-risk of the treatments. Thus, no statistical penalty will be imposed since efficacy analyses will not be the basis for any potential early trial termination.

Measures are in place to ensure blinding of the Sponsor and all other trial participants. The Sponsor will remain blinded until after the last patient completes the Week 52 visit. See Section 7.4 for more information. The tasks and responsibilities of the DMC will be specified in a charter. The DMC will maintain written records of all its meetings.


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 3.1.3 MACE Adjudication Committee

An independent adjudication committee will be used to adjudicate all observed cardio- and cerebro-vascular and thrombotic events reported during the conduct of the study to assure

consistent assessment of major adverse cardiovascular events (MACE). This review will be blinded to treatment allocation; the events that are to be adjudicated and the adjudication process will be detailed in the MACE Adjudication Committee Charter.

### 3.2 DISCUSSION OF TRIAL DESIGN, INCLUDING THE CHOICE OF CONTROL GROUP(S)

This is a randomized double blind, placebo controlled, parallel design study. This design is appropriate for assessing the safety and efficacy of BI 655066 compared to placebo in patients with moderate to severe chronic plaque psoriasis. While there is a low rate of response with placebo treatment, it is important to have a placebo control early in the study to control for confounding factors, such as potential investigator bias or regression to the mean in PASI scoring.

In order to enroll patient participants, it is necessary to allow patients initially assigned to placebo to receive active treatment. Thus, only adverse events reported during the first 16 weeks of the trial can be directly compared to placebo. In this trial, patients originally randomized to BI 655066 who are considered to be BI 655066 responders will be rerandomized to receive either placebo or continued BI 655066 starting at Week 28. Patients in this phase of the study will be assessed for an additional 76 weeks for a total of 104 weeks. This is necessary to adequately capture the loss of response for patients taking BI 655066. Furthermore, patients losing response will be retreated with BI 655066 and response after retreatment will be assessed.

#### 3.3 SELECTION OF TRIAL POPULATION

A total of approximately 500 patients is planned to be randomized in this trial. A sufficient number of patients will be screened to meet this randomized goal. Patients will be recruited at multiple investigative sites in multiple countries. Approximately 85 sites are planned with approximately 5-10 patients to be randomized per site. Recruitment will be competitive.

A log of all patients enrolled into the trial (i.e. signed informed consent) will be maintained in the ISF at the investigational sites, whether these patients have been treated with investigational drug or not.

#### 3.3.1 Main diagnosis for trial entry

Patients must have moderate to severe chronic plaque psoriasis, defined as  $\geq 10\%$  body surface area involvement, a Psoriasis Area and Severity Index  $\geq 12$  and static Physician Global Assessment score  $\geq 3$ .

Please refer to <u>Section 8.3.1</u> (Source Documents) for the documentation requirements pertaining to the inclusion and exclusion criteria.


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 3.3.2 Inclusion criteria

1. Male or female patients. Women of childbearing potential\* must be ready and able to use highly effective methods of birth control per ICH M3(R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.

\*Women of childbearing potential are defined as:

- Having experienced menarche and are
- **Not** postmenopausal (12 months with no menses without an alternative medical cause) **and are**
- **Not** permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral oophorectomy or bilateral salpingectomy).
- 2. Age  $\geq$  18 years at screening
- 3. Have a diagnosis of chronic plaque psoriasis (with or without psoriatic arthritis) at least 6 months before the first administration of study drug. Duration of diagnosis may be reported by the patient.
- 4. Have stable moderate to severe chronic plaque psoriasis with or without psoriatic arthritis at both Screening and Baseline (Randomisation);
  - Have an involved body surface area (BSA)  $\geq 10\%$  and
  - Have a Psoriasis Area and Severity Index (PASI)  $\geq$  12 and
  - Have a static Physician Global Assessment (sPGA) score of  $\geq 3$ .
- 5. Must be a candidate for systemic therapy or phototherapy for psoriasis treatment, as assessed by the investigator
- 6. Signed and dated written informed consent prior to admission to the study and performance of any study procedures in accordance with GCP and local legislation

#### 3.3.3. Exclusion criteria

- 1. Patients with
  - nonplaque forms of psoriasis (including guttate, erythrodermic, or pustular)
  - current drug-induced psoriasis (including a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium)
  - active ongoing inflammatory diseases other than psoriasis and psoriatic arthritis that might confound trial evaluations according to the investigator's judgment

Boehringer Ingelheim BI Trial No.: 1311.0004 c03357704-04

Trial Protocol


11 Oct 2016

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- 2. Previous exposure to BI 655066
- 3. Currently enrolled in another investigational study or less than 30 days (from screening) since completing another investigational study (participation in observational studies is permitted).
- 4. Use of any restricted medication as noted in <u>Table 4.2.2.1:1</u> or any drug considered likely to interfere with the safe conduct of the study.
- 5. Major surgery performed within 12 weeks prior to randomisation or planned within 12 months after screening (e.g. hip replacement, removal aneurysm, stomach ligation,).
- 6. Known chronic or relevant acute infections, such as HIV (Human Immunodeficiency Virus), \viral hepatitis, or tuberculosis. QuantiFERON® TB test or Purified Protein Derivative (PPD) skin test will be performed during screening. Patients with a positive test result may participate in the study if further work up (according to local practice/guidelines) establishes conclusively that the patient has no evidence of active tuberculosis. If presence of latent tuberculosis is established, patients who are at low risk of reactivation, defined by local guidelines and investigator judgment, do not need to be treated with prophylactic anti-tuberculosis prior to or during the trial.
- 7. Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma or squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix.
- 8. Evidence of a current or previous disease (including chronic alcohol or drug abuse), medical condition other than psoriasis, surgical procedure (i.e., organ transplant), medical examination finding (including vital signs and ECG), or laboratory value at the screening visit outside the reference range that in the opinion of the Investigator, is clinically significant and would make the study participant unable to adhere to the protocol or to complete the trial, compromise the safety of the patient, or compromise the quality of the data.
- 9. History of allergy/hypersensitivity to a systemically administered biologic agent or its excipients.
- 10. Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
- 11. Previous enrolment in this trial.

#### 3.3.4 Removal of patients from therapy or assessments

#### 3.3.4.1 Removal of individual patients

All patients have the right to withdraw from the study at any time without the need to justify their decision. The investigator has the right to remove patients from the study for non-


#### Trial Protocol

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies compliance, administrative or other reasons. It should be clearly understood that an excessive rate of withdrawals can render the study results uninterpretable. The sponsor reserves the right to remove any study patient from the trial for non-compliance.

Given the patient's agreement, the patient will undergo the procedures for early treatment discontinuation and follow up as outlined in the Flow Charts and Section 6.2.3.

An individual patient is to be withdrawn from study medication if:

- The patient withdraws consent for study treatment or study participation, without the need to justify the decision.
- The patient can no longer be treated with study medication for other medical reasons (such as surgery, adverse events, other diseases, or pregnancy).
- Development of a toxicity or adverse event that warrants BI 655066 discontinuation including but not limited to SAEs or SUSARs
- If prohibited medication is used during the study for any indication, the patient must discontinue use of the prohibited medication if he/she wants to continue in this study. In case of undue safety risk for the subject, the subject should discontinue study treatment at the discretion of the investigator. If the subject received a live virus vaccination during the study, the subject must discontinue study treatment.
- If the patient experiences an intolerable increase of psoriasis during the course of the trial the patient will be discontinued from the trial to receive rescue treatment as deemed appropriate by the investigator.

Of note: Discontinuation of study medication should not necessarily lead to withdrawal from the study. If possible the patient should complete all study visits and procedures as initially planned.

If a patient becomes pregnant during a trial, the study medication needs to be discontinued, and the patient will complete EOT Visit procedures, and Follow-up 2 (EOO) Visit procedures. The patient will be followed up until birth or otherwise termination of the pregnancy. Patients who discontinue the trial after receiving the first dose of study medication at visit 2 will not be replaced.

For all patients the reason for withdrawal (e.g. adverse events) must be recorded in the eCRF. These data will be included in the trial database and reported.

#### Vital Status

For randomized patients leaving the study early (before the planned EOO in their current applicable flow chart), vital status should be collected every 12 months after discontinuation up to the planned EOO.

#### 3.3.4.2 Discontinuation of the trial by the sponsor

AbbVie/Boehringer Ingelheim reserves the right to discontinue the trial overall or at a particular trial site at any time for the following reasons:

1. Failure to meet expected enrolment goals overall or at a particular trial site,

Boehringer Ingelheim BI Trial No.: 1311.0004 c03357704-04

11 Oct 2016

**57704-04** Trial Protocol 
Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- 2. Emergence of any efficacy/safety information that could significantly affect continuation of the trial, or any other administrative reasons, i.e. problems with availability of the study medication, discontinuation of development of BI 655066
- 3. Violation of GCP, the CTP, or a Contract disturbing the appropriate conduct of the trial. The investigator / trial site will be reimbursed for reasonable expenses incurred in case of trial termination (except in case of the third reason).

#### 4. TREATMENTS

#### 4.1 TREATMENTS TO BE ADMINISTERED

Multiple doses of BI 655066 and/or Placebo to match BI 655066 will be administered subcutaneously. All products will be supplied by Boehringer Ingelheim.

#### 4.1.1 Identity of BI investigational product and reference product

Table 4.1.1:1 BI 655066

| Substance | BI 655066: Anti-human IL-23p19 mAb |
|---|---|
| Pharmaceutical formulation: | |
| Source: | Boehringer Ingelheim Pharma GmbH & Co. KG |
| Chemical form | Anti-human IL-23p19 mAb |
| Molecular weight | Approximately 148 kDa |
| Unit strength: | 75 mg BI 655066 in a pre-filled syringe (concentration 90 mg/mL) |
| Posology | Week 0, Week 4, then every 12 weeks with last injection at Week 88 |
| Route of administration: | Subcutaneous injection |

Table 4.1.1:2 Placebo to BI 655066

| Substance: | Placebo to match BI 655066 |
|---|---|
| Pharmaceutical formulation: | |
| Source: | Boehringer Ingelheim Pharma GmbH & Co. KG |
| Chemical form | N.A |
| Molecular weight | N.A |
| Unit strength: | Sodium chloride solution in a pre-filled syringe |
| Posology | Week 0, Week 4, then every 12 weeks with last injection at Week 88 |
| Route of administration: | Subcutaneous injection |

11 Oct 2016

**Trial Protocol** 


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 4.1.2 Method of assigning patients to treatment groups

During Visit 2 and after the patient's eligibility has been confirmed, the treatment will be assigned via Interactive Response Technology (IRT). To facilitate the use of the IRT, the Investigator will receive all necessary instructions.

Patients will be randomised to receive BI 655066 150 mg or matching placebo in a ratio of 4:1. Randomisation will be stratified by weight ( $\leq 100 \text{ kg vs.} > 100 \text{ kg}$ ) and prior exposure to TNF antagonists (0 vs.  $\geq 1$ ).

At each subsequent visit where study medication is to be administered the site is required to complete the medication resupply module in the IRT. At randomisation as well as subsequent medication administration visits, IRT will assign medication numbers. Site personnel will enter the medication numbers in the eCRF.

Re-randomisation will occur at Week 28 for those patients who have met the responder criteria in Arm 1 (c.f. Section 7.6). Re-randomisation will be stratified by weight ( $\leq 100 \text{ kg vs.} > 100 \text{ kg}$ ) and prior exposure to TNF antagonists (0 vs.  $\geq 1$ ). For Week 28 responders in Arm 2, blinded BI 655066 treatment will be assigned from IRT to maintain blinding. Details regarding the use of the IRT are described in the site-user manual available in the ISF.

#### 4.1.3 Selection of doses in the trial

The dose selection strategy for phase III involved analyses of data from the completed phase I study (Trial 1311.1), (c02434648-01) the ongoing phase II study (Trial 1311.2), (c03272682-01) and PK-PD modelling of all available data from phase I and II.

The phase I and phase II data demonstrated an exposure-response relationship for BI 655066 where doses less than 0.25 mg/kg (intravenously or subcutaneously) were associated with lower clinical efficacy (assessed as decrease from baseline in the PASI score) while doses greater than 1.0 mg/kg achieved near maximal efficacy.

This exposure-response relationship was confirmed in the Phase II study where the 18 mg single injection of BI 655066 (approximately equivalent to 0.25 mg/kg in a 90 kg patient) had the lowest efficacy, while the 90 mg dose (approximately equivalent to 1 mg/kg) given at 0, 4 and 16 weeks had considerably higher efficacy (90% reduction in PASI achieved in 73.2% vs. 32.6%, p < 0.01). Thus the dose-response (range) from 0.25 to 1.0 mg/kg identified in the phase I trial was roughly replicated in the phase II trial.

Furthermore, the 180 mg dose of BI 655066 was associated with a numerically higher proportion of patients achieving PASI 90, compared to the 90 mg dose (81.0% vs. 73.2%). Although not statistically significant, this improved efficacy was noted in every endpoint (PASI 90, PASI 100 and sPGA) at each time point and was not associated with a safety issue.

#### PK-PD Modelling to Support Dose Selection

A semi-mechanistic, indirect response PK-PD model was developed using available PK and PASI data across all currently available 1311.1 and 1311.2 PASI time course data. Similar PK-PD models for efficacy have been utilized across many development programs in psoriasis.

#### **Trial Protocol**


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

A model-based assessment of exposure vs. safety response was not currently feasible, as no dose-dependent AEs have been observed currently.

The current PK-PD modelling results indicate BI 655066 pharmacokinetics are linear with respect to time and dose, and are comparable to other IgG monoclonal antibodies binding soluble targets. PASI pharmacodynamics reflect endogenous psoriatic plaque formation rate similar to the reported literature values. The half-maximal inhibition (IC<sub>50</sub>) concentration in the range of 1 ng/mL confirms the high (in vivo) potency of BI 655066.

The PK-PD modelling confirmed the conclusions of the clinical data that 180 mg provided optimal efficacy, defined at least 70% of patients achieving PASI 90. Doses above 180 mg were also modelled and these results indicated minimal improvements (<5%) in the proportion of patients achieving PASI 90. For example a dose of 300 mg was predicted to yield a PASI 90 at Week 12 of 71% (63 - 78%) compared to 68% (61 - 76%) for 180 mg. The modelling also predicted that inclusion of the additional dose at Week 4 ("loading dose") would provide higher PASI 90 response rates at earlier time points e.g. Week 12 and Week 16 compared to regimens without this additional dose.

The model was also used to examine alternative dosing regimens, both longer (i.e. every 16 weeks) or shorter (i.e. every 8-week) dosing intervals. Compared to every 12 weeks dosing, decreases in efficacy were predicted when the 16 week dosing interval was examined, while increasing the dosing frequency to every 8 weeks provided only minor improvement in efficacy, i.e. 3-5% increase in the proportion of patients achieving PASI 90. Finally, the modelling predicts that at a dose of 180 mg administered at Weeks 0, 4 and 16 the effect of body weight on PASI response rates was minimal, when this covariate was included as part of the PK model.

In addition to the observed clinical data (safety and efficacy) and PK-PD modelling, the final dose selection for Phase III was influenced by formulation and patient acceptability factors. The highest concentration of BI 655066 that can be formulated in 1 mL (and thus administered with a single injection) is 150 mg. Given that administration involving more than one injection on an ongoing basis could limit patient acceptability, modelling was used to predict PASI responses for a 150 mg dose administered at Weeks 0, 4 and every 12 weeks thereafter.

PK-PD analyses indicated no relevant reduction in efficacy when the dose was changed from 180 mg to 150 mg (based on interpolation). In summary, taking into consideration expert advisor recommendation and prescriber preferences, the proposed dosing for BI 655066 in the upcoming phase 3 trials is 150 mg at Weeks 0 and 4, followed by every 12 weeks. This regimen is anticipated to provide a favourable risk-benefit profile with a dosing schedule that is consistent with standard clinical practice.

In this trial the 150 mg dose will be administered as two prefilled syringes of 75 mg active drug each, as the 150 mg/mL formulation of BI 655066 is still being developed.

#### 4.1.4 Drug assignment and administration of doses for each patient

IRT will be used to allocate medication to patients. At randomisation as well as subsequent medication administration visits, IRT will assign medication numbers. At visits where study medication is to be administered (Refer to Flow Chart) study sites will be required to complete the appropriate module in the IRT system.

Study medication will be administered exclusively at the study site, by the investigator or authorized study personnel (e.g. study nurse).

BI 655066 and/or matching placebo will be administered as a subcutaneous injection in the abdomen, thighs, gluteal regions, or upper arms.

Injections should be at least 2 cm. apart and should not be close to a vein. The injection sites should avoid sites of psoriasis involvement as well as sites where the skin is tender, bruised, erythematous, or indurated, and should be alternated to other areas for subsequent doses.

Injections will be given in a double blind fashion with each patient receiving 2 injections of BI 655066 or matching placebo administered within approximately 5 minutes at each dosing visit as indicated in the Flow Charts.

In the eCRF, the study drug administration time is always the time of the first injection.

Further information regarding the technique of injection and injection materials (syringes, needles) will be provided in the ISF.

Patients should be closely monitored for signs and symptoms of hypersensitivity reactions for approximately 2 hours after the last injection at Visit 2 and for approximately 1 hour after the last injection at all other visits where drug is administered. Hypersensitivity reactions should be treated according to medical standards. Pre-medications for further injections might be considered and will be agreed on between investigator and BI clinical monitor.

The injections at each dosing visit are presented in Table 4.1.4: 1.

Table 4.1.4:1 Dosing schedule

| | Day 1 +<br>Week 4 | Week 16 | Week 28, 40, 52, 64, 76, 88 |
|---|---|---|---|
| Arm 1<br>BI<br>655066<br>150 mg | (2) ml (75 mg)<br>BI 655066<br>(blinded) | (2) ml (75 mg)<br>BI 655066<br>(blinded) | (2) ml (75 mg)<br>blinded or open label BI 655066<br>Or<br>(2) PTM ml (75 mg)<br>BI 655066 (blinded) |
| Arm 2 Placebo to BI 655066 150 mg | (2) PTM ml (75 mg)<br>BI 655066<br>(blinded) | (2) ml (75 mg)<br>BI 655066<br>(blinded) | (2) ml (75 mg)<br>blinded or open label BI 655066 |

PTM= Placebo to match


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 4.1.5 Blinding and procedures for unblinding

#### 4.1.5.1 Blinding

During "Part A" of this trial all patients receive double-blind treatment. Patients, investigators and everyone involved in trial conduct or analyses of this double-blind study will remain blinded with regard to the randomized treatment assignments.

Arm 1 refers to patients originally randomized to BI 655066, and Arm 2 refers to patients originally randomized to placebo at Visit 2.

At Week 28, the start of "Part B", non-responders (sPGA≥ 2) from Arm 1 and 2 will receive open label drug and will know future treatments are BI 655066.

At Week 28, responders (sPGA of 0 or 1) from Arm 1 in "Part A" will be re-randomized to either maintain treatment of BI 655066 or to receive placebo; these treatments will also be double-blinded to ensure that patients and investigators remain blinded to re-randomized treatment during "Part B." To maintain blinding, if a patient in Arm 2 reaches a sPGA of 0 or 1 at Week 28, she/he will continue to receive blinded BI 655066 treatment assigned from IRT.

After the last patient has been in the study for 52 weeks (or has discontinued), the Sponsor will be unblinded in order to summarize the trial. Blinded treatment assignments will not be disseminated to the sites, investigators, and patients until the end of study database lock.

The randomisation code will be kept secret by Clinical Trial Support up to database lock. Refer to Section 4.1.5.2 for rules of breaking the blinding code for an individual or for all patients in emergency situations.

The randomisation codes will be provided to bioanalytics prior to last patient out to allow them to exclude PK samples taken from placebo patients from the bioanalytical analyses. Bioanalytics will not disclose the randomisation code or the results of their measurements until the study is officially unblinded.

Serum drug levels and demographic data together with treatment assignments and dosing information may be made available to individuals outside of the trial team for the purpose of PK dataset generation and analysis in accordance with sponsor's standard procedures.

#### 4.1.5.2 Unblinding and breaking the code

Emergency unblinding will be available to the Investigator / Pharmacist / investigational drug storage manager via IRT. It must only be used in an emergency situation when the identity of the trial drug must be known to the Investigator in order to provide appropriate medical treatment or otherwise assure safety of trial participants. The reason for unblinding must be documented in the source documents and/or appropriate CRF page along with the date and the initials of the person who broke the code.

If the treatment code for a patient is broken, the sponsor must be informed immediately. Due to the requirements to report Suspected Unexpected Serious Adverse Reactions (SUSARs), it may be necessary for a representative from BI's drug safety group to access the randomisation code for individual patients during study conduct via the IRT system. In such cases, access to the code will only be permitted by authorised drug safety representatives.
Boehringer Ingelheim BI Trial No.: 1311.0004

11 Oct 2016

c03357704-04 Trial Protocol 

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

For Japan only:

In this blinded trial, an emergency code break will be available to the Investigator via the IRT system. This code break may only be accessed in emergency situations when the identity of the trial drug must be known to the Investigator in order to provide appropriate medical treatment or if required to assure the safety of trial participants. Each site receives a manual from the IRT provider that contains instructions on how to

unblind the treatment of a patient via the IRT (via 24-hour Emergency helpline). If the code break for a patient is accessed, the sponsor must be informed immediately. The reason for accessing the code break, together with the date, must be documented on the appropriate eCRF page. In case a third party needs to break the code when the Investigator cannot be reached, the code can be opened by calling emergency code manager.

## 4.1.6 Packaging, labelling, and re-supply

BI 655066 and placebo supplies will be provided by Boehringer Ingelheim Pharma GmbH & Co KG, Biberach, Germany (see Section 4.1.1 for more details). Pre-filled syringes of study medication will be provided in individual boxes identified with the trial number, batch and medication number. Supply of study medication will be managed by the IRT.

For details of packaging and the description of the label, refer to the ISF.

There are approximately four re-supply campaigns planned. IRT will manage the inventory and re-supply of study medication.

## 4.1.7 Storage conditions

Drug supplies will be kept in their original packaging and in a secure limited access storage area according to the recommended storage conditions on the medication label. A temperature log must be maintained for documentation.

If the storage conditions are found to be outside the specified range, the local clinical monitor (as provided in the list of contacts) must be contacted immediately.

Trial medication must be securely stored, e.g. in a locked refrigerator or at a pharmacy. The medication may only be dispensed to trial patients according to the CTP by authorized personnel as documented in the trial staff list.

#### 4.1.8 Drug accountability

Drug supplies will be provided by the sponsor.

The Investigator < and/or > pharmacist < and/or > investigational drug storage manager will receive the investigational drugs delivered by the Sponsor when the following requirements are fulfilled:

- Approval of the trial protocol by the IRB / ethics committee,
- Availability of a signed and dated clinical trial contract between the Sponsor and the head of the investigational site,
- Approval/notification of the regulatory authority, e.g. competent authority,
- Availability of the curriculum vitae of the principal Investigator,
- Availability of a signed and dated clinical trial protocol
- Availability of the proof of a medical license for the principal Investigator
- Availability of Form 1572 (only for US sites)

11 Oct 2016

**Trial Protocol** 


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

All unused medication must be returned to the sponsor. Used medication will be destroyed per local guidelines. Account must be given for any discrepancies.

Receipt, usage, and return must be documented. Account must be given for any discrepancy. These records will include dates, quantities, batch / serial numbers, expiry ('use- by') dates, and the unique code numbers assigned to the investigational product and trial patients. The Investigator / pharmacist / investigational drug storage manager will maintain records that document adequately that the patients were provided the doses specified by the CTP and reconcile all investigational products received from the Sponsor. At the time of return to the Sponsor < and/or > appointed CRO, the Investigator / pharmacist / investigational drug storage manager must verify that all unused or partially used drug supplies are not remaining in the Investigator's possession.

# 4.2 CONCOMITANT THERAPY, RESTRICTIONS, AND RESCUE TREATMENT

# 4.2.1 Rescue medication, emergency procedures, and additional treatment(s)

There are no special emergency procedures to be followed.

Stable doses of concomitant therapies for chronic conditions, for which neither the condition nor the treatment are judged to exclude the patient from participation (cf. Section 3.3), are permissible. All concomitant medications should be carefully evaluated by the investigator, and the CML should be contacted when there are questions regarding concomitant medications.

If the patient experiences an intolerable increase of psoriasis during the course of the trial as deemed by the investigator, the patient will be discontinued from the trial to receive rescue treatment.

In case of adverse events in need of treatment symptomatic therapy according to investigator judgment will be permitted. All concomitant and/or rescue therapies will be recorded on the appropriate pages of the eCRF.

## 4.2.2 Restrictions

## 4.2.2.1 Restrictions regarding concomitant treatment

The medications (or classes of medications) listed in <u>Table 4.2.2.1:1</u> must not be taken for the specified times prior to randomisation and for the whole duration of the study. If prohibited medication is used during the study for any indication, the patient must discontinue use of the prohibited medication if he/she wants to continue in this study. If a patient receives a live virus during the study, they must be discontinued.

**Trial Protocol** 


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies Table 4.2.2.1:1 Restricted medications

| Medication or class of medications | Restriction duration (through EOO Visit) |
|---|---|
| guselkumab, tildrakizumab | not allowed prior or during trial participation |
| briakinumab, secukinumab (Cosentyx®), ustekinumab (Stelara®) | 6 months prior to randomisation |
| brodalumab, ixekizumab | 4 months prior to randomisation |
| adalimumab (Humira®), infliximab (Remicade®) | 12 weeks prior to randomisation |
| investigational products for psoriasis (non biologics) | |
| etanercept (Enbrel®) | 6 weeks prior to randomisation |
| live virus vaccinations | 6 weeks prior to randomisation |
| investigational device or product (excludes psoriasis products) | |
| other systemic immunomodulating treatments (e.g. methotrexate, cyclosporine A, corticosteroids <sup>1</sup> ,cyclophosphamide, tofacitinib (Xeljanz <sup>®</sup> ), apremilast (Otezla <sup>®</sup> ) | 30 days prior to randomisation |
| other systemic psoriasis treatments (e.g. retinoids, fumarates, any other drug known to possibly benefit psoriasis) | |
| photochemotherapy (e.g., PUVA) | |
| phototherapy (e.g., UVA, UVB) | 14 days prior to randomisation |
| topical treatment for psoriasis or any other skin condition (e.g. corticosteroids <sup>2</sup> , vitamin D analogues, vitamin A analogues, pimecrolimus, retinoids, salicylvaseline, salicylic acid, lactic acid, tacrolimus, tar, urea, andanthralin, $\alpha$ -hydroxy, fruit acids) | |

<sup>&</sup>lt;sup>1</sup> No restriction on corticosteroids with only a topical effect (e.g. inhalant corticosteroids to treat asthma or corticosteroid drops used in the eye or ear).

## 4.2.2.2 Restrictions on diet and life style

Patients should be fasted for at least 8 hours prior to the collection of all safety laboratory samples starting with Visit 2.

<sup>&</sup>lt;sup>2</sup> **Exception**: Topical steroids of US class 6 (mild, such as Desonide) or US class 7 (least potent, such as hydrocortisone) will be permitted for use limited to the face, axilla, and/or genitalia with a restriction of use within 24 hours prior to clinic visits when PASI is assessed.

11 Oct 2016

**57704-04** Trial Protocol 
Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Moisturizers/emollients containing retinoids and the use of tanning beds are not allowed during the study.

## 4.2.2.3 Restrictions regarding women of childbearing potential

Female patients of childbearing potential need to follow inclusion criterion 1 in <u>Section 3.3.2</u> of this CTP and the informed consent form with regard to acceptable contraception.

## 4.3 TREATMENT COMPLIANCE

Study medication will be administered in accordance with the protocol by authorized study personnel (e.g. study nurse). The measured plasma concentrations will provide additional information about compliance.

Any missed dose has to be documented and reported to the CML.

c03357704-04

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 5. VARIABLES AND THEIR ASSESSMENT

#### 5.1 TRIAL ENDPOINTS

## 5.1.1 Primary Endpoint(s)

There are co-primary endpoints to assess the efficacy of BI 655066 for the treatment of moderate to severe plaque psoriasis. These are as follows:

- Achievement of  $\geq 90\%$  reduction from baseline PASI score (PASI 90) at Week 16
- Achievement of an sPGA score of clear or almost clear (0 or 1) at Week 16

At the trial level, the co-primary endpoints will be the proportion of patients achieving PASI 90 and an sPGA score of clear or almost clear at Week 16 in each of the treatment groups.

None of the primary endpoints are safety issues.

## 5.1.2 Secondary Endpoints

None of the Secondary endpoints are safety issues.

## **Key Secondary Endpoints:**

The key secondary endpoints are as follows:

- Achievement of 75% reduction from baseline PASI score (PASI 75) at Week 16
- Achievement of 100% reduction from baseline PASI score (PASI 100) at Week 16
- Achievement of an sPGA score of clear (0) at Week 16
- Achievement of a Dermatology Life Quality Index (DLQI) score of 0 or 1 at Week 16
- Achievement of an sPGA score of clear or almost clear (0 or 1) at Week 52

## **Other Secondary Endpoints:**

The secondary endpoints are as follows:

- Achievement of PASI 75 at Week 52
- Achievement of PASI 90 at Week 52
- Achievement of PASI 100 at Week 52

Note that all key and other secondary endpoints at Week 52 will only be assessed for patients re-randomised at Week 28.

#### **5.1.3.** Further Endpoints

The further endpoints are as follows:

- Achievement of PASI 50 at all visits collected
- Achievement of PASI 75 at all visits collected
- Achievement of PASI 90 at all visits collected
- Achievement of PASI 100 at all visits collected
- Time until the first achievement of PASI 50, PASI 75, PASI 90, and PASI 100

11 Oct 2016

57704-04 Trial Protocol 

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

• Time until loss of PASI 50, PASI 75, PASI 90, and PASI 100 response for patients rerandomised at Week 28

- Change and percent change from baseline in PASI at all visits collected
- Absolute PASI of < 3 at all visits collected
- Achievement of an sPGA score of clear or almost clear at all visits collected
- Achievement of an sPGA score of clear at all visits collected
- Time until the first achievement of sPGA of 0 or 1
- Time until loss of sPGA of 0 or 1 response for patients re-randomised at Week 28
- Time until sPGA score of  $\geq$  3 (relapse) for patients re-randomised at Week 28
- Change from baseline in DLQI at all visits collected
- Achievement of a DLQI score of 0 or 1 at all visits collected
- Achievement of a reduction of 5 or more points from baseline in DLQI score at all visits collected
- Change from baseline in HAQ-DI at all visits collected, in patients selected for PsA assessment.
- Change and percent change from baseline on patient Pain VAS
- Change and percent change from baseline on patient Global Assessment VAS
- Change from baseline in Swollen or Tender Joint Count (28 joints) at all visits collected in patients selected for PsA assessment.
- Change from baseline in DAS28 at all visits collected in patients selected for PsA assessment.
- Change and percent change from baseline in Nail Psoriasis Severity Index (NAPSI) at all visits collected
- Change and percent change from baseline in Palmoplantar Psoriasis Severity Index (PPASI) at all visits collected
- Change and percent change from baseline in Psoriasis Scalp Severity Index (PSSI) at all visits collected
- Change of metabolic risk factors from baseline (waist circumference, body weight, HOMA-index)

See the Flow Chart for when the above measures are collected. The above endpoints will be analyzed, where appropriate, for re-randomized subjects after receiving open-label study drug for retreatment (Flow Chart 2 and 3).

## 5.2 ASSESSMENT OF EFFICACY

- The skin condition will be assessed by using the PASI, sPGA, and other relevant scores as described in CTP Section 5.1, Appendix 10, and the ISF.
- Symptoms, quality of life, and physical function will be assessed by DLQI and HAQ-DI.

Details of the efficacy assessments are listed in the Appendix (Section 10).

### 5.3 ASSESSMENT OF SAFETY

Safety will be assessed descriptively based on:

11 Oct 2016


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

**Trial Protocol** 

- Adverse events
- Serious adverse events
- Clinical laboratory values (haematology, clinical chemistry and urinalysis)
- Intensity of adverse events will be assessed by Rheumatology Common Toxicity Criteria (RCTC) version 2.0 (refer to ISF for details)

## 5.3.1 Physical examination

Complete physical examinations will be performed at visits noted in the Flow Charts. A complete physical examination will include vital sign assessment, and general appearance as well as evaluation of all relevant organ systems.

A targeted physical examination will be performed at visits noted in the Flow Charts. This includes vital sign assessment as well as an evaluation of the organ systems associated with AE(s) symptoms or laboratory abnormalities.

Clinically relevant abnormal findings will be reported as baseline conditions or AE's.

#### 5.3.1.1 Waist circumference

Waist circumference measurements should be made around a patient's bare midriff, after the patient exhales while standing without shoes and with both feet touching and arms hanging freely. The tape should be placed perpendicular to the long axis of the body and horizontal to the floor and applied with sufficient tension to conform to the measurement surface. Waist circumference should be determined by measuring the midpoint between the lowest rib and the iliac crest.

#### 5.3.1.2. Body weight

The scale used to capture body weight for each patient should remain consistent during the trial. In order to get comparable body weight values, it should be performed in the following way:

- Fasting (except for the screening visit);
- After the urine sampling (body weight after bladder voiding);
- Shoes and coat/jackets should be taken off; and
- Pockets should be emptied of heavy objects (i.e. keys, coins etc.)

## 5.3.2 Vital Signs

Vital sign evaluations will be performed at every visit as shown in the Flow Charts and includes temperature, pulse rate, systolic/diastolic blood pressure and respiratory rate. Respiratory rate, pulse rate, and blood pressure will be measured after patients have been sitting comfortably for at least five minutes. Measurement of vital signs should precede blood sampling to avoid the impact of blood sampling on the vital measurements. At dosing visits vital sign evaluations will be performed pre-dose. In addition at Visit 2 and Visit 3 vital sign evaluations will be taken at approximately 5 minutes post-dose (5 minutes after last injection) and approximately 60 minutes post-dose (60 minutes after last injection).

Patients should be closely monitored for signs and symptoms of hypersensitivity reactions for approximately 2 hours after the last injection at Visit 2 and for approximately 1 hour after the

11 Oct 2016

Trial Protocol 

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

last injection at all other visits where drug is administered. Hypersensitivity reactions should be treated according to medical standards. Pre-medications for further injections might be considered and will be agreed on between investigator and BI clinical monitor.

## 5.3.3 Safety laboratory parameters

For the visit schedule requiring safety laboratory sampling, see the Flow Charts. The laboratory tests listed in <u>Table 5.3.3: 1</u> will be performed at the central laboratory service provider. A local laboratory may be used for selected tests in exceptional cases. Patients should be fasting for at least 8 hours prior to the blood sample being taken (except screening visit).

Instructions regarding sample collection, sample handling/ processing and sample shipping are provided in the Laboratory Manual in the ISF.

Laboratory results (i.e. all safety laboratory and clinical laboratory data relevant for current clinical practice of psoriasis patients) of the patients will be available in real time to the respective investigator (via laboratory reports) and to the sponsor (via the central laboratory website) and selected abnormal laboratory alerts will be flagged to the site and sent to sponsor in real time.

Clinically relevant abnormal findings will be reported as baseline conditions or AE's. A clinically relevant value may be either inside or outside the reference range. Clinically relevant abnormal laboratory test results must be confirmed using an unscheduled visit laboratory kit and should be repeated until normalisation or stabilisation or until an alternative explanation has been found. Abnormal laboratory values will be also graded for intensity by using RCTC Version 2.0 criteria (R13-3515).

**57704-04** Trial Protocol 
Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies Table 5.3.3:1 Laboratory tests

| Category<br>Haematology | Hematocrit (Hct)<br>Hemoglobin (Hb) |
|---|---|
| | Hemoglobin (Hb) |
| | Glycosylated Hb (HbA1c) |
| | Red Blood Cell Count/ Erythrocytes |
| | Reticulocyte Count |
| | White Blood Cells / Leukocytes |
| | Platelet Count/ Thrombocytes |
| Diff. Automatic | Neutrophils (relative and absolute count) |
| DIII. Automatic | Eosinophils (relative and absolute count) |
| | Basophils (relative and absolute count) |
| | Monocytes (relative and absolute count) |
| | Lymphocytes (relative and absolute count) |
| Diff. Manual (if Diff Automatic is abnormal) | Neutrophils, bands (Stabs) |
| Diff. Manual (II Diff Automatic is automat) | |
| | Neutrophils, polymorphonuclear (PMN) |
| | Eosinophils |
| | Basophils |
| | Monocytes |
| | Lymphocytes |
| Coagulation | Activated Partial Thromboplastin Time (aPTT) |
| | Prothrombin time (INR) |
| | Fibrinogen |
| Enzymes | AST(GOT) |
| · | ALT(GPT) |
| | Alkaline Phosphatase (AP) |
| | Creatine Kinase (CK) |
| | CK-MB, (Only if CK is elevated) |
| | Gamma-Glutamyl Transferase (GGT/γ-GT) |
| | Lactic Dehydrogenase (LDH) |
| | Amylase |
| | Lipase |
| Electrolytes | Calcium |
| Licentrytes | Sodium |
| | Potassium |
| | Chloride |
| | Bicarbonate |
| Substrates | Glucose |
| | BUN |
| | Uric acid |
| | Creatinine |
| | eGFR (estimated by CKD-EPI formula) |
| | Bilirubin Total |
| | Bilirubin Direct (if total is elevated) |
| | Bilirubin Indirect (if total is elevated) |
| | Troponin (Reflex when CK is elevated) |
| | Albumin |
| | C-Reactive Protein (high sensitivity) |
| | Cholesterol, total |
| | Triglycerides |
| | LDL-Cholesterol (calculated) |
| | HDL-Cholesterol |
| | HOMA-IR (V2, V9, V15, V19, EOO) |
| Urine Pregnancy test <sup>1</sup> | Human Chorionic Gonadotropin in the urine |
| | * |
| Serum Pregnancy test <sup>2</sup> | Human Serum Chorionic Gonadotropin |

**Trial Protocol** 


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies Table 5.3.3:1 Laboratory tests

| Category | Test name |
|---|---|
| Hormones (screening) | TSH, |
| <del>-</del> | (free T3 and free T4 in case of abnormal TSH |
| | results) |
| Autoantibodies (screening) | Rheumatoid Factor |
| H: 1 : (G:) | TI ' YE'' |
| Urinalysis (Stix) | Urine Nitrite |
| | Urine Protein |
| | Urine Glucose |
| | Urine Ketone |
| | Urobilinogen |
| | Urine Bilirubin |
| | Urine RBC/ Erythrocytes |
| | Urine WBC/ Leukocytes |
| | Urine pH |
| Urine-Sediment (microscopic examination, only if | Urine Sediment Bacteria |
| urine analysis abnormal) | Urine Cast in Sediment |
| | Urine Squamous Epithelial Cells |
| | Urine Sed. Crystals., Unspecified |
| | Urine Sediment RBC/ Erythrocytes |
| | Urine Sediment WBC/ Leucocytes |
| Urinalysis | Albumin (quantitative) |
| • | Creatinine |
| | Albumin/Creatinine ratio |
| Infection Testing (Screening <sup>3</sup> V15, EOO) | Hepatitis B Surface Antigen (qualitative) |
| | Hepatitis C Antibodies (qualitative) |
| | HIV-1, and HIV-2 Antibody (qualitative) |
| | QuantiFERON®-TB <sup>3</sup> |

- 1. Urine pregnancy test performed on-site at all dosing visits (pre-dose) as well as EOT and EOO. (only for female patients of childbearing potential)
- 2. Serum pregnancy test at screening as well as confirmation of positive urine pregnancy test. (only for female patients of child bearing potential at screening as well as reflex for positive urine pregnancy test)
- 3. At Screening only TB testing is required. There is the site option to perform a PPD skin test, although this will not be provided or performed at Central Lab

## 5.3.4 Electrocardiogram

The 12-lead ECGs will be performed as scheduled in the Flow Chart(s).

ECGs will be recorded after the patients have rested for at least 5 minutes in a supine position and will always precede blood sampling. Six limb leads, as specified by Einthoven (I, II and III) and Goldberger (aVR, aVL, aVF), and six pre-cordial leads (V1–V6), according to Wilson, will be used.

ECGs will be read and evaluated by a central vendor. The study site will be informed about the results of the assessment of the ECG obtained at screening and if there are findings that would exclude the patient from study participation according to <a href="Exclusion Criterion#8"><u>Exclusion Criterion#8</u></a>. The electronic version of the ECG is regarded as source data.

**Trial Protocol** 


11 Oct 2016

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

ECGs may be repeated for quality reasons and the repeat used for analysis. Additional ECGs may be collected for safety reasons. Clinically significant abnormal findings will be reported as AE's.

Information about the details of ECG collection and the parameters assessed will be provided in the ISF.

## 5.3.5 Other safety parameters

#### 5.3.5.1 Local Tolerability

Local tolerability at the administration sites of the subcutaneous injections will be assessed according to "swelling", "induration", "heat", "redness", "pain", or "other findings" at the specified visits during the treatment period according to the flow chart. On visits where drug is administered this assessment should be done pre-dose. Clinically relevant findings will be reported as AE's.

#### 5.3.6 Assessment of adverse events

#### 5.3.6.1 Definitions of AEs

#### Adverse event

An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation patient administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment.

An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

#### Serious adverse event

A serious adverse event (SAE) is defined as any AE which:

- results in death,
- is life-threatening,
- requires inpatient hospitalisation or prolongation of existing hospitalisation,
- results in persistent or significant disability or incapacity,
- is a congenital anomaly/birth defect, or
- Is to be deemed serious for any other reason if it is an important medical event when based upon appropriate medical judgment which may jeopardize the patient and may require medical or surgical intervention to prevent one of the other outcomes listed in the above definitions.

11 Oct 2016

57704-04 Trial Protocol 
Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Life-threatening in this context refers to an event in which the patient was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if more severe.

For Japan only, the following events will be handled as "deemed serious for any other reason". An AE which possibly leads to disability will be reported as an SAE.

## AEs considered "Always Serious"

In accordance with the European Medicines Agency initiative on Important Medical Events, Boehringer Ingelheim has set up a list of AEs, which by their nature, can always be considered to be "serious" even though they may not have met the criteria of an SAE as given above.

The latest list of "Always Serious AEs" can be found in the Remote Data Capture (RDC) system. These events should always be reported as SAEs.

## Adverse events of special interest (AESIs)

The term AESI relates to any specific AE that has been identified at the project level as being of particular concern for prospective safety monitoring and safety assessment within this trial, e.g. the potential for AEs based on knowledge from other compounds in the same class. AESI need to be reported to the Sponsor's Pharmacovigilance Department within the same timeframe that applies to SAE, see Section 5.3.7.

The following are considered as AESIs:

## Hepatic injury

A hepatic injury is defined by the following alterations of hepatic laboratory parameters:

- an elevation of AST and/or ALT <u>></u>3 fold upper limit of normal (ULN) combined with an elevation of total bilirubin <u>></u>2 fold ULN measured in the same blood draw sample, and/or
- marked peak aminotransferase (ALT, and/or AST) elevations ≥10 fold ULN

These lab findings constitute a hepatic injury alert and the patients showing these lab abnormalities need to be followed up according to the "DILI checklist" provided in the ISF and the RDC-system.

In case of clinical symptoms of hepatic injury (icterus, unexplained encephalopathy, unexplained coagulopathy, right upper quadrant abdominal pain, etc.) without lab results (ALT, AST, total bilirubin) available, the investigator should make sure these parameters are analysed, if necessary in an unscheduled blood test. Should the results meet the criteria of hepatic injury alert, the procedures described in the DILI checklist should be followed.

#### **Intensity of AEs**

The intensity grading of AEs will be performed according to Rheumatology Common Toxicity Criteria (RCTC) Version 2.0 developed by OMERACT (R13-3515). Refer to the ISF for intensity/severity classification.

Intensity options are:

Grade 1: MILD

Grade 2: MODERATE

Grade 3: SEVERE

Grade 4: LIFE-THREATENING


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### Causal relationship of AEs

Medical judgment should be used to determine the relationship, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases and relevant history. Assessment of causal relationship should be recorded in the case report forms.

Yes: There is a reasonable causal relationship between the investigational product administered and the AE.

No: There is no reasonable causal relationship between the investigational product administered and the AE.

The causal relationship must be provided by the Investigator for all potential trial drugs, i.e. the BI trial drug and for all other trial drugs (such as any active comparator or placebo and for trial procedure).

<u>For Japan</u>, the reason for the decision on causal relationship for unlisted AEs needs to be provided in the eCRF

## 5.3.7 Adverse event collection and reporting

#### **AE Collection**

The following must be collected and documented in the eCRF by the Investigator:

- From signing the informed consent onwards through the Residual Effect Period until a patient's end of trial participation, all AEs (serious and non-serious), and AESIs must be collected.
- After the individual patient's completion of trial:

  The investigator does not need to actively monitor the patient for AEs, but should only report relevant SAEs and relevant AESIs of which the investigator may become aware of.

The REP is defined as 15 weeks after the last trial medication administration. All AEs that occur during the treatment phase and throughout the REP will be considered as on treatment (see Section 7.3.4). Events that occur after the REP will be considered as post treatment events.



#### Trial Protocol


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The Investigator must report SAEs, AESIs, and non-serious AEs which are relevant for the reported SAE or AESI, on the BI SAE form via fax immediately (within 24 hours ) to the Sponsor's unique entry point (country specific contact details will be provided in the ISF). The same timeline applies if follow-up information becomes available. In specific occasions the Investigator could inform the Sponsor upfront via telephone. This does not replace the requirement to complete and fax the BI SAE form.

In Japan, all SAEs and AESIs must be reported immediately to the head of the trial site. With receipt of any further information to these events, a follow-up SAE form has to be provided. For follow-up information the same rules and timeline apply as for initial information.

## **Information required**

For each AE, the Investigator should provide the information requested on the appropriate eCRF pages and the BI SAE form, e.g. onset, end date, intensity, treatment required, outcome, seriousness, and action taken with the investigational drug(s). The Investigator should determine the causal relationship to the trial medication, and the trial procedures outlined under Section 6.2.

The following should also be recorded as an (S)AE in the eCRF and SAE form (if applicable):

- Worsening of the underlying disease or of other pre-existing conditions
- Changes in vital signs, ECG, physical examination and laboratory test results, if they are judged clinically relevant by the Investigator.

If such abnormalities already pre-exist prior trial inclusion they will be considered as baseline conditions.

All (S)AEs, including those persisting after individual patient's end of trial must be followed up until they have resolved, have been sufficiently characterized, or no further information can be obtained.

#### **Screening failures:**

SAEs which occurred <u>during</u> the screening period are to be reported according to standard procedures.

#### **Pregnancy**

In the rare case that a female patient participating in this clinical trial becomes pregnant after having taken trial medication, the Investigator must report immediately (within 24 hours) the drug exposure during pregnancy (DEDP) to the Sponsor's unique entry point (country-specific contact details will be provided in the ISF). The Pregnancy Monitoring Form for Clinical Trials (Part A) should be used.

If a patient becomes pregnant during a trial, the study medication needs to be discontinued, and the patient will complete the EOT Visit procedures and Follow-up 1 and Follow-up 2 (EOO) Visit procedures. The patient will be followed up until birth or otherwise termination of the pregnancy.

The outcome of the pregnancy associated with the drug exposure during pregnancy must be followed up and reported to the Sponsor's unique entry point on the Pregnancy Monitoring Form for Clinical Trials (Part B).

**Trial Protocol** 


11 Oct 2016

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

As pregnancy itself is not to be reported as an AE, in the absence of an accompanying SAE, only the Pregnancy Monitoring Form for Clinical Trials and not the SAE form is to be completed. If there is an SAE associated with the pregnancy then the SAE has to be reported on the SAE form in addition.

The ISF will contain the Pregnancy Monitoring Form for Clinical Trials (Part A and B).

## 5.4 DRUG CONCENTRATION MEASUREMENTS AND PHARMACOKINETICS

#### 5.4.1 Assessment of Pharmacokinetics

BI 655066 concentrations will be reported descriptively. No PK parameters will be calculated. PK data will be incorporated into a larger pharmacometric analysis with other trials of BI 655066 project. The relationship between PK and selected efficacy endpoints, biomarkers and AEs may be assessed.

PK and demographic data together with treatment assignments and dosing information may be made available to individuals outside of the trial team for the purpose of PK dataset generation in accordance with sponsor's standard procedures.

Refer to the Flow Charts for the visits requiring PK and ADA sampling. The date and exact clock time of drug administration and PK and ADA sampling will be recorded on the eCRF. These actual administration and sampling times will be used for determination of PK parameters. On visits with study medication dosing, PK and ADA sampling should be collected prior to administration of study drug.

After completion of the study, PK and ADA plasma samples may be used for further methodological investigations, e.g., stability testing. However, only data related to the analyte will be generated by these additional investigations.

## 5.4.2 Methods of sample collection

## 5.4.2.1 Plasma sampling for pharmacokinetic analysis

For quantification of analytic plasma concentrations, approximately 2.5 mL of blood will be taken at the time points listed in the Flow Chart under PK sampling.

Detailed instructions for pharmacokinetic sampling, handling, and shipment of plasma samples are provided in the laboratory manual.

## 5.4.2.2 Plasma sampling for ADA

For ADA assessment, approximately 2.5 mL of blood will be taken at the time points listed in the Flow Chart under ADA sampling. Detailed instructions for ADA sampling, handling, and shipment of plasma samples are provided in the laboratory manual.

#### 5.4.3 Analytical determinations

BI 655066 concentrations will be determined by a validated Enzyme Linked Immunosorbent Assay (ELISA).

The presence of ADA to BI 655066 will be assessed via a tiered approach using a validated electrochemiluminescence assay (screening, confirmatory, and titration analysis as appropriate).

**Trial Protocol** 


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Samples that are confirmed positive may be further characterized in a validated neutralizing antibody (NAb) assay.

## 5.4.4 Pharmacokinetic-Pharmacodynamic Relationship

Refer to Section 7.3.6.

#### 5.5 ASSESSMENT OF EXPLORATORY BIOMARKERS

## 5.5.1 Assessment of soluble protein biomarkers in blood

Serum will be collected pre and post treatment with BI 655066 to assess changes in protein levels of disease specific markers such as but not limited to  $\beta$ -defensin 2, neutrophil gelatinase associated lipocalin-2 (NGAL) and S-100 A8 protein.

In addition changes in levels of biomarkers related to metabolic syndrome, such as leptin, resistin, TNFa, IL-6 and vascular endothelial growth factor (VEGF) will be explored.

Blood samples will be stored for a maximum of 3 years (under consideration of local legislation) upon signature of the final study report unless the patient agrees to long-term storage (15 years) of the biomarker samples for biomarker sample banking (Section 5.5.3).

## 5.5.1.1 Methods of sample collection

For the assessment of soluble protein biomarkers in serum, approximately 12.5 ml of blood will be collected at the time points indicated in the flow charts. Samples should be collected prior to the administration of study drug at dosing visits. For details on sample collection, processing and logistics refer to the ISF (Laboratory Manual).

#### 5.5.1.2 Analytical determinations

These biomarkers are considered exploratory and respective assays will need to be qualified to meet the required performance criteria.

## 5.5.2 DNA Banking

Participation in the DNA Banking sampling is voluntary and not a prerequisite for participation in the trial. The patient must provide informed consent for participation in this optional testing prior to any blood sampling used for DNA Banking.

The DNA Banking sample will be stored in accordance with local ethical and regulatory requirements.

## 5.5.2.1. Methods of sample collection

One blood sample for DNA banking will be taken at Visit 2. A maximum of 8.5 mL blood will be collected per PaxGene DNA blood sampling tube. For details on sample handling and logistics refer to the ISF (Laboratory Manual).

11 Oct 2016

Trial Protocol 

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 5.5.2.2. Analytical determinations

The DNA Banking sample, derived from the original blood sample, will be stored at AbbVie or a third party delegate (e.g. Boehringer Ingelheim Pharma GmbH & Co. KG; Birkendorfer Str. 65, 88397 Biberach, Germany). The stored DNA may be retrospectively analysed, e.g. to identify whether there are other genetic factors that could contribute to a better therapeutic outcome or a higher risk of developing treatment-related adverse drug reactions.

## 5.5.3 Biomarker sample banking

After completion of the study any unused serum, collected for biomarker sampling as listed in <u>Section 5.5.1.</u> may be used for further investigations, (e.g., additional biomarkers for immunological & inflammatory diseases) if informed consent for biomarker sample banking is agreed upon by the patient.

Declination to allow storage and use of these unused samples will not preclude participation in this study. The study samples will be stored for a maximum period of 15 years (under consideration of local legislation and if consented by the patient) upon archiving of the final study report after study termination.

#### 5.6 OTHER ASSESSMENTS

Not applicable

#### 5.7 APPROPRIATENESS OF MEASUREMENTS

All measurements performed during this trial are standard measurements in psoriasis treatment trials and will be performed in order to monitor safety aspects or assess treatment response in an appropriate way.

Information about race should be obtained from all study participants as allowed by local regulations. This is because the prevalence and characteristics of psoriasis differ widely between patients of different racial origin. It will thus be worthwhile to assess if patients of different race will respond differently to the study treatment.

c03357704-04

**Trial Protocol** 


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 6.0 INVESTIGATIONAL PLAN

#### 6.1 VISIT SCHEDULE

All patients have to adhere to the visit schedule as specified in the Flow Charts. Each visit date (with its window) is to be counted from Day 1.

If any visit has to be rescheduled, subsequent visits should follow the original visit date scheduled. Additional visits for the purpose of re-testing of laboratory parameters or AE monitoring may be included as deemed necessary by the investigator.

For detailed description of the trial procedures, please refer to the Flow Charts.

#### 6.2 DETAILS OF TRIAL PROCEDURES AT SELECTED VISITS

Study procedures to be performed at each visit are listed in the Flow Charts and the respective protocol sections. Refer to Section 5.3 and the Appendix Section 10 for explanations of the procedures. Additional details on select procedures are provided below.

Patients should be seen for all visits on the designated day within the allowed "visit window" as specified in the Flow Charts. Measurement of vital signs should precede blood sampling and be assessed pre-dose at all dosing visits. Patient reported outcomes (PROs) should be completed electronically during clinic visits by the patient on his/her own in the following order, as programmed in the electronic device:

- (1) DLQI
- (2) HAQ-DI [for psoriatic arthritis patients at selected sites]
- (3) Pain VAS [for psoriatic arthritis patients at selected sites]
- (4) Patient Global Assessment (PtGA) VAS [for psoriatic arthritis patients at selected sites]

PROs should be completed by the patient in a quiet area/room before any other visit assessments or treatments, and, when possible, before any interaction with the investigator or other members of the study team. Timing for downloading the data of PROs will be available in the ISF.

The following psoriasis efficacy assessments (PASI, sPGA, NAPSI, PPASI and PSSI) and psoriatic arthritis assessments (CASPAR and Tender or Swollen joint counts (TJC/SJC)) will be performed by a qualified efficacy assessor at the site by direct capture using an electronic device. Efficacy assessor qualifications and The Group for Research and Assessment of Psoriasis and Psoriatic Arthritis (GRAPPA) training requirements will be available in the ISF.

#### Tuberculosis (TB) Testing

Patients will be tested for TB (Quantiferon or PPD) at Screening, Week 52 and EOO. Patients who test positive and are at low risk of TB reactivation, per local guidelines and investigator judgment, do not need to be treated with prophylactic anti-tuberculosis medication and can be entered or continue in the trial.

#### 6.2.1 Screening period

After patients have been informed about the trial, written informed consent in accordance with GCP and the local legislation must be obtained prior to performing any study related procedures. Once they have consented, the patient is considered to be enrolled in the trial and have started screening. The patient should be recorded on the enrolment log and be registered

11 Oct 2016

Trial Protocol 

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

in IRT as a screened patient. Patients will be assigned a patient number and enrolment must be recorded in eCRF pages.

The Screening period is defined as the period from the Screening visit to Randomisation (first study drug administration). The screening period should be no longer than 42 days and no less than 7 days and will be used to assess eligibility of the patients and to taper the patients off disallowed medications. Thus patients will not be randomized until all screening procedures are completed and results are reviewed to verify study eligibility. Screening procedures may be extended to more than 1 physical visit if needed.

## Re-Screening

Re-screening will not be permitted. Patients who fail screening following Visit 1 assessments should be registered as a screen failure in IRT within the protocol defined screening period. For the comprehensive list of the trial procedures required at the Screening Visit (Visit 1) please refer to Flow Chart #1.

## **Demographics**

Informed consent date, HIPAA status (US patients only), sex, ethnicity and race (if allowed by local law) will be collected and reported in the eCRF.

## **Baseline Conditions**

Chronic diseases, current observable conditions, any new clinically relevant findings discovered from the Physical Exam, ECG, safety labs, and any condition requiring therapy (excluding psoriasis) will be reported on the Baseline Condition eCRF page.

## **History for Psoriatic Arthritis**

At Visit 1, all patients at all sites will be evaluated for history of psoriatic arthritis.

#### Psoriatic Arthritis Diagnosis Assessment

At Visit 1 at pre-selected study sites, all patients with a positive medical history of psoriatic arthritis will be further evaluated for psoriatic arthritis (PsA) diagnosis based on CASPAR (Classification of Psoriatic Arthritis) criteria. See <u>Appendix 10.6</u> for further details

#### IRT

All patients that are screened must be registered with IRT. If the patient results in a screen failure, IRT should be notified as soon as possible and within the 42- day screening period. Details of IRT procedures can be found in the IRT manual located in the ISF

## 6.2.2 Treatment period

The Treatment period consists of a maximum of 20 visits (Visits 2-21). Visit 2 is the Randomisation Visit and Visit 21 is end of treatment (EOT) visit, where the last dose of medication will be administered.

#### Unscheduled Visits

During the treatment period patients may be seen at an unscheduled visit if they experience deterioration of psoriasis (i.e. between Weeks 32 and 88 for patients in the double blind portion of the study to assess relapse), or have AEs that in the opinion of the investigator need intervention or repeated laboratory testing.

11 Oct 2016

**Trial Protocol** 


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## Safety laboratory testing

All visits after screening requiring safety laboratory sampling will be performed in a fasted state (8 hours no food and only water). If a patient comes in non-fasted where a fasting condition is required, the visit should be performed, the non-fasted condition documented on the laboratory requisition, and the patient reminded about the expected conditions.

#### Pregnancy testing

Urine pregnancy testing for all woman of childbearing potential will be conducted on-site prior to every dosing and must be negative to further treat the patient. A positive urine test must be confirmed with a serum pregnancy test.

#### Psoriatic arthritis assessments (at selected study sites)

Refer to the Flow charts as well as Appendix 10.6 for timing and assessments.

## C-Reactive protein (CRP)

Safety laboratory assessments include CRP testing. The result of the CRP will be used to calculate the DAS28 at the associated visit. See also Appendix 10.6.1.

At treatment period visits all the study procedures described in the Flow-Charts will be performed before the administration of the study medication.

## Randomisation (Visit 2)

Randomisation via IRT and administration of the first dose of study medication should be the last activity at Visit 2.

#### Week 28 Visit

At Week 28, each patient's sPGA score will be entered into IRT. Refer to the ISF for details pertaining to IRT procedures and requirements.

All patients that are responding to treatment (sPGA of 0 or 1) at Week 28 will be dispensed blinded medication kits; see (Section 7.6.).

All patients who are non-responders (sPGA  $\geq 2$ ) at week 28, regardless of initial treatment arm, should continue in this trial and will be dispensed open label BI 655066 medication kits until the end of the treatment period (Week 88).

## Randomized withdrawal period (Re-randomized patients)

Between Week 32 and Week 82, at scheduled or unscheduled visits, once any Week 28 responder's sPGA increases to  $\geq 3$  (relapse) the site will enter this result into IRT, and IRT will immediately dispense open label BI 655066 medication. The patient will immediately follow Flowchart #2 or Flowchart #3 depending on the time of relapse. The patient will be re-treated for a maximum of 16 weeks and then have the opportunity to roll-over to the OLE study for further treatment. (See Section 6.2.3). All patients following Flow Chart 2 or Flow Chart 3 will receive a loading dose 4 weeks after the first re-treatment.

Patients relapsing at either an unscheduled visit between Week 82 and Week 88 or at the scheduled Week 88 visit will have the EOT visit procedures performed and return for Follow-up 1 and Follow-up #2 visits as scheduled. A loading dose will not be administered. These patients will also have the opportunity to rollover to the OLE study (See Section 6.2.3)

**Trial Protocol** 


11 Oct 2016

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## **6.2.3** Follow up Period and Trial Completion

For all randomized patients termination of trial medication and trial completion must be recorded on the corresponding eCRF.

The follow-up period within this trial is 16 weeks after receiving the last dose of study medication. Refer to the flow charts for the list of procedures required.

## Early treatment and trial termination

If study medication is discontinued prior to the planned Flow Chart EOT visit, every effort should be made to have the patient continue in the trial and complete all of the remaining Treatment Period Visits, as well as Follow-Up 1 and Follow-Up 2 Visits. Trial termination should be completed at Follow-Up 2 Visit.

If a patient cannot or will not continue in the trial, the patient should complete EOT visit procedures instead of the planned treatment period visit and return to the clinic for Follow-Up 2/End of Observation (FU2/EOO) Visit 16 weeks after last dose of study medication.

Patients who discontinue treatment early should be registered as withdrawn/discontinued in IRT and will not have the option to participate in the OLE trial.

## Successful trial completion

Patients who complete treatment according to the applicable planned Flow Chart visit schedule will return to the clinic for Follow-up Visit 1, (6 weeks after last dose of study medication) and for the EOO visit (16 weeks after last dose of study medication). Trial completion is defined as patients completing the EOO visit within the specified window per the flow charts, and who have not discontinued drug prematurely. These patients should be registered as completed in IRT at the EOO visit. These patients will have the option to participate in the open label extension (OLE) trial once EOO procedures are completed.

Refer to ISF for OLE trial entry details.

#### Vital Status

For randomized patients leaving the study early (before the planned EOO in their current applicable flow chart), vital status should be collected every 12 months after discontinuation up to the planned EOO.

c03357704-04

11 Oct 2016

#### **Trial Protocol**


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 7.0 STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

## 7.1 STATISTICAL DESIGN - MODEL

This is a confirmatory, multicenter, randomized, double-blind, placebo controlled study with randomized withdrawal and re-treatment, evaluating the efficacy and safety of BI 655066 in patients with moderate to severe chronic plaque psoriasis. The primary objectives of this trial are to assess the safety and efficacy of BI 655066 in comparison to placebo in patients with moderate to severe chronic plaque psoriasis. The primary efficacy will be evaluated at 16 weeks. In addition, the maintenance of response following drug withdrawal will be assessed after Week 28 through Week 104. Subsequent to drug withdrawal, patients who experience relapse (sPGA  $\geq$ 3) will be retreated with BI 655066 to assess response after retreatment. Randomisation will be stratified by weight ( $\leq$  100 kg vs.  $\geq$ 100 kg) and prior exposure to TNF antagonists (0 vs.  $\geq$ 1). Based upon these design considerations and the binary nature of the coprimary endpoints of PASI 90 and sPGA 0 or 1, the trial will be analysed using the Cochran-Mantel-Haenszel risk difference estimate stratified by the randomisation factors mentioned previously. Baseline refers to the measurement recorded at randomisation (Visit 2); if data at Visit 2 is missing or not collected per protocol, then data from Visit 1 will be considered baseline.

In addition, this trial will assess PK and the emergence of anti-drug antibodies (ADA) and their effect on efficacy and safety. Moreover, it will be explored how the use of BI 655066 may influence gene and protein expression levels and disease specific protein markers. More details on these analyses will be provided in the Trial Statistical Analysis Plan (TSAP).

The percent reduction from baseline is calculated by % PASI reduction from baseline = ((PASI at baseline - PASI at Visit Y) / PASI at baseline) \* 100, at all follow up visits. Achieving an X% or larger reduction from baseline PASI score is denoted as PASI X.

Re-randomisation at Week 28 will also be stratified by weight ( $\leq 100 \text{ kg vs.} > 100 \text{ kg}$ ) and prior exposure to TNF antagonists (0 vs.  $\geq 1$ ).

#### 7.2 NULL AND ALTERNATIVE HYPOTHESES

The primary hypotheses are that BI 655066 is different than placebo in achieving  $\geq 90\%$  reduction from baseline in the Psoriasis Area and Severity Index score (PASI 90) and sPGA of 0 or 1 at Week 16 in participants with moderate to severe chronic plaque psoriasis. For the primary analyses, this study has 2 treatment arms:

- Arm 1 Patients randomised at visit 2 to receive 150 mg of BI 655066
- Arm 2 Patients randomised at visit 2 to receive placebo

For Part B of the trial, patients randomised to receive BI 655066 at visit 2 and have an sPGA response of 0 or 1 at Week 28 will be re-randomised to one of the following treatment arms:

Arm A – Patients re-randomised to continue to receive BI 655066 during Part B

Arm B – Patients re-randomised to receive placebo during Part B

**Trial Protocol** 


11 Oct 2016

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The following null hypotheses will be tested in a hierarchical order using two-sided tests with a type I error of 0.05. The two co-primary endpoints need to be significant simultaneously, therefore no alpha adjustment is necessary.

- 1. BI 150 mg (Arm 1) is not different from placebo (Arm 2) with respect to PASI 90 or sPGA 0 or 1 response at Week 16
- 2. BI 150 mg (Arm 1) is not different from placebo (Arm 2) with respect to PASI 75 response at Week 16
- 3. BI 150 mg (Arm 1) is not different from placebo (Arm 2) with respect to PASI 100 response at Week 16
- 4. BI 150 mg (Arm 1) is not different from placebo (Arm 2) with respect to achieving an sPGA score of clear (0) at Week 16
- 5. BI 150 mg (Arm 1) is not different from placebo (Arm 2) with respect to achieving a DLOI score of 0 or 1 at Week 16.

For the re-randomized patients, the following null hypothesis will be performed with a type I error of 0.05.

• Arm A (patients re-randomised to BI 655066) is not different from Arm B (patients re-randomised to placebo) with respect to sPGA 0 or 1 response at Week 52.

#### 7.3 PLANNED ANALYSES

The efficacy analyses will be based on the intent-to-treat principle, comprising all participants who were randomized and received at least one dose during the trial. Misrandomized patients are by definition screening failures and therefore are not included in the intended to treat population. Efficacy analyses will be based on the planned treatment (i.e., the treatment assigned at randomisation); this set of patients is called the Full Analysis Set (FAS). Safety analyses will be based on the actual treatment received at the randomisation visit; this set of patients is called the Safety Set (SAF).

All efficacy analyses will be conducted on the FAS. All safety analyses will be conducted on the SAF.

Important violations of the protocol will include key inclusion and exclusion violations, incorrect medications taken, compliance with study medication, incorrectly re-randomized or not re-randomized, concomitant use of restricted medications, and any other violations of the protocol deemed important by the study team. All decisions concerning important protocol violations will be made prior to unblinding of the database. A per-protocol set (PPS) will be defined excluding patients with violations that affect Week 16 efficacy. A secondary re-randomized per-protocol set (RRS-PPS) will be defined excluding those patients with violations affecting Week 52 efficacy of randomized withdrawal. The hypothesis tests as described in Section 7.2 will be repeated on the PPS or RRS-PPS populations, as appropriate.

## 7.3.1 Primary endpoint analyses

The achievement of PASI90 at Week 16 is the first co-primary endpoint and is a binary variable with values of 0 or 1. The difference in proportion responding between the BI 150 mg arm and placebo arm will be estimated and tested using the Cochran-Mantel-Haenszel risk difference

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

estimate stratified by the randomisation factors of weight ( $\leq$  100 kg vs. >100 kg) and prior exposure to TNF antagonists (0 vs.  $\geq$ 1) with weights proposed by Greenland & Robins, which is calculated as follows:

$$\hat{\delta}_{MH} = \frac{\sum_{i=1}^{u} w_i \cdot \hat{\delta}_i}{\sum_{i=1}^{u} w_i} \text{ , where }$$
 
$$\hat{\delta}_i = \frac{x_i}{n_i} - \frac{y_i}{m_i} \text{ denotes the risk difference in stratum } i, i = 1, \cdots, u$$
 
$$w_i = \frac{n_i \cdot m_i}{n_i + m_i} \text{ denotes the weight of stratum } i, i = 1, \cdots, u$$

 $x_i$  denotes the number of patients with event in treatment<sub>1</sub>in stratum i,  $i=1,\cdots,u$   $y_i$  denotes the number of patients with event in treatment<sub>2</sub>in stratum i,  $i=1,\cdots,u$   $n_i$  denotes the number of patients on treatment<sub>1</sub>in stratum i,  $i=1,\cdots,u$   $m_i$  denotes the number of patients on treatment<sub>2</sub>in stratum i,  $i=1,\cdots,u$ 

The estimated variance of  $\hat{\delta}_{MH}$  is calculated as:

$$\begin{split} \widehat{var}\big(\hat{\delta}_{MH}\big) &= \frac{\sum_{i=1}^{u} L_i}{(\sum_{i=1}^{u} w_i)^2} \\ \text{where } L_i &= \frac{x_i(n_i - x_i) \ m_i^3 + y_i(m_i - y_i) \ n_i^3}{n_i \cdot m_i \cdot (n_i + m_i)^2} \ \text{, } i = 1, \cdots \text{, } u \end{split}$$

Assuming a normal distribution of  $\hat{\delta}_{MH}$ , an approximate 95% CI is given as follows, where  $z_{0.975}$  is the 97.5% quantile of the standard normal distribution:

$$CI = \left[\hat{\delta}_{MH} \pm z_{0.975} \cdot \sqrt{\widehat{var}(\hat{\delta}_{MH})}\right]$$

Also, the approximate p-value can be calculated using the following:

pvalue = 
$$2 \cdot \Pr \left[ Z > \frac{\hat{\delta}_{MH}}{\sqrt{\widehat{var}(\hat{\delta}_{MH})}} \right]$$
, where  $Z \sim N(0, 1)$ 

If there is a stratum for a treatment group that has 0 patients in it, the 0 count will be replaced by 0.1 in order to prevent dividing by 0 in the above equations, as suggested in Greenland & Robins (R09-1299). Pairwise comparisons of the BI 150 mg arm and placebo arm will include both a p-value and 95% confidence interval.

The achievement of an sPGA score of clear or almost clear at Week 16 is the second coprimary endpoint and is a binary variable with values of 0 or 1. The analysis of the sPGA coprimary endpoint will be identical to that of the PASI90 co-primary endpoint detailed above.

#### 7.3.2 Secondary endpoint analyses

#### **Key Secondary Endpoints:**

The achievement of PASI75 at Week 16 is a binary variable with values of 0 or 1. The analysis of this endpoint will be identical to that of the PASI90 co-primary endpoint detailed in <u>Section 7.3.1</u>.

The achievement of PASI100 at Week 16 is a binary variable with values of 0 or 1. The analysis of this endpoint will be identical to that of the PASI90 co-primary endpoint detailed in Section 7.3.1.

## Trial Protocol 

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The achievement of an sPGA score of clear at Week 16 is a binary variable with values of 0 or 1. The analysis of this endpoint will be identical to that of the PASI90 co-primary endpoint detailed in Section 7.3.1.

The achievement of a DLQI score of 0 or 1 at Week 16 is a binary variable with values of 0 or 1. The analysis of this endpoint will be identical to that of the PASI90 co-primary endpoint detailed in Section 7.3.1.

The achievement of an sPGA score of clear or almost clear at Week 52 is a binary variable with values of 0 or 1. The analysis of this endpoint will be identical to that of the PASI90 co-primary endpoint detailed in Section 7.3.1. Note that this endpoint will only be analysed for patients rerandomised at Week 28 (i.e., only for Arm A and Arm B defined in Section 7.2).

## **Other Secondary Endpoints:**

All of the other secondary endpoints are binary variables with values of 0 or 1. The analysis of these endpoints will be identical to that detailed in Section 7.3.1.

Note that all other secondary endpoints will only be analysed for patients re-randomised at Week 28 (i.e., only for Arm A and Arm B defined in Section 7.2).

## 7.3.3 Further endpoint analyses

Further endpoints will be summarized, with number and proportion of responders for dichotomous endpoints and mean, median, SD and IQR presented for continuous variables. Time to onset of *Endpoint*, the time to event will be calculated as:

- Time to first onset (with observed event) = [date of first onset] [date of first active treatment] + 1
- If a patient never attains *Endpoint* (e.g., PASI75 or PASI90), then that patient's time to first onset will be censored at the last visit where the *Endpoint* was measured (e.g., PASI).

Time to Loss of *Endpoint* will only be performed for patients that are re-randomised at Week 28 (i.e., Arms A and B defined in Section 7.2), where day 0 is defined as the date of the Week 16 visit. Time to loss is defined using the following algorithm:

- a) Never attains *Endpoint* (Failure at day 0)
- b) After achieving *Endpoint*, patient will be a failure if they subsequently do not achieve *Endpoint* and either discontinue from the study or switch therapy while still not achieving *Endpoint*. Time to failure will be calculated using date of first failure to achieve *Endpoint*.
- c) Patients that take prohibited meds to treat Psoriasis will be counted as failures at the time when they first take the prohibited med.
- d) Patients that switch therapy while maintaining response will be censored at their last measurement prior to switching treatment. A switch from active medication to Placebo does not constitute a change in treatment.
- e) Patients who maintain *Endpoint* throughout the study will be censored at their last measurement.

Time to Loss of *Endpoint* (from time of achieving *Endpoint* or from specific point in time) will be defined as above but only for those patients that have achieved *Endpoint*.

11 Oct 2016

#### Trial Protocol


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

All Time to Event endpoints will be presented using Kaplan-Meier curves with comparisons made between treatment groups using stratified Log-Rank test. Further information will be provided in the TSAP.

## 7.3.4 Safety analyses

Adverse events will be coded using the Medical Dictionary for Drug Regulatory Activities (MedDRA) coding dictionary. Standard AbbVie summary tables and listings will be produced. All adverse events with an onset between start of treatment and end of the residual effect period (REP), a period of 15 weeks days after the last dose of trial medication, will be assigned to the treatment period for evaluation.

All treated patients will be included in the safety analysis. In general, safety analyses will be descriptive in nature and will be based on AbbVie standards. No hypothesis testing is planned.

Statistical analysis and reporting of adverse events will concentrate on treatment-emergent adverse events. To this end, all adverse events occurring between start of treatment and end of the residual effect period will be considered 'treatment-emergent'. Adverse events that start before first drug intake and deteriorate under treatment will also be considered as 'treatment-emergent'.

Frequency, severity, and causal relationship of adverse events will be tabulated by system organ class and preferred term after coding according to the current version of the Medical Dictionary for Drug Regulatory Activities (MedDRA).

Laboratory data will be analysed both quantitatively as well as qualitatively. The latter will be done via comparison of laboratory data to their reference ranges. Values outside the reference range as well as values defined as clinically relevant will be highlighted in the listings. Treatment groups will be compared descriptively with regard to distribution parameters as well as with regard to frequency and percentage of patients with abnormal values or clinically relevant abnormal values.

Vital signs, physical examinations, or other safety-relevant data observed at screening, baseline, during the course of the trial and at the end-of-trial evaluation will be assessed with regard to possible changes compared to findings before start of treatment.

More information on the analysis of safety will be given in the TSAP.

## 7.3.5 Pharmacokinetic analyses

Descriptive statistics of BI 655066 concentration measurements by treatment group and visit will be provided.

Pharmacokinetic data will be analyzed using population pharmacokinetic approaches. For this purpose, data may also be combined with data from other trials.

#### 7.3.6 Pharmacodynamic analysis

No formal analysis of pharmacokinetic-pharmacodynamic relationships is planned. As the data from previous trials with BI 655066 suggest a pharmacokinetic (PK)-pharmacodynamic (PD)

Boehringer Ingelheim BI Trial No.: 1311.0004

11 Oct 2016

c03357704-04 Trial Protocol 

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Proprietary confidential information © 2016 Boenringer Ingelineim International Gmoh or one or more of its artiflated companies

relationship for efficacy endpoints such as PASI, population PK-PD analyses will be performed. For this purpose, data may also be combined with data from other trials. Model-based analyses will be planned and documented separately according to internal and external guidelines and SOPs. Other exploratory analyses of drug concentration, biomarker or safety data may be performed using data obtained as part of this trial.

All modeling activities will be planned and documented separately according to internal and external guidelines and SOP.

## 7.3.7 Biomarker analyses

Changes in serum protein biomarker levels over time will be described by treatment group. The details of these analyses will be included in the TSAP.

#### 7.4 INTERIM ANALYSES

There will not be an interim analysis from a statistical standpoint. An analysis will be conducted after the last patient either has been in the study for 52 weeks or discontinues from the study. All primary and key secondary endpoints are collected by Week 52; hence no alpha adjustment is required at this analysis. For this analysis all efficacy endpoints and safety will be analysed. The Sponsor will be unblinded to perform this analysis. Blinded treatment assignments will not be disseminated to the sites, investigators, and patients until the end of study database lock. If needed, more details about this analysis will be specified in the TSAP.

## 7.5 HANDLING OF MISSING DATA

Every effort should be made to collect complete data at all visits.

The following rules will be used to impute for missing data:

- For all non-binary endpoints, last observation carried forward (LOCF) will be used to impute missing values
- For all binary endpoints (i.e. endpoints that are either 1 (patient responded) or 0 (patient did not respond)):
  - If no data after that visit\*, then impute as failure (NRI [No Response Imputation])
- If data at visits\* before and after, only impute as success if both visits are successes; else impute as failure
- \* Patients that take prohibited medications to treat Psoriasis will be treated the same as those that discontinued from the trial i.e. subsequent visits following start of prohibited medication will be considered as failure for binary endpoints.

Missing items from the PRO questionnaires will be handled according to the measure instructions (Section 10.7). If there is no data for a particular visit, then it will be imputed following the same rules as described above.

Sensitivity analyses to assess the robustness of the hypothesis testing results will include the following methods where applicable:

- LOCF (for binary endpoints)
- Logistic regression

**Trial Protocol** 


11 Oct 2016

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Mixed effect Model Repeat Measurement (MMRM) (for continuous endpoints)

• Multiple imputation (for binary endpoints)

Of note, for randomized withdrawal analyses, subjects who received retreatment will be counted as non-responders in all visits after the date of retreatment.

#### 7.6 RANDOMISATION

At Visit 2, patients will be randomized in blocks to double-blind treatment to either BI 655066 150 mg or placebo in a 4:1 ratio. Randomisation will be stratified with respect to weight ( $\leq$  100 kg vs.  $\geq$ 100 kg) and prior exposure to TNF antagonists (0 vs.  $\geq$ 1).

At week 28, patients will be separated into "responder" and "non-responder" groups. A patient will be considered as a "responder" if the week 28 sPGA is clear or almost clear (0 or 1); otherwise the patient will be considered a "non-responder".

Among responders, patients originally randomized to BI 655066 150 mg (Arm 1) will be rerandomized in a 1:2 ratio to either 150 mg of BI 655066 or placebo in a second double-blinded portion (Part B) of the trial. Re-randomisation will be stratified by weight (≤ 100 kg vs. >100 kg) and prior exposure to TNF antagonists (0 vs. ≥1). Patients originally randomized to placebo (Arm 2) will continue to receive blinded study drug every 12 weeks in Part B of the trial, to maintain the blind to the original randomized treatment arm.

Regardless of originally randomized treatment group, non-responders will receive open label BI 655066 every 12 weeks, starting at Week 28, for the remainder of the trial. BI will arrange for the randomisation and the packaging and labelling of trial medication. The randomisation lists will be generated using a validated system, which involves a pseudo-random number generator so that the resulting treatment will be both reproducible and non-predictable. The block sizes will be documented in the Clinical Trial Report (CTR). Access to the codes will be controlled and documented.

#### 7.7 DETERMINATION OF SAMPLE SIZE

This study is designed to show a difference between BI 655066 and placebo in terms of PASI90 response and sPGA scores of clear or almost clear at Week 16. However, this study was also powered to show a difference in sPGA response at Week 52 between the patients randomized to continue on BI 655066 vs. patients randomized to placebo at Week 28.

Based on the interim results from 1311.2 (c03272682-01), it is assumed at most 10% of the patients in the re-randomized BI 655066 arm will lose sPGA response of clear or almost clear (0 or 1) at Week 52 whereas approximately 25% of patients in the re-randomized placebo arm will lose response. Using a 1:2 re-randomisation scheme (BI 655066:placebo), 102 patients in the BI 655066 arm and 204 patients in the placebo arm will provide at least 90% power to detect the difference in sPGA response rate at Week 52. Assuming that 80% of patients on BI 655066 at baseline will achieve sPGA of clear or almost clear at Week 28, the total sample size required for the initial BI 655066 arm at Visit 2 is (102)(3)÷0.8=383. See Table 7.7:1 for more sample size calculations to have at least 90% power.


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 7.7:1 Sample sizes for randomized withdrawal comparison

| Response Rate at Week 52 | | Randomisation ratio at Week 28 active:placebo = Total N | Total N at randomisation | |
|---|---|---|---|---|
| Active | Placebo | Delta | 1:2 | |
| 90% | 72.5% | 17.5% | 79:158 = 237 | 297 |
| 90% | 75% | 15% | 102:204 = 306 | 383 |
| 90% | 77.5% | 12.5% | 138:276 = 414 | 518 |

Calculated using ADDPLAN Version 6.0.4.

Thus 400 patients in the original BI 655066 arm, provide at least 90% power for the randomized withdrawal comparison. Using a 4:1 randomisation will yield a total sample size of 500 = 400:100 for BI 655066: placebo.

Based on the outcome from trials 1311.1 and 1311.2, the PASI90 response rate at Week 16 is assumed to be at least 65% in the BI 655066 arm and approximately 5% for placebo. For sPGA clear or almost clear at Week 16, the response rate for the BI 655066 arm is assumed to be at least 80% and approximately 5% for placebo. This trial will have >99% power for comparing each BI 655066 arm to placebo on both of these endpoints.

All calculations were performed using ADDPLAN Version 6.0.4, an Aptiv Solutions Company.

c03357704-04


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 8.0 INFORMED CONSENT, DATA PROTECTION, TRIAL RECORDS

The trial will be carried out in compliance with the protocol, the ethical principles laid down in the Declaration of Helsinki, in accordance with the ICH Harmonized Tripartite Guideline for Good Clinical Practice (GCP), relevant BI Standard Operating Procedures (SOPs), the EU regulation 536/2014, the Japanese GCP regulations (Ministry of Health and Welfare Ordinance No. 28, March 27, 1997) and other relevant regulations.

The Investigator will inform the Sponsor immediately of any urgent safety measures taken to protect the trial patients against any immediate hazard, and also of any serious breaches of the protocol or of ICH GCP.

The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract. As a general rule, no trial results should be published prior to finalization of the Clinical Trial Report.

Insurance Cover: The terms and conditions of the insurance cover are made available to the investigator and the patients via documentation in the ISF.

Standard medical care (prophylactic, diagnostic and therapeutic procedures) remains in the responsibility of the treating physician of the patient.

# 8.1 TRIAL APPROVAL, PATIENT INFORMATION, AND INFORMED CONSENT

This trial will be initiated only after all required legal documentation has been reviewed and approved by the respective Institutional Review Board (IRB) / Independent Ethics Committee (IEC) and competent authority (CA) according to national and international regulations. The same applies for the implementation of changes introduced by amendments.

Prior to patient participation in the trial, written informed consent must be obtained from each patient (or the patient's legally accepted representative) according to ICH / GCP and to the regulatory and legal requirements of the participating country. Each signature must be personally dated by each signatory and the informed consent and any additional patient-information form retained by the Investigator as part of the trial records. A signed copy of the informed consent and any additional patient information must be given to each patient or the patient's legally accepted representative."

## The following paragraph pertains to Japan only:

The Investigator must give a full explanation to trial patients including the items listed below in association with the use of the patient information form, which is prepared avoiding the use of technical terms and expressions. The patient is given sufficient time to consider participation in the trial. The Investigator obtains written consent of the patient's own free will with the informed consent form after confirming that the patient understands the contents. The Investigator must sign (or place a seal on) and date the informed consent form. If a trial collaborator has given a supplementary explanation, the trial collaborator also signs (or places a seal on) and dates the informed consent.

Re-consenting may become necessary when new relevant information becomes available and should be conducted according to the sponsor's instructions.

11 Oct 2016

Trial Protocol


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 8.2 DATA QUALITY ASSURANCE

A quality assurance audit/inspection of this trial may be conducted by the Sponsor, Sponsor's designees, or by IRB / IEC or by regulatory authorities. The quality assurance auditor will have access to all medical records, the Investigator's trial-related files and correspondence, and the informed consent documentation of this clinical trial.

#### 8.3 RECORDS

Case Report Forms (CRFs) for individual patients will be provided by the sponsor via remote data capture. See <u>Section 4.1.5.2</u> for rules about emergency code breaks. For drug accountability, refer to Section 4.1.8.

#### 8.3.1 Source documents

Source documents provide evidence for the existence of the patient and substantiate the integrity of the data collected. Source documents are filed at the investigator's site.

Data reported on the CRF must be consistent with the source data or the discrepancies must be explained. The Investigator may need to request previous medical records or transfer records, depending on the trial; current medical records must also be available. For eCRFs all data must be derived from source documents.

#### 8.3.2 Direct access to source data and documents

An adaptive approach to clinical trial monitoring will be utilised. This is initiated by an assessment of the risk associated with the trial combined with identification of critical data and processes. An Integrated Quality and Risk Management Plan documents the strategies involved with the implementation of onsite, offsite and central monitoring activities in order to direct focus to the areas of greatest risk which have the most potential impact to patient safety and data quality. Trial oversight is achieved by regular review of a report of risk, which then influences any monitoring adaptations.

The Investigator / institution will permit trial-related monitoring, audits, IRB / IEC review and regulatory inspection, providing direct access to all related source data / documents. eCRF and all source documents, including progress notes and copies of laboratory and medical test results must be available at all times for review by the Sponsor's clinical trial monitor, auditor and inspection by health authorities (e.g. FDA). The Clinical Research Associate (CRA) / on site monitor and auditor may review all eCRF, and written informed consents.

## 8.3.3 Storage period of records (Applicable to Japan only)

#### Trial site(s):

The trial site(s) must retain the source documents and essential documents for a period defined by the Japanese GCP regulation and trial site's contract with the sponsor.

#### Sponsor:

The Sponsor must retain the essential documents according to the Sponsor's SOPs. When it is no longer necessary for the trial site to retain the source documents and essential documents, the Sponsor must notify the head of trial site.

c03357704-04

11 Oct 2016

**Trial Protocol** 


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 8.4 LISTEDNESS AND EXPEDITED REPORTING OF ADVERSE EVENTS

#### 8.4.1 Listedness

To fulfil the regulatory requirements for expedited safety reporting, the Sponsor evaluates whether a particular adverse event is "listed", i.e. is a known side effect of the drug or not. Therefore, a unique reference document for the evaluation of listedness needs to be provided. For the study drug BI 655066, this is the current version of the Investigator's Brochure (c01569420-06), which is provided in the ISF.

No AEs are classified as listed for matching placebo, trial design, or invasive procedures

## 8.4.2 Expedited reporting to health authorities and IEC / IRB

Expedited reporting of serious adverse events, e.g. suspected unexpected serious adverse reactions (SUSAR) to health authorities and IEC / IRB, will be done according to local regulatory requirements.

#### 8.5 STATEMENT OF CONFIDENTIALITY

Individual patient medical information obtained as a result of this trial is considered confidential and disclosure to third parties is prohibited with the exceptions noted below. Patient confidentiality will be ensured by using patient identification code numbers. Treatment data may be given to the patient's personal physician or to other appropriate medical personnel responsible for the patient's welfare. Data generated as a result of the trial need to be available for inspection on request by the participating physicians, the Sponsor's representatives, by the IRB / IEC and the regulatory authorities.

#### 8.6 END OF TRIAL

The end of the trial is defined as written in <u>Section 6.2.3</u>.

The IEC / competent authority in each participating EU member state will be notified about the end or early termination of the trial.

For Japan: When the trial is completed, the Investigator should inform the head of the trial site of the completion in writing, and the head of the trial site should promptly inform the IRB and Sponsor of the completion in writing.

#### 8.7 PROTOCOL VIOLATIONS

This Section is applicable to Japan only

The investigator should document any deviation from the protocol regardless of their reasons. Only when the protocol was not followed in order to avoid an immediate hazard to trial patients or for other medically compelling reason, the principal investigator should prepare and submit the records explaining the reasons thereof to the sponsor, and retain a copy of the records.

11 Oct 2016


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 8.8 COMPENSATION AVAILABLE TO THE PATIENT IN THE EVENT OF TRIAL RELATED INJURY

**Trial Protocol** 

This Section is applicable to Japan only In the event of health injury associated with this trial, the Sponsor is responsible for compensation based on the contract signed by the trial site. Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 9.0 REFERENCES

#### 9.1 PUBLISHED REFERENCES

- R05-2548 Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI) a simple practical measure for routine clinical use. Joint Ann Mtg of the British Association of Dermatologists and the Canadian Dermatology Association, Oxford, 6 10 Jul 1993 Clin Exp Dermatol 1994. 19:210-216.
- R08-1089 Lowes MA, Bowcock AM, Krueger JG. Pathogenesis and therapy of psoriasis. Nature 2007; 445(7130):866-873.
- R09-1299 Greenland S, Robins M. Estimation of a common effect parameter from sparse follow-up data, Biometrics 41, 55-68, 1985
- R11-1257 Nestle FO, Kaplan DH, Barker J. Mechanisms of disease: psoriasis. N Engl J Med 2009; 361(5):496-509.
- R11-1259 Menter A, Griffiths CEM. Psoriasis 2: current and future management of psoriasis. Lancet 2007; 370:272-284.
- R11-1547 Smith RLI, Warren RB, Eyre S, Ho P, Ke X, Young HS, Griffiths CEM, Worthington J. Polymorphisms in the IL-12beta and IL-23R genes are associated with psoriasis of early onset in a UK cohort. J Invest Dermatol 2008. 128:1325-1327.
- R13-3515 Woodworth T, Furst DE, Alten R, Bingham C, Yocum D, Sloan V, Tsuji W, Stevens R, Fries J, Witter J, Johnson K, Lassere M, Brooks P. Standardizing assessment and reporting of adverse effects in rheumatology clinical trials II: the Rheumatology Common Toxicity Criteria v.2.0. J Rheumatol 2007. 34(6):1401-1414.
- R14-5159 Reich K, Puig L, Paul C, Kragballe K, Luger T, Lambert J, Chimenti S, Girolomoni G, Nicolas JF, Rizova E, Brunori M, Mistry S, Bergmans P, Barker J, TRANSIT Investigators. One-year safety and efficacy of ustekinumab and results of dose adjustment after switching from inadequate methotrexate treatment: the TRANSIT randomized trial in moderate-to-severe plaque psoriasis. Br J Dermatol 2014. 170(2):435-444.
- R15-1001 Taylor W, Gladman D, Helliwell P, Marchesoni A, Mease P, Mielants H; CASPAR Study Group. Classification criteria for psoriatic arthritis: development of new criteria from a large international study. Arthritis Rheum 2006;54:2665-73.
- R15-1393 Davidovici BB, Sattar N, Joerg PC, Puig L, Emery P, Barker JN, Kerkhof P van de, Stahle M, Nestle FO, Girolomoni G, Krueger JG, Psoriasis Education and Learning Syllabus (PEARLS). Psoriasis and systemic inflammatory diseases: potential mechanistic links between skin disease and co-morbid conditions. J Invest Dermatol 2010. 130(7):1785-1796.

11 Oct 2016

Trial Protocol 

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

R15-3846 Bruce B, Fries JF. The Stanford Health Assessment Questionnaire: a review of its history, issues, progress, and documentation. J Rheumatol 2003. 30(1):167-178. The Health Assessment Ouestionnaire (HAO) and the improved HAO (formerly R15-3849 called the PROMIS HAQ) (revised June 2009). http://aramis.stanford.edu/downloads/HAQ%20Instructions%20(ARAMIS)%20 6-30-09.pdf (access date: 15 July 2015); Stanford: Stanford University School of Medicine, Division of Immunology & Rheumatology 2009 R15-5200 Langley RGB, Feldman SR, Nyirady J, Kerkhof P van de, Papavassilis C. The 5point Investigator's Global Assessment (IGA) scale: a modified tool for evaluating plaque psoriasis severity in clinical trials. J Dermatol Treat 2015. 26(1):23-31. R15-5488 Khader SA, Pearl JE, Sakamoto K, Gilmartin L, Bell GK, Jelley-Gibbs DM, et al. IL-23 compensates for the absence of IL-12p70 and is essential for the IL-17 response during tuberculosis but is dispensable for protection and antigenspecific IFN-v responses if IL-12p70 is available. J of Immunol 2005; 175:788-795. R15-5495 O'Garra A, Redford PS, McNab FW, Bloom CI, Wilkinson RJ, Berry MPR. The immune response in tuberculosis. Annu Rev Immunol 2013; 31:475-527. R15-5497 Tsai TF, Blauvelt A, Gong Y, Huang J, Fox T. Secukinumab treatment shows no evidence for reactivation of previous or latent TB infection in subjects with psoriasis: A pooled phase 3 safety analysis. J Am Acad Dermatol 2015; 607. R16-2653 Tuong W, Armstrong AW. Scalp Psoriasis: Clinical Features and Assessment, In: Adebajo A, Boehncke WH, Gladman DD, Mease PJ, editors. Psoriatic Arthritis and Psoriasis: Pathology and Clinical Aspects. Cham: Springer, 139 – 141 (2016) R16-2654 Rich P, Scher RK. Nail Psoriasis Severity Index: A useful tool evaluation of nail psoriasis. J AM Acad Dermatol 49 (2), 206 – 212 (2003) R96-3541 Fredriksson T, Pettersson U. Severe psoriasis - oral therapy with a new retinoid. Dermatologica 1978; 157:238-244.

#### 9.2 UNPUBLISHED REFERENCES

c01569420-06 Investigator's Brochure BI 655066, Psoriasis, Crohn's Disease, Ankylosing Spondylitis, Asthma, Psoriatic Arthritis 1311.P1/1311.P2/1311.P3/1311.P4/1311.P5

c03272682-01 Summary report of interim analysis at Week 48, Trial 1311.2. 05 May 2015

Trial Protocol


11 Oct 2016

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

c02434648-01 Dorleacq, N., Steimle-Goerttler, C., Bai, X., Joseph, D. Safety, tolerability, efficacy, pharmacokinetics, and pharmacodynamics of single rising i.v. (Stage 1) and s.c. (Stage 2) doses of BI 655066 in male and female patients with moderate to severe psoriasis (randomised, double-blind, placebo controlled within dose groups). Clinical Trial Report.


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 10 APPENDICES

### 10.1 PASI DEFINITIONS AND USE

The PASI is an established measure of clinical efficacy for psoriasis medications. (R96-3541) The PASI is a tool that provides a numeric scoring for patients overall psoriasis disease state, ranging from 0 to 72. It is a linear combination of percent of surface area of skin that is affected and the severity of erythema, infiltration, and desquamation over four body regions.

The endpoints used are based on the percent reduction from baseline, generally summarized as a dichotomous outcome based on achieving over an X% reduction (or  $PASI_X$ ), where X is 50, 75, 90 and 100.

To calculate the PASI, the four main body areas are assessed: **head (h), trunk (t), upper extremities (u) and lower extremities (l).** These correspond to 10, 30, 20 and 40% of the total body area respectively.

The **area of psoriatic involvement** of these four areas (Ah, At, Au, and Al) is given a numerical value: 0 = no involvement, 1 = <10%, 2 = 10 to <30%, 3 = 30 to <50%, 4 = 50 to <70%, 5 = 70 to <90%, and 6 = 90 to 100% involvement.

The signs of severity, erythema (E), infiltration (I) and desquamation (D) of lesions are assessed using a numeric scale 0-4 where 0 is a complete lack of cutaneous involvement and 4 is the severest possible involvement; scores are made independently for each of the areas, h, t, u and l and represents a composite score for each area. An illustration of judging erythema follows: 0 = no erythema, 1 = slight erythema, 2 = moderate erythema, 3 = striking erythema, and 4 = exceptionally striking erythema.

The PASI score is calculated according to the following formula:

PASI = 0.1(Eh + Ih + Dh)Ah + 0.3(Et + It + Dt)At + 0.2(Eu + Iu + Du)Au + 0.4(El + Il + Dl)Al


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 10.2 STATIC PHYSICIAN GLOBAL ASSESSMENT (SPGA)

The sPGA is a 5 point score ranging from 0 to 4, based on the physician's assessment of the average thickness, erythema, and scaling of all psoriatic lesions (R15-5200).

The assessment is considered "static", which refers to the patients disease state at the time of the assessments, without comparison to any of the patient's previous disease states, whether at Baseline or at a previous visit.

A lower score indicates less body coverage, with 0 being clear and 1 being almost clear.

# Erythema

- 0 Normal (post-inflammatory hyper/hypopigmentation may be present)
- 1 Faint, diffuse pink or slight red coloration
- 2 Mild (light red coloration)
- 3 Definite red coloration (Dull to bright red)
- 4 Bright to Deep red coloration of lesions

# Induration (plaque elevation)

- 0 None
- 1 Just detectable (slight elevation above normal skin)
- 2 Mild thickening (slight but definite elevation, typically edges are indistinct or sloped)
- 3 Clearly distinguishable to moderate thickening (marked definite elevation with rough or sloped edges)
- 4 Severe thickening with hard edges (marked elevation typically with hard or sharp edges)

# Scaling

- 0 No scaling
- 1 Minimal focal scaling (surface dryness with some desquamation)
- 2 Predominately fine scaling (fine scale partially or mostly covering lesions)
- 3 Moderate scaling (coarser scale covering most or all of the lesions)
- 4 Severe /coarse scaling covering almost all or all lesions (coarse, non-tenacious scale predominates)

### **Scoring:**

Clear 0 = 0 for all three Almost clear 1 = mean > 0, <1.5Mild 2 = mean > = 1.5, <2.5Moderate 3 = mean > = 2.5, <3.5Severe 4 = mean > = 3.5 Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# sPGA Rating Scale for Overall Psoriatic Disease

| Score | Short description | Detailed description |
|---|---|---|
| 0 | clear | No signs of psoriasis. Post-inflammatory hyper/hypopigmentation may be present |
| 1 | Almost clear | Normal to pink coloration; Just detectable (possible slight elevation above normal skin) No to minimal focal scaling |
| 2 | mild | Pink to light red coloration Mild thickening (slight but definite elevation, typically edges are indistinct or sloped) Predominantly fine scaling |
| 3 | moderate | Dull to bright red coloration Clearly distinguishable to moderate thickening Moderate scaling |
| 4 | severe | Bright to deep dark red coloration; Severe thickening with hard edges Severe coarse scaling covering almost all or all lesions |

The scale used was static, i.e., it referred exclusively to the patient's disease state at the time of the assessments, without comparison to any of the patient's previous disease states, whether at Baseline or at a previous visit.

### **Trial Protocol**


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 10.3 NAPSI – NAIL PSORIASIS SEVERITY INDEX

The NAPSI assesses how much of the fingernail is affected with psoriasis with scores ranging from 0 to 80. (R16-2654)

If a patient has nail psoriasis, the physician will assess the nail psoriasis at each protocol defined time point. Fingers (5) on each hand will be individually examined for two distinct assessments and are graded as follows:

### Nail Matrix Assessment:

- 0 = None
- 1 = present in 1 quadrant of nail
- 2 = present in 2 quadrants of nail
- 3 = present in 3 quadrants of nail
- 4 = present in 4 quadrants of nail

# Nail Bed Assessment:

- 0 = None
- 1 = present in 1 quadrant of nail
- 2 = present in 2 quadrants of nail
- 3 = present in 3 quadrants of nail
- 4 = present in 4 quadrants of nail

The sum of the scores will be added resulting a range of 0 to 80. If an individual finger assessment is missing (not done), the average of the remaining measured digits will be imputed and added to the sum. If < 50% of the finger assessments are missing the imputation will be performed. If more than 50% of the assessments are missing then the sum of the scores will be left as missing.


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 10.4 PPASI – PALMOPLANTAR PSORIASIS SEVERITY INDEX

The PPASI provides a numeric scoring for psoriasis affecting the hands and feet with scores ranging from 0 to 72. It is a linear combination of percent of surface area of hands and feet that are affected and the severity of erythema, induration, and desquamation.

If a patient has palmoplantar psoriasis, the physician will assess the psoriasis at each protocol defined time point. Both palms and soles on each hand and foot will be individually assessed for erythema, induration, desquamation and percentage of area affected as follows:

Erythema, Induration and Desquamation:

0 = None

1 = Slight

2 = Moderate

3 = Severe

4 = Very Severe

Percent of Palm and Sole Area Covered:

0 = Clear

1 = < 10%

2 = 10-29%

3 = 30-49%

4 = 50-69%

5= 70-89%

6= 90-100%

The PPASI is a composite score and will be computed for each palm and sole, left and right and is derived from the sum of the scores for erythema (E), induration (I) and desquamation (D) multiplied by the score recorded for the extent of palm and sole area involved. PPASI is calculated as follows: (sum of scores for E+I+D)\*Area \*0.2(location: right palm) + (sum of scores for E+I+D)\*Area \*0.2(location: left palm) + (sum of scores for E+I+D)\*Area \*0.3(location: right sole) + (sum of scores for E+I+D)\*Area \*0.3(location: left sole). The range is 0 to 72.

### **Trial Protocol**


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 10.5 PSORIASIS SCALP SEVERITY INDEX (PSSI)

If a patient has scalp psoriasis, the physician will assess the erythema (redness), induration (hardness), desquamation (shedding of skin) and percent of scalp covered at each protocol defined time point. (R16-2653).

Erythema, Induration and Desquamation:

- 0 = None
- 1 = Slight
- 2 = Moderate
- 3 = Severe
- 4 = Very Severe

# Percent of Scalp Covered:

- 1 = < 10%
- 2 = 10-29%
- 3 = 30-49%
- 4 = 50-69%
- 5 = 70-89%
- 6 = 90-100%

The PSSI is a composite score derived from the sum of the scores for erythema, induration and desquamation multiplied by the score recorded for the extent of scalp area involved. The range is 0 to 72.

c03357704-04


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 10.6 DIAGNOSIS AND ASSESSMENTS FOR PATIENTS WITH PSORIATIC ARTHRITIS (AT SELECTED SITES ONLY)

At Visit 1 <u>at selected study sites</u>, patients with a positive history of PsA or suspected to have PsA will be further evaluated for PsA diagnosis based on CASPAR (Classification of Psoriatic Arthritis) criteria (R15-1001).

To be classified has having PsA, a patient must have inflammatory articular disease (joint, spine, or entheseal) with at least 3 points total from the 5 categories in Table 10.6: 1, All trial participants will have 2 points assigned due to evidence of current psoriasis per trial entry criteria and will require at least one additional point for diagnosis of PsA.

Table 10.6:1 CASPAR criteria

| Category | Point assignment |
|---|---|
| Evidence of current psoriasis, a personal history of psoriasis, or a family history of psoriasis | 2 points |
| Typical psoriatic nail dystrophy, including onycholysis, pitting, or hyperkeratosis observed on current physical examination | 1 point |
| A negative test result for rheumatoid factor by any method except latex | 1 point |
| Either current dactylitis, defined as swelling of an entire digit, or a history of dactylitis recorded by a rheumatologist | 1 point |
| Radiographic evidence of juxta-articular new bone formation appearing as ill-defined ossification near joint margins (but excluding osteophyte formation) on plain radiographs of the hand or foot | 1 point |

If a diagnosis of PsA is confirmed by CASPAR and the patient meets all study entry criteria for participation, the following will be performed at Visit 2.

- HAQ-DI (see Appendix 10.7.2)
- Pain VAS (see <u>Appendix 10.7.3</u>)
- Patient global assessment VAS (see Appendix 10.7.4)
- Tender or Swollen joint counts (TJC/SJC) on 28 joints (refer to <u>Table 10.6: 2</u>)
- Entry of data for calculation of DAS28 on electronic device (Refer to Appendix 10.6.1)

During the treatment period and EOO the following will continue to be performed at the visits noted in the Flow Charts if the TJC/SJC is  $\geq 3$  at Visit 2.

- HAQ-DI (see Appendix 10.7.2)
- Pain VAS (see Appendix 10.7.3)
- Patient global assessment VAS (see Appendix 10.7.4)
- Tender or Swollen joint counts (TJC/SJC) on 28 joints (refer to Table 10.6: 2)
- Entry of data for calculation of DAS28 on electronic device (Refer to Appendix 10.6.1)

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies Table 10.6:2 Tender or Swollen Joint Count (28)

| Joint | Right | | Left | |
|------------------|--------|---------|--------|---------|
| | Tender | Swollen | Tender | Swollen |
| Shoulder | | | | |
| Elbow | | | | |
| Wrist | | | | |
| MCP1 | | | | |
| MCP2 | | | | |
| MCP3 | | | | |
| MCP4 | | | | |
| MCP5 | | | | |
| IP of the thumb | | | | |
| PIP of fingers 2 | | | | |
| PIP of fingers 3 | | | | |
| PIP of fingers 4 | | | | |
| PIP of fingers 5 | | | | |
| Knee | | | | |

Metacarpal-phalangeal joints (MCP); Interphalangeal joints (IP); Proximal interphalangeal joints (PIP)

Tenderness and swelling will be evaluated as "0" absent or "1" present.

# 10.6.1 Disease Activity Score in 28 Joints (DAS 28)

DAS28, which stands for "disease activity score," is a modified version of the original DAS. DAS28 will be calculated using a formula that includes the number of tender joints and swollen joints (28 joints), CRP (C-reactive protein) and a patient self-assessment (patient global health-VAS).

DAS 28 will be calculated using the following formula from the electronic device where the VAS pertains to the patient's global assessment of disease VAS:

• DAS28= $0.56*\sqrt{\text{ (tender joint count)}} + 0.28*\sqrt{\text{ (swollen joint count)}} + 0.36*\text{Ln(CRP+1)} + 0.014* (patient global assessment VAS) + 0.96$ 

For the DAS 28 calculation, the CRP value from laboratory report of current visit will be entered on the electronic device. Data from swollen and tender joint count (28 joints) and the patient global assessment VAS will have already been recorded on the electronic device.


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 10.7 HEALTH OUTCOMES/QUALITY OF LIFE

# 10.7.1 Dermatology Life Quality Index

The DLQI is a patient-administered, ten-question, quality of life questionnaire that covers six domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment (R05-2548). The DLQI has a one-week recall period. Response categories include "not relevant" (score of 0), "not at all" (score of 0), "a little" (score of 1), "a lot" (score of 2) and "very much" (score of 3). Question 7 is a "yes"/ "no" question where "yes" is scored as 3.

The DLQI will be self-administered by the patient at visits indicated in the flowchart.

The DLQI will be analysed under six headings as follows (R05-2548):

| Domain | Question Number | Score |
|------------------------|-------------------|-----------------|
| Symptoms and feelings | Questions 1 and 2 | Score maximum 6 |
| Daily activities | Questions 3 and 4 | Score maximum 6 |
| Leisure | Questions 5 and 6 | Score maximum 6 |
| Work and school | Question 7 | Score maximum 3 |
| Personal relationships | Questions 8 and 9 | Score maximum 6 |
| Treatment | Question 10 | Score maximum 3 |

DLQI total score is calculated by summing the scores of each question resulting in a range of 0 to 30 where 0-1 = no effect on patient's life, 2-5 = small effect, 6-10 = moderate effect, 11-20 = very large effect, and 21-30 = extremely large effect on patient's life. The higher the score, the more the quality of life is impaired. If the answer to one question in a domain is missing, that domain is treated as missing. If 2 or more questions are left unanswered (missing), DLQI total score is treated as missing. A 5-point change from baseline is considered a clinically important difference.

**Trial Protocol** 


c03357704-04 Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies DERMATOLOGY LIFE QUALITY INDEX DLQI Hospital No: Date: Name: Score: Address: Diagnosis: The aim of this questionnaire is to measure how much your skin problem has affected your life OVER THE LAST WEEK. Please tick one box for each question. Over the last week, how itchy, sore, Very much painful or stinging has your skin A lot been? A little Not at all Over the last week, how embarrassed Very much or self conscious have you been because A lot A little of your skin? Not at all Over the last week, how much has your Very much skin interfered with you going A lot A little shopping or looking after your home or garden? Not at all Not relevant Over the last week, how much has your Very much skin influenced the clothes A lot you wear? A little Not at all Not relevant Over the last week, how much has your 5. Very much skin affected any social or A lot leisure activities? A little Not at all Not relevant 6. Over the last week, how much has your Very much skin made it difficult for A lot you to do any sport? A little Not at all Not relevant Over the last week, has your skin prevented Yes you from working or studying? Not relevant If "No", over the last week how much has A lot A little your skin been a problem at work or studying? Not at all Over the last week, how much has your Very much skin created problems with your A lot partner or any of your close friends A little or relatives? Not at all Not relevant Over the last week, how much has your Very much skin caused any sexual A lot difficulties? A little Not at all Not relevant Over the last week, how much of a Very much problem has the treatment for your A lot skin been, for example by making A little your home messy, or by taking up time? Not at all Not relevant Please check you have answered EVERY question. Thank you. SAY Finlay, GK Khan, April 1992 www.dermatology.org.uk, this must not be copied without the permission of the authors

11 Oct 2016

57704-04 Trial Protocol 

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 10.7.2 Health Assessment Questionnaire Disability Index (HAQ-DI)

The HAQ-DI will be self-administered by the patient [for psoriatic arthritis patients at selected sites] at visits indicated in the flowchart.

The HAQ-DI is a twenty-item patient reported outcome instrument that assesses current physical function/ disability. The HAQ-DI covers eight categories (dressing and grooming, hygiene, arising, reach, eating, grip, walking and common daily activities). There are four response options, ranging from 0 (no difficulty) to 3 (unable to do). HAQ-DI score is reported as a mean score between 0 and 3 by dividing the total score by the number of items answered (R15-3849).

The HAQ-DI has been the most-widely used instrument to assess physical function clinical trials of treatments for rheumatoid and psoriatic arthritis and has extensive evidence of its validity and other psychometric properties in this context (R15-3846).

11 Oct 2016

# **Trial Protocol**


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| HEALTH ASSESSMENT QUESTIONNAIRE | | | | | |
|---|---|---|---|---|---|
| Name Dat | te | | | | PATKEY#QUESTDAT |
| In this section we are interested in learning how your illness affect add any comments on the back of this page. | s your ability to | o function in d | laily <mark>life. Pleas</mark> | e feel free to | HAQADMIN |
| Please check the response which best describes your usual a | abilities OVER | THE PAST | WEEK: | | QUESTYPE |
| DRESSING & GROOMING Are you able to: | Without<br>ANY<br><u>Difficulty</u> | With<br>SOME<br><u>Difficulty</u> | With<br>MUCH<br><u>Difficulty</u> | UNABLE<br>To Do | PMSVISRASTUDYQUESTNUM |
| <ul> <li>Dress yourself, including tying shoelaces and doing<br/>buttons?</li> </ul> | 3 <del></del> | 18 | <del></del> | | |
| - Shampoo your hair? | <del></del> | - | <del>2</del> 2 | <del>2 - 2</del> | DRESSNEW |
| ARISING | | | | | |
| Are you able to: | | | | | |
| - Stand up from a straight chair? | | | | | |
| - Get in and out of bed? | | | | | RISENEW |
| EATING | | | | | |
| Are you able to: | | | | | _ |
| - Cut your meat? | | | | | |
| - Lift a full cup or glass to your mouth? | | | | | |
| - Open a new milk carton? | | | | | EATNEW |
| WALKING | | | | | |
| Are you able to: | | | | | |
| - Walk outdoors on flat ground? | | | | | |
| - Climb up five steps? | | | | | WALKNEW |
| Please check any AIDS OR DEVICES that you usually use for | | | | | - |
| Cane Devices used long-handled s | | | pper pull, | | |
| Walker Built up or spe | cial utensils | | | | |
| Crutches Special or buil | | | | | |
| Wheelchair Other (Specify | r: | | _) | | DRSGASST |
| | | | | | RISEASST |
| Please check any categories for which you usually need HEL | P FROM ANO | THER PERS | ON: | | |
| Dressing and Grooming Eating | | ON COLUMN TWO IS NOT THE OWNER. | occupility | | EATASST |
| Arising Walking | | | | | WALKASST |

### 11 Oct 2016

### **Trial Protocol**


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Please check the response which best describes your usual abilities OVER THE PAST WEEK: Without With With UNABLE ANY SOME MUCH To Do **Difficulty** <u>Difficulty</u> **Difficulty HYGIENE** Are you able to: - Wash and dry your body? - Take a tub bath? - Get on and off the toilet? HYGNNEW\_ REACH Are you able to: - Reach and get down a 5 pound object (such as a bag of sugar) from just above your head? - Bend down to pick up clothing from the floor? REACHNEW\_ **GRIP** Are you able to: - Open car doors? - Open jars which have been previously opened? GRIPNEW - Turn faucets on and off? ACTIVITIES Are you able to: - Run errands and shop? - Get in and out of a car? ACTIVNEW\_ - Do chores such as vacuuming or yardwork? Please check any AIDS OR DEVICES that you usually use for any of these activities: Raised toilet seat \_\_\_\_Bathtub bar Bathtub seat Long-handled appliances for reach Jar opener (for jars Long-handled appliances in bathroom previously opened) \_\_Other (Specify: \_\_ Please check any categories for which you usually need HELP FROM ANOTHER PERSON: **HYGNASST** Hygiene Gripping and opening things RCHASST Reach Errands and chores GRIPASST\_

ACTVASST\_

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### **10.7.3** Pain VAS

The Pain VAS will be self-administered by the patient [for psoriatic arthritis patients at selected sites] at visits indicated in the flowchart.

The patient's assessment of pain will be performed using a horizontal 15cm visual analog scale (VAS), ranging from 0 (no pain) to 100 (severe pain) after the question:

"How much pain have you had because of your psoriatic arthritis in the past week? Place a vertical ( | ) mark on the line to indicate the severity of the pain."

# 10.7.4 Patient global assessment VAS

The patient global assessment VAS will be self-administered by the patient [for psoriatic arthritis patients at selected sites] at visits indicated in the flowchart.

The patient's global assessment of disease activity will be performed using a horizontal 15cm VAS, ranging from 0 (very well) to 100 (very poor) after the question:

"Considering all the ways your psoriatic arthritis affects you, how would you rate the way you felt over the past week? Place a vertical ( ) mark on the line to indicate how you felt."

**Trial Protocol** 


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 11. DESCRIPTION OF GLOBAL AMENDMENTS

| Number of global amendment | | 1.0 |
|---|---|---|
| Date of CTP revision | | 11-Mar-2016 |
| EudraCT number | | 2014-005102-38 |
| BI Trial number | | 1311.4 |
| BI Investigational Product(s) | | BI 655066 |
| Title of protocol | | BI 655066 (risankizumab) versus placebo In a |
| | | Multicenter randomized double-blind study in patients with Moderate to severe chronic plaque psoriasis evaluating the efficacy and safety with randomized withdrawal and re-treatment (IMMhance) |
| To be implemented only after | X | |
| approval of the IRB / IEC / | | |
| Competent Authorities | | |
| To be implemented immediately in order to eliminate hazard – IRB / IEC / Competent Authority to be notified of change with request for approval | | |
| Can be implemented without | | |
| IRB / IEC / Competent | | |
| Authority approval as changes | | |
| involve logistical or | | |
| administrative aspects only | | |
| Section to be changed | | Flow Chart 1 |
| Description of Change | | <ol> <li>Added Infection Testing (TB) to Screening.</li> <li>Footnote #23 added for clarification to TB.</li> </ol> |
| | | 3.ADA sampling added to Week 4 4. Footnote #5, Visit 28 corrected to Week 28 5. Footnote #17, Visit 32 and Visit 70 corrected to Week 32 and Week 70 6.Text regarding hypersensitivity removed from Footnote #13 and placed accordingly in a new footnote #24 7. Line item "biologic therapy history" changed to "psoriasis therapy history 8. Footnote #22 was re-worded |

| c03357704-04 | Trial Protocol |
|---|---|
| Proprietary confidential information © 2016 | Boehringer Ingelheim International GmbH or one or more of its affiliated companies |
| | 9. % BSA involvement added as a line item |
| Rationale for change | 1.Request from Health Authorities 2. Request from Health Authorities 3. Request from Health Authorities 4. Error in original CTP 5. Error in original CTP 6. Clarification 7. Clarification 8. Clarification 9. % BSA is collected on the electronic device at screening and prior to randomization as an inclusion criteria |
| Section To be changed | All Flow Charts |
| Description of change | 1. Footnote #6 The criterion for missing more than 1 study |
| | treatment was removed from the completer definition for entry into the OLE study. |
| | "Patients who have completed the study (which is defined as patients completing the EOO visit within the specified window per the flow charts.) and who also meet the eligibility criteria will be offered to roll over into an open label extension (OLE) trial. |
| | 2. Footnote #7- PK and ADA samples are to be taken within 60 minutes before the subcutaneous injection 3. Footnote #3 Re-written as well as DLQI removed from flow chart 2 and 3 footnote 3 |
| Rationale for change | 1. Clarification |
| | <ul><li>2. Clarification</li><li>3. DLQI not needed for flow Chart #2 and Flow Chart #3. Also footnote as originally written was redundant</li></ul> |
| Section to be changed | Flow Charts 2 and 3 (Footnote #10) |
| Description of change | Vital Status information: patients must follow their current flow chart for 'planned EOO'') |
| Rational for change | Clarification for relapsed and re-treated patients with respect to Vital Status as they follow Flow |

| c03357704-04 | Trial Protocol 6 Boehringer Ingelheim International GmbH or one or more of its affiliated companies |
|---|---|
| Proprietary confidential information © 2016 | Charts 2 and 3 which do not have an EOO at 104 weeks. |
| Section to be changed | Flow Chart #2 and Flow Chart #3 |
| Description of change | Removed DLQI from Footnote #3 |
| Rationale for change | Error in original CTP footnote |
| Section to be changed | Section 2.3-Benefit Risk Assessment |
| Description of change | Provided justification for not treating latent TB |
| Rationale for change | Due to update of Exclusion #6 for TB |
| Section to be changed | Section 3.1.2-Data Monitoring |
| Description of change | Clarification on how efficacy data will be used upon submission to the DMC as well as additional information on unblinding |
| Rationale for change | Clarification |
| Section to be changed | Section 3.1.3, MACE Adjudication Committee |
| Description of change | Added "thrombotic events" |
| Rationale for change | Clarification |
| Section to be changed | Section 3.3.3- Exclusion Criteria #6 |
| Description of change | Updated exclusion criteria to clarify latent TB and treatment for TB. "Patients with a positive test result may participate in the study if further work up (according to local practice/guidelines) establishes conclusively that the patient has no evidence of active tuberculosis. If presence of latent tuberculosis is established, patients who are at low risk of reactivation, defined by local guidelines and investigator judgment, do not need to be treated with prophylactic anti-tuberculosis prior to or during the trial". |
| Rationale for change | Due to inclusion of TB testing at Screening |
| Section to be changed | Section 3.3.4.1, Removal of Individual Patients |
| Description of change | 1.Patients discontinuing treatment early should remain in the study |

| c03357704-04 | Trial Protocol 6 Boehringer Ingelheim International GmbH or one or more of its affiliated companies |
|---|---|
| Proprietary confidential information © 201 | 2. Updated Vital Status to clarify that EOO is the current applicable flow chart |
| Rationale for change | 1. When possible patients should continue with remaining visits |
| | 2. To clarify and distinguish relapse and re-treated patients following flow charts #2 and #3 |
| Section to be changed | Section 4.1.4, Drug assignment and administration |
| Description of change | Added additional areas and wording for subcutaneous injection "(gluteal and upper arms) as well as contralateral to PK/ADA sampling" |
| Rationale for change | Omitted from original CTP |
| Section to be changed | Table 4.2.2.1:1, restricted medications |
| Description of change | 1.Added the following medications tofacitinib (Xeljanz®), apremilast (Otezla®) |
| | 2. Removed efalizumab (Raptiva®) |
| Rational for Change | <ul><li>1.Additional medications requiring washout</li><li>2. Medication not available</li></ul> |
| Section to be changed | Section 5.1.3-Further Endpoints |
| Description of change | Added "absolute PASI of <3 at all visits collected |
| Rationale for change | Change to CTP |
| Section to be changed | Laboratory Table 5.3.3:1 |
| <b>Description of Change</b> | The requirement for TB at screening was added to the Infection Testing category and footnote #3 |
| Rationale for change | Request from Health Authorities |
| Section to be changed | Section 6.2, Details of Trial Procedures |
| Description of change | Added a paragraph for TB testing: "Patients will be tested for TB (Quantiferon or PPD) at Screening, Week 52 and EOO. Patients who test positive and are at low risk of TB reactivation, per local guidelines and investigator judgment, do not need to be treated with prophylactic antituberculosis medication and can be entered or continue in the trial". |
| Rational for change | New screening procedure and information on |

| c03357704-04 Proprietary confidential information © | Trial Protocol 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies |
|---|---|
| 1 | treatment upon testing positive. |
| Section to be changed | Section 6.2.1, Screening period |
| Description of change | The maximum of 2 visits that a patient may need for screening was deleted |
| Rationale for change | Patients may require more than 2 visits to the clinic during screening |
| Section to be changed | Section 6.2.3, Follow-up Period and Trial Completion |
| Description of change | 1.Vital status- patients must follow their current flow chart for EOO |
| | <ul><li>2. Removed criteria for missing one dose for eligibility for OLE study</li><li>3. Patients discontinuing treatment early should continue in the study</li></ul> |
| Rationale for change | 1. Clarification for relapse and re-treated patients following FC#2 and FC#3 |
| | <ul><li>2. Clarification</li><li>3. Added for Clarification</li></ul> |
| Section for change | Section 7.2 Null and Alternative Hypothesis |
| Description of change | Separated out re-randomized hypothesis from hypotheses tested on all randomized patients |
| Rationale for change | The re-randomized portion of the trial can be treated as a separate study and thus tested with its own alpha = $0.05$ . |
| Section for change | Section 7.3- Planned Analysis |
| <b>Description of change</b> | 1.Clarifying the definition of analysis sets |
| | <ol> <li>deleted wording that IPV's would be provided in TSAP and added verbiage about IPVs and PPS sensitivity analyses</li> <li>Added "The hypothesis tests as described in Section 7.2 will be repeated on the PPS or RRS-PPS populations, as appropriate".</li> </ol> |
| Rationale for change | In response to questions from Health Authorities. |
| Section for change | Section 7.4-Interim analysis |
| <b>Description of change</b> | Removal of DMC information |

357704-04 Trial Protocol 

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Rationale for change | Redundant as included in DMC section |
|---|---|
| Section for change | Section 7.5 Handling of Missing data |
| Description of change | Removed sentence that additional information may be included in TSAP and added information pertaining to the sensitivities analyses that will be done |
| Rationale for change | Provide as much information concerning primary and secondary endpoints to be pre-defined in the protocol. |
| Section to be changed | Appendix 10.6 |
| Description of change | Order of PsA assessments changed at Visit 2 |
| Rationale for change | To match order of assessments on the electronic device and due to requirement to perform joint counts last |
| Section for change | Section 1.2, Drug Profile, Listedness Section 8.4.1, and Unpublished Reference Section 9.2 |
| Description of change | Document ID for the new version of the Investigator Brochure has changed to "c01569420-06" |
| Rationale for change | Updated Document ID |
| Section for change | Published Reference Section 9.1 |
| Description of change | Three references added,R15-5488, R15-5495, R15-5497 |
| Rationale for change | Due to addition information added to Section 2.3 |
| Section for change | Pages 1,2 Title pages |
| Description of change | Added risankizumab after BI 655066 |
| Rationale for change | New name added for completeness |

357704-04 Trial Protocol 

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Number of global amendment | 2.0 |
|---|---|
| Date of CTP revision | 28-Jul-2016 |
| EudraCT number | 2014-005102-38 |
| BI Trial number | 1311.4 |
| BI Investigational Product(s) | BI 655066 (risankizumab) |
| Title of protocol | BI 655066 (risankizumab) versus placebo In a |
| | Multicenter randomized double-blind study in |
| | patients with Moderate to severe chronic plaque |
| | psoriasis evaluating the efficacy and safety with randomized withdrawal and re-treatment |
| | (IMMhance) |
| To be implemented only after | X |
| approval of the IRB / IEC / | |
| Competent Authorities | |
| To be implemented immediately | |
| in order to eliminate hazard – | |
| IRB / IEC / Competent | |
| Authority to be notified of | |
| change with request for | |
| approval | |
| Can be implemented without | |
| IRB / IEC / Competent | |
| Authority approval as changes | |
| involve logistical or | |
| administrative aspects only | |
| Section To be changed | Title Page and Synopsis |
| Description of change | Added (risankizumab) to BI investigational product |
| Description of change | on title page and to active ingredient section in |
| | Synopsis |
| Rationale for change | New name added for completeness |
| Section To be changed | Throughout document |
| Description of change | The following abbreviations are now spelled out due |
| Description of change | to first use in the text: ECG (synopsis); RDC |
| | (5.3.6.1); PPD (3.3.3); VEGF (5.5.1);ULN (5.3.6.1); |
| | GRAPPA (6.2); NRI, LOCF, MMRM (7.5); CTR |
| | (7.6); CTP (flowchart #1 footnote 6) |
| Rationale for change | Omitted from original CTP |
| Section to be changed | All Flow Charts |
| Description of Change | a. Added to footnote #6 " who have not discontinued |
| | drug prematurely" |
| | <b>b</b> . Revision to footnote #24 on FC #1, footnote #12 |
| | on FC #2 and footnote #11 on FC #3, "Patients |

Trial Protocol 

| Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies | |
|---|---|
| | should be closely monitored for signs and symptoms |
| | of hypersensitivity reactions for approximately 2 |
| | hours after the last injection at Visit 2 and for |
| | approximately one hour after the last injection at all |
| | other visits where drug is administered |
| Rationale for change | a. Additional criteria for a study completer and entry |
| | into OLE study |
| | <b>b</b> . Provide additional details of monitoring |
| | hypersensitivity with respect to injection times |
| Section To be changed | Flow Chart 1 |
| Description of change | Added to Footnote #15 |
| | "Patients that terminate trial medication early should |
| | remain in the trial and complete all remaining |
| | Treatment Period visits and, FU1 and FU2 Visits. |
| | Termination of trial medication eCRF should be |
| | completed and end of study registered as a non- |
| | completer in IRT. Refer to Section 6.2.3 for details |
| | and further instruction if patient cannot or will not |
| | continue in the trial. |
| Rationale for change | Additional clarification needed for proper procedure |
| | when a patient discontinues treatment but remains in |
| | the study |
| Section to be changed | Flow Chart #1 |
| Description of change | Added the following to Footnote #13 "(after last |
| | injection)" |
| Rationale for change | To clarify when vitals post dose are expected at |
| | Visits 2 and 3 |
| Section to be changed | Abbreviations |
| Description of change | Added the following abbreviations: aPTT, CRO, |
| | PPD, RCTC, Nab, NGAL, VEGF, TJC/SJC, |
| | GRAPPA, CRP, PPS, RBC, RRS-PPS, NRI, |
| | MMRM, AP, BUN, CK, CK-MB, eGFR, GGT, Hb, |
| | Hct, HDL, LDL, TSH, INR, RDC |
| | Abbreviation PoC corrected to PoCC |
| | Abbreviation OPU corrected to "Operative" |
| Rationale for change | Omitted from original or CTP V 2.0 |
| Section to be changed | Table of Contents |
| Description of change | Formatting update to title of sections 5.3.5.1, 5.4.2.1, |
| | 5.4.2.2, 5.5.1.2 and 7.3.7 in order to show in the table |
| D.C. L.C. | of contents |
| Rationale for change | Formatting error in original CTP |
| Section to be changed | Section 3.1- Overall Trial Design and Plan |
| Description of change | Section re-written and Figure 3.1:1 was replaced with |
| | new trial design. In summary: At the Week 28 |
| | visit, all patients will be assessed for responsiveness. |
| | Patients not meeting the protocol defined response |
| | criteria (sPGA is $\geq 2$ ) (Week 28 non-responders), |
| | will receive open label BI 655066 150 mg from |

**Trial Protocol** 


| Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies | |
|---|---|
| | Week 28 until the end of the treatment period (Week |
| | 88), regardless of originally randomized treatment |
| | arm. Patients who meet the protocol defined |
| | responder criteria (sPGA of 0 or 1) (Week 28 |
| | responders), will continue to receive blinded drug. In |
| | Arm 1, patients will be re-randomized; in Arm 2, |
| | they will continue to receive blinded BI655066 |
| | treatment as described in Section 7.6. |
| | Starting with Week 32, Week 28 responders will |
| | have their sPGA assessed for protocol defined |
| | relapse (sPGA of $\geq$ 3). |
| Rationale for change | This change is to be implemented to ensure that no |
| g | bias is introduced by knowing patients' original |
| | treatment assignment after the Week 28 visit |
| Section to be changed | 3.1 Overall Trial Design and Plan |
| Description of change | "a primary endpoint analysis will be conducted <u>after</u> |
| l line of the second of the se | the last patient has been in the study for 52 weeks (or |
| | discontinued)". The previous wording was "when |
| | the last patient completes the Week 52 visit. |
| Rationale for change | To incorporate the possibility that patients may |
| | discontinue from the study prior to Week 52. |
| Section to be changed | Section 3.1.1 Administrative structure of the trial |
| Description of change | Operating unit changed to Operative Unit |
| Rationale for change | Protocol template error |
| Section to be changed | 3.3.4.1 Removal of individual patients |
| Description of change | The word "necessarily" was added to: |
| Description of change | "Discontinuation of study medication should not |
| | necessarily lead to withdrawal from the study". |
| Rationale for change | Clarification as patients that discontinue study |
| Rationale for change | medication should complete all study visits and |
| | procedures as initially planned, if possible |
| Section to be changed | 3.3.4.2 |
| Description of change | Bullet #2 re-written to "Emergence of any |
| Description of change | efficacy/safety information that could significantly |
| | affect continuation of the trial, or any other |
| | administrative reasons, i.e. problems with availability |
| | of the study medication, discontinuation of |
| | development of BI 655066 Original Bullet #3 removed "Emergence of any |
| | Original Bullet #3 removed "Emergence of any efficacy/safety information invalidating the earlier |
| | positive benefit-risk-assessment that could |
| | significantly affect the continuation of the trial |
| | (including those based on DMC recommendation) |
| | (mending mose based on DIVIC recommendation) |
| Rationale for change | Error in original CTP |
| Section to be changed | Section 4.1.2 Methods of assigning patients to |
| Section to be changed | treatment groups |
| Description of change | Section re-written according to new study design to |
| Description of change | section to written according to new study design to |

| c03357704-04 | Trial Protocol 116 Boehringer Ingelheim International GmbH or one or more of its affiliated companies |
|---|---|
| Proprietary confidential information © 20 | be consistent with section 3.1 |
| Rationale for change | Design change |
| Section to be changed | Section 4.1.3 Selection of doses in the trial |
| <b>Description of change</b> | 650666 changed to 655066 |
| Rationale for change | Error in original CTP |
| Section to be changed | 4.1.4 Drug assignment and administration of doses for each patient |
| Description of change | <ul> <li>a. Added that the 2 injections need to be administered within approximately 5 minutes.</li> <li>b. Added that the IMP time in the eCRF is the time of injection # 1.</li> <li>c. Added the underlined words to the sentence; "Patients should be closely monitored for signs and symptoms of hypersensitivity reactions for approximately 2 hours after the last injection at Visit 2 and for approximately one hour after the last injection at all other visits where drug is administered.</li> <li>d. Deleted: (contra-lateral to that used for PK/PD samples) from sentence "BI 655066 and/or matching placebo will be administered as a subcutaneous injection in the abdomen, thighs, gluteal regions, or upper arms".</li> </ul> |
| Rationale for change | <ul> <li>a,b. Provide clarity and further details on timing of injections and eCRF completion</li> <li>c.To specify timing of monitoring hypersensitivity with respect to injection times.</li> <li>d. not required as PK samples are only taken predose (trough)</li> </ul> |
| Section to be changed | 4.1.5.1 Blinding |
| Description of change | Section re-written according to new study design to be consistent with section 3.1, clarifying the criteria for receiving open label drug and knowing future treatments are BI 655066. |
| Rationale for change | New study design as noted in section 3.1 |
| Section to be changed | 4.2.2.3 Restrictions regarding women of childbearing potential |
| Description of change | Deleted reference to Section 3.3.3, and corrected to 3.3.2 |
| Rationale for change | Error in original protocol |
| Section to be changed | 5.1.3 Further endpoints |
| <b>Description of change</b> | Text added "The above endpoints will be analyzed, |

357704-04 Trial Protocol 

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| where appropriate, for re-randomized subjects after receiving open-label study drug for retreatment (Flow Chart 2 and 3)". Rationale for change To clarify that these endpoints will also be analyzed among retreatment patients at visits collected. Section to be changed Description of change The underlined wording was added to the following sentences. "In addition at Visit 2 and Visit 3 vital sign evaluations will be taken at approximately 5 minutes post-dose (5 minutes after last injection) and approximately 60 minutes post-dose (60 minutes after last injection) and approximately 60 minutes post-dose (60 minutes after last injection) and approximately 2 hours after the last injection at Visit 2 and for approximately one hour after the last injection at all other visits where drug is administered Rationale for change To specify timing of vitals relative to injection times and also timing of monitoring hypersensitivity with respect to injection times. Section to be changed Description of change Added absolute count to differential Added "activated to aPTT Deleted "Creatinine" from urinalysis stix Added "calculated" to LDL Deleted "Creatinine" from urinalysis stix Added "creatinine" rom urinalysis stix Added "creatinine" rom urinalysis Added Albumin/creatinine ratio to Urinalysis Rationale for change Section to be changed 6.2 Details of Trial Procedures At Selected Visits Description of change Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Rationale for change Omitted from original CTP Section to be changed Section to be changed Omitted from original CTP Section to be changed Section to Rationale patients) |
|---|
| Rationale for change Bection to be changed Description of change The underlined wording was added to the following sentences. "In addition at Visit 2 and Visit 3 vital sign evaluations will be taken at approximately 5 minutes post-dose (5 minutes after last injection) and approximately 60 minutes post-dose (60 minutes after last injection). "Patients should be closely monitored for signs and symptoms of hypersensitivity reactions for approximately 2 hours after the last injection at all other visits where drug is administered. Rationale for change To specify timing of vitals relative to injection times and also timing of monitoring hypersensitivity with respect to injection times. Section to be changed Description of change Added absolute count to differential Added "activated to aPTT Deleted "MB" from Troponin reflex Added "calculated" to LDL Deleted "creatinine" from urinalysis stix Added "creatinine" from urinalysis Added Albumin/creatinine ratio to Urinalysis Rationale for change Rationale for change Bection to be changed Captalis of Trial Procedures At Selected Visits Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Rationale for change Section to be changed Omitted from original CTP |
| Rationale for change Section to be changed Description of change To clarify that these endpoints will also be analyzed among retreatment patients at visits collected. 5.3.2 Vital Signs The underlined wording was added to the following sentences. "In addition at Visit 2 and Visit 3 vital sign evaluations will be taken at approximately 5 minutes post-dose (5 minutes after last injection) and approximately 60 minutes post-dose (60 minutes after last injection). "Patients should be closely monitored for signs and symptoms of hypersensitivity reactions for approximately 2 hours after the last injection at Visit 2 and for approximately one hour after the last injection at all other visits where drug is administered. Rationale for change To specify timing of vitals relative to injection times and also timing of monitoring hypersensitivity with respect to injection times. Section to be changed Description of change Added absolute count to differential Added "activated to aPTT Deleted "MB" from Troponin reflex Added "calculated" to LDL Deleted "creatinine" from urinalysis stix Added "creatinine" from urinalysis stix Added "creatinine" and original CTP or needed further clarification Section to be changed Description of change Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Omitted from original CTP Section to be changed Omitted from original CTP |
| among retreatment patients at visits collected. Section to be changed Description of change The underlined wording was added to the following sentences. "In addition at Visit 2 and Visit 3 vital sign evaluations will be taken at approximately 5 minutes post-dose (5 minutes after last injection) and approximately 60 minutes post-dose (60 minutes after last injection). "Patients should be closely monitored for signs and symptoms of hypersensitivity reactions for approximately 2 hours after the last injection at Visit 2 and for approximately one hour after the last injection at all other visits where drug is administered Rationale for change To specify timing of vitals relative to injection times and also timing of monitoring hypersensitivity with respect to injection times. Section to be changed Table 5.3.3:1 laboratory tests Added absolute count to differential Added "activated to aPTT Deleted "MB" from Troponin reflex Added "creatinine" from urinalysis stix Added "creatinine" from urinalysis stix Added "creatinine" from urinalysis Added Albumin/creatinine ratio to Urinalysis Rationale for change Was omitted from original CTP or needed further clarification Section to be changed Observiption of change Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Omitted from original CTP Section to be changed Omitted from original CTP Section to be changed Omitted from original CTP Section to be changed Omitted from original CTP Section to be changed Omitted from original CTP Section to be changed Omitted from original CTP |
| Section to be changed Description of change The underlined wording was added to the following sentences. "In addition at Visit 2 and Visit 3 vital sign evaluations will be taken at approximately 5 minutes post-dose (5 minutes after last injection) and approximately 60 minutes post-dose (60 minutes after last injection). "Patients should be closely monitored for signs and symptoms of hypersensitivity reactions for approximately 2 hours after the last injection at Visit 2 and for approximately one hour after the last injection at all other visits where drug is administered and also timing of monitoring hypersensitivity with respect to injection times. Section to be changed Table 5.3.3:1 laboratory tests |
| The underlined wording was added to the following sentences. "In addition at Visit 2 and Visit 3 vital sign evaluations will be taken at approximately 5 minutes post-dose (5 minutes after last injection) and approximately 60 minutes post-dose (60 minutes after last injection). "Patients should be closely monitored for signs and symptoms of hypersensitivity reactions for approximately 2 hours after the last injection at Visit 2 and for approximately 2 hours after the last injection at Visit 2 and for approximately one hour after the last injection at all other visits where drug is administered. Rationale for change To specify timing of vitals relative to injection times and also timing of monitoring hypersensitivity with respect to injection times. Section to be changed Description of change Added absolute count to differential Added "activated to aPTT Deleted "MB" from Troponin reflex Added "activated to aPTT Deleted "Creatinine" from urinalysis stix Added "creatinine" to urinalysis Added Albumin/creatinine ratio to Urinalysis Added Albumin/creatinine ratio to Urinalysis and Visits Added Albumin/creatinine ratio to Urinalysis Patients of the Creating of the CPP or needed further clarification Section to be changed Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Omitted from original CTP Section to be changed Omitted from original CTP Section to be changed Section to be changed Omitted from original CTP Section to be changed Section to be changed withdrawal period (Re-randomized patients) |
| sentences. "In addition at Visit 2 and Visit 3 vital sign evaluations will be taken at approximately 5 minutes post-dose (5 minutes after last injection) and approximately 60 minutes post-dose (60 minutes after last injection). "Patients should be closely monitored for signs and symptoms of hypersensitivity reactions for approximately 2 hours after the last injection at Visit 2 and for approximately one hour after the last injection at all other visits where drug is administered and also timing of vitals relative to injection times and also timing of monitoring hypersensitivity with respect to injection times. Section to be changed Description of change Added absolute count to differential Added "activated to aPTT Deleted "MB" from Troponin reflex Added "calculated" to LDL Deleted "creatinine" from urinalysis stix Added "creatinine" from urinalysis Added Albumin/creatinine ratio to Urinalysis Added Albumin/creatinine ratio to Urinalysis Rationale for change Was omitted from original CTP or needed further clarification Section to be changed Omitted from original CTP Section to be changed Omitted from original CTP Section to be changed Section 6.2.2, Week 28 Visit and Randomized withdrawal period (Re-randomized patients) |
| sign evaluations will be taken at approximately 5 minutes post-dose (5 minutes after last injection) and approximately 60 minutes post-dose (60 minutes after last injection). "Patients should be closely monitored for signs and symptoms of hypersensitivity reactions for approximately 2 hours after the last injection at Visit 2 and for approximately one hour after the last injection at all other visits where drug is administered Rationale for change To specify timing of vitals relative to injection times and also timing of monitoring hypersensitivity with respect to injection times. Section to be changed Description of change Added absolute count to differential Added "activated to aPTT Deleted "MB" from Troponin reflex Added "calculated" to LDL Deleted "creatinine" from urinalysis stix Added "creatinine" from urinalysis Added Albumin/creatinine ratio to Urinalysis Rationale for change Was omitted from original CTP or needed further clarification Section to be changed 6.2 Details of Trial Procedures At Selected Visits Description of change Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Omitted from original CTP Section to be changed Section 6.2.2, Week 28 Visit and Randomized withdrawal period (Re-randomized patients) |
| minutes post-dose (5 minutes after last injection) and approximately 60 minutes post-dose (60 minutes after last injection). "Patients should be closely monitored for signs and symptoms of hypersensitivity reactions for approximately 2 hours after the last injection at Visit 2 and for approximately one hour after the last injection at all other visits where drug is administered Rationale for change To specify timing of vitals relative to injection times and also timing of monitoring hypersensitivity with respect to injection times. Section to be changed Description of change Added absolute count to differential Added "activated to aPTT Deleted "MB" from Troponin reflex Added "calculated" to LDL Deleted "creatinine" from urinalysis stix Added "creatinine" from urinalysis Added Albumin/creatinine ratio to Urinalysis Rationale for change Was omitted from original CTP or needed further clarification Section to be changed 6.2 Details of Trial Procedures At Selected Visits Description of change Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Rationale for change Section to be changed Omitted from original CTP Section to be changed Section 6.2.2, Week 28 Visit and Randomized withdrawal period (Re-randomized patients) |
| approximately 60 minutes post-dose (60 minutes after last injection). "Patients should be closely monitored for signs and symptoms of hypersensitivity reactions for approximately 2 hours after the last injection at Visit 2 and for approximately one hour after the last injection at all other visits where drug is administered and also timing of vitals relative to injection times and also timing of monitoring hypersensitivity with respect to injection times. Section to be changed Description of change Added absolute count to differential Added "activated to aPTT Deleted "MB" from Troponin reflex Added "calculated" to LDL Deleted "creatinine" from urinalysis stix Added "creatinine" from urinalysis Added Albumin/creatinine ratio to Urinalysis Added Albumin/creatinine ratio to Urinalysis Pation to be changed Section to be changed Description of change Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Rationale for change Omitted from original CTP Section to be changed Omitted from original CTP Section to be changed Omitted from original CTP Section to be changed Omitted from original CTP Section to be changed Omitted from original CTP |
| Last injection]. "Patients should be closely monitored for signs and symptoms of hypersensitivity reactions for approximately 2 hours after the last injection at Visit 2 and for approximately one hour after the last injection at all other visits where drug is administered and also timing of vitals relative to injection times and also timing of monitoring hypersensitivity with respect to injection times. Section to be changed |
| for signs and symptoms of hypersensitivity reactions for approximately 2 hours after the last injection at Visit 2 and for approximately one hour after the last injection at all other visits where drug is administered and also timing of vitals relative to injection times and also timing of monitoring hypersensitivity with respect to injection times. Section to be changed Description of change Added absolute count to differential Added "activated to aPTT Deleted "MB" from Troponin reflex Added "calculated" to LDL Deleted "creatinine" from urinalysis stix Added "creatinine" from urinalysis stix Added "creatinine" to urinalysis Added Albumin/creatinine ratio to Urinalysis Rationale for change Was omitted from original CTP or needed further clarification Section to be changed 6.2 Details of Trial Procedures At Selected Visits Description of change Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Rationale for change Omitted from original CTP Section to be changed Section 6.2.2, Week 28 Visit and Randomized withdrawal period (Re-randomized patients) |
| for approximately 2 hours after the last injection at Visit 2 and for approximately one hour after the last injection at all other visits where drug is administered To specify timing of vitals relative to injection times and also timing of monitoring hypersensitivity with respect to injection times. Section to be changed Table 5.3.3:1 laboratory tests Added absolute count to differential Added "activated to aPTT Deleted "MB" from Troponin reflex Added "calculated" to LDL Deleted "creatinine" from urinalysis stix Added "creatinine" to urinalysis Added Albumin/creatinine ratio to Urinalysis Added Albumin/creatinine ratio to Urinalysis Rationale for change Was omitted from original CTP or needed further clarification Section to be changed 6.2 Details of Trial Procedures At Selected Visits Description of change Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Rationale for change Omitted from original CTP Section to be changed Section 6.2.2, Week 28 Visit and Randomized withdrawal period (Re-randomized patients) |
| Visit 2 and for approximately one hour after the last injection at all other visits where drug is administered To specify timing of vitals relative to injection times and also timing of monitoring hypersensitivity with respect to injection times. Section to be changed Table 5.3.3:1 laboratory tests Added absolute count to differential Added "activated to aPTT Deleted "MB" from Troponin reflex Added "calculated" to LDL Deleted "creatinine" from urinalysis stix Added "creatinine" from urinalysis Added Albumin/creatinine ratio to Urinalysis Rationale for change Was omitted from original CTP or needed further clarification Section to be changed 6.2 Details of Trial Procedures At Selected Visits Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Rationale for change Section to be changed Omitted from original CTP Section to be changed Section 6.2.2, Week 28 Visit and Randomized withdrawal period (Re-randomized patients) |
| Injection at all other visits where drug is administered To specify timing of vitals relative to injection times and also timing of monitoring hypersensitivity with respect to injection times. Section to be changed Table 5.3.3:1 laboratory tests |
| Rationale for change To specify timing of vitals relative to injection times and also timing of monitoring hypersensitivity with respect to injection times. Section to be changed Description of change Added absolute count to differential Added "activated to aPTT Deleted "MB" from Troponin reflex Added "calculated" to LDL Deleted "creatinine" from urinalysis stix Added "creatinine" to urinalysis Added Albumin/creatinine ratio to Urinalysis Rationale for change Was omitted from original CTP or needed further clarification Section to be changed Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Rationale for change Section to be changed Omitted from original CTP Section to be changed Section (Re-randomized patients) |
| and also timing of monitoring hypersensitivity with respect to injection times. Section to be changed Description of change Added absolute count to differential Added "activated to aPTT Deleted "MB" from Troponin reflex Added "calculated" to LDL Deleted "creatinine" from urinalysis stix Added "creatinine" to urinalysis Added Albumin/creatinine ratio to Urinalysis Rationale for change Was omitted from original CTP or needed further clarification Section to be changed 6.2 Details of Trial Procedures At Selected Visits Description of change Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Rationale for change Omitted from original CTP Section to be changed Section 6.2.2, Week 28 Visit and Randomized withdrawal period (Re-randomized patients) |
| respect to injection times. Table 5.3.3:1 laboratory tests Added absolute count to differential Added "activated to aPTT Deleted "MB" from Troponin reflex Added "calculated" to LDL Deleted "creatinine" from urinalysis stix Added "creatinine" to urinalysis Added Albumin/creatinine ratio to Urinalysis Rationale for change Was omitted from original CTP or needed further clarification Section to be changed 6.2 Details of Trial Procedures At Selected Visits Description of change Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Rationale for change Omitted from original CTP Section to be changed Section 6.2.2, Week 28 Visit and Randomized withdrawal period (Re-randomized patients) |
| Table 5.3.3:1 laboratory tests Added absolute count to differential Added "activated to aPTT Deleted "MB" from Troponin reflex Added "calculated" to LDL Deleted "creatinine" from urinalysis stix Added "creatinine" to urinalysis Added Albumin/creatinine ratio to Urinalysis Was omitted from original CTP or needed further clarification Section to be changed Description of change Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Omitted from original CTP Section to be changed Section to be changed Omitted from original CTP Section to be changed Omitted from original CTP Section to be changed Section to Be changed Omitted from original CTP Section to Be changed Section to Be changed Omitted from original CTP Section to Be changed Section to Be changed Omitted from original CTP |
| Added absolute count to differential Added "activated to aPTT Deleted "MB" from Troponin reflex Added "calculated" to LDL Deleted "creatinine" from urinalysis stix Added "creatinine" to urinalysis Added Albumin/creatinine ratio to Urinalysis Was omitted from original CTP or needed further clarification Section to be changed 6.2 Details of Trial Procedures At Selected Visits Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Omitted from original CTP Section to be changed Section to be changed Omitted from original CTP Section to be changed Section 6.2.2, Week 28 Visit and Randomized withdrawal period (Re-randomized patients) |
| Added "activated to aPTT Deleted "MB" from Troponin reflex Added "calculated" to LDL Deleted "creatinine" from urinalysis stix Added "creatinine" to urinalysis Added Albumin/creatinine ratio to Urinalysis Was omitted from original CTP or needed further clarification Section to be changed 6.2 Details of Trial Procedures At Selected Visits Description of change Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Omitted from original CTP Section to be changed Section 6.2.2, Week 28 Visit and Randomized withdrawal period (Re-randomized patients) |
| Deleted "MB" from Troponin reflex Added "calculated" to LDL Deleted "creatinine" from urinalysis stix Added "creatinine" to urinalysis Added Albumin/creatinine ratio to Urinalysis Was omitted from original CTP or needed further clarification Section to be changed 6.2 Details of Trial Procedures At Selected Visits Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Rationale for change Omitted from original CTP Section to be changed Section 6.2.2, Week 28 Visit and Randomized withdrawal period (Re-randomized patients) |
| Added "calculated" to LDL Deleted "creatinine" from urinalysis stix Added "creatinine" to urinalysis Added Albumin/creatinine ratio to Urinalysis Was omitted from original CTP or needed further clarification Section to be changed 6.2 Details of Trial Procedures At Selected Visits Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Omitted from original CTP Section to be changed Section 6.2.2, Week 28 Visit and Randomized withdrawal period (Re-randomized patients) |
| Deleted "creatinine" from urinalysis stix Added "creatinine" to urinalysis Added Albumin/creatinine ratio to Urinalysis Rationale for change Was omitted from original CTP or needed further clarification Section to be changed 6.2 Details of Trial Procedures At Selected Visits Description of change Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Rationale for change Omitted from original CTP Section to be changed Section 6.2.2, Week 28 Visit and Randomized withdrawal period (Re-randomized patients) |
| Added "creatinine" to urinalysis Added Albumin/creatinine ratio to Urinalysis Rationale for change Was omitted from original CTP or needed further clarification Section to be changed 6.2 Details of Trial Procedures At Selected Visits Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Rationale for change Omitted from original CTP Section to be changed Section 6.2.2, Week 28 Visit and Randomized withdrawal period (Re-randomized patients) |
| Added Albumin/creatinine ratio to Urinalysis Was omitted from original CTP or needed further clarification Section to be changed 6.2 Details of Trial Procedures At Selected Visits Description of change Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Omitted from original CTP Section to be changed Section 6.2.2, Week 28 Visit and Randomized withdrawal period (Re-randomized patients) |
| Rationale for change Was omitted from original CTP or needed further clarification Section to be changed 6.2 Details of Trial Procedures At Selected Visits Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Rationale for change Omitted from original CTP Section to be changed Section 6.2.2, Week 28 Visit and Randomized withdrawal period (Re-randomized patients) |
| clarification Section to be changed 6.2 Details of Trial Procedures At Selected Visits Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Rationale for change Omitted from original CTP Section to be changed Section 6.2.2, Week 28 Visit and Randomized withdrawal period (Re-randomized patients) |
| Section to be changed Description of change Added paragraph to note that efficacy questionnaires are direct data capture on an electronic device Rationale for change Omitted from original CTP Section to be changed Section 6.2.2, Week 28 Visit and Randomized withdrawal period (Re-randomized patients) |
| Description of changeAdded paragraph to note that efficacy questionnaires are direct data capture on an electronic deviceRationale for changeOmitted from original CTPSection to be changedSection 6.2.2, Week 28 Visit and Randomized withdrawal period (Re-randomized patients) |
| are direct data capture on an electronic device Rationale for change Omitted from original CTP Section to be changed Section 6.2.2, Week 28 Visit and Randomized withdrawal period (Re-randomized patients) |
| Rationale for change Omitted from original CTP Section to be changed Section 6.2.2, Week 28 Visit and Randomized withdrawal period (Re-randomized patients) |
| Section to be changed Section 6.2.2, Week 28 Visit and Randomized withdrawal period (Re-randomized patients) |
| withdrawal period (Re-randomized patients) |
| <b>Description of change</b> Wording revised due to implementation of continuing |
| blinded treatment |
| Rationale for change Design change for Week 28 |
| Section to be changed Section 6.2.2 Treatment period |
| <b>Description of change</b> Added "a maximum of" 20 visits |
| Rationale for change Clarification as patients who relapse and get retreated |
| may have less visits during treatment depending on |
| time of relapse |
| Section to be changed Section 6.2.3 Early Treatment and trial termination |
| <b>Description of change</b> Further instructions given for staying in the trial or |
| terminating from the trial when a patient ends |
| treatment early |

| c03357704-04 | Trial Protocol |
|---|---|
| | chringer Ingelheim International GmbH or one or more of its affiliated companies |
| Rationale for change | Update to original CTP |
| Section to be changed | Section 6.2.3 Successful Trial Completion |
| Description of change | Added "and who have not discontinued drug |
| Dationals for shange | prematurely" to definition of trial completion |
| Rationale for change | Clarifying definition of trial completion Section 7.1 |
| Section to be changed | 2 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 |
| Description of change | "or not collected per protocol" was added to the last sentence in first paragraph |
| Rationale for change | clarification |
| Section to be changed | Section 7.3 Planned Analyses |
| Description of change | Second to last sentence of last paragraph wording "the patients included in the Week 52 assessment of randomized withdrawal "Replaced with "affecting Week 52 efficacy of randomized withdrawal. |
| Rationale for change | To clarify that this per-protocol set will exclude patients with violations affecting their efficacy evaluation, not affecting patients in general. |
| Section to be changed | 7.3.3 Further endpoint analyses |
| Description of change | "descriptively" removed from "Further endpoints |
| | will be summarized descriptively |
| Rationale for change | "summarized" already means that descriptive/summary statistics will be provided, the word "descriptively" seems duplicated here and is removed. |
| Section to be changed | 7.4 Interim Analyses |
| Description of change | <ul> <li>a. Updated to "An analysis will be conducted after the last patient either has been in the study for 52 weeks or discontinues from study".</li> <li>b. Updated to: "hence no alpha adjustment is required at this analysis".</li> </ul> |
| Rationale for change | <ul> <li>a. To incorporate the possibility that patients may discontinue from the study prior to Week 52.</li> <li>b. To clarify that this analysis will not require type-I error rate adjustment.</li> </ul> |
| Section to be changed | 7.5 Handling of Missing Data |
| Description of change | <ul> <li>a. Added "Of note, for randomized withdrawal analyses, subjects who received retreatment will be counted as non-responders in all visits after the date of retreatment."</li> <li>b. Added "the following methods where applicable" to the end of this sentence, "Sensitivity analyses to assess the robustness of the hypothesis testing results will include":</li> </ul> |
| Rationale for change | <b>a.</b> To clarify that patients who received retreatment |
| | will be counted as non-responders, since the decision |

c03357704-04 Trial Protocol 

| Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies | |
|---|---|
| | of retreatment is due to lack of efficacy. |
| | <b>b.</b> To clarify that the listed methods for sensitivity |
| | analyses will be conducted based on data availability |
| | and method validity, because not all methods are |
| | applicable at all cases. |
| Section to be changed | 7.6 Randomisation |
| Description of change | Section re-written according to new study design to |
| | be consistent with section 3.1 |
| Rationale for change | CTP update |
| Section to be changed | Table 7.7.1 |
| Description of change | Changed PBO to "placebo" |
| Rationale for change | "placebo" used throughout CTP |
| Section to be changed | Section 9.1 Published References |
| Description of change | Added R16-2653 and R16-2654 |
| Rationale for change | Omitted from original CTP |
| Section to be changed | 10.3 NAPSI-Nail Psoriasis Severity Index |
| Description of change | Addition of Reference number R16-2654 |
| Rationale for change | Update to CTP |
| Section to be changed | 10.4 PPASI-Palmoplantar psoriasis severity index |
| Description of change | Correction of wording from "scored" to "scores" |
| Rationale for change | Correction |
| Section to be changed | 10.5 Psoriasis scalp severity index (PSSI) |
| Description of change | Addition of Reference number R16-2653 |
| Rationale for change | Omitted from original CTP |
| Section to be changed | 10.7.1 Dermatology life quality index (DLQI) |
| Description of change | Correction of response categories |
| Rationale for change | Update from original CTP |
| Section to be changed | 3.1 Overall Trial Design and Plan and 4.1.5.1 |
| | Blinding |
| Description of change | Removed wording noting that data for all patients |
| | through week 16 must be entered into the eCRF prior |
| | to the patients receiving treatment at the week 28 |
| | visit." |
| Rationale for change | As this amendment removes the blind break for week |
| | 28 responders, this is no longer a requirement and is |
| | accordingly removed from the protocol. |

| c03357704-04 Proprietary confidential information © 2016 | | | |
|---|---|---|---|
| Number of global amendment | 3. | - | ore or its armiated companies |
| Date of CTP revision | | 1-Oct-2016 | |
| EudraCT number | 20 | 2014-005102-38 | |
| BI Trial number | 13 | 1311.4 | |
| BI Investigational Product(s) | B | I 655066/ABBV-066 (risanl | kizumab) |
| Title of protocol | M<br>pa<br>ps<br>ra | I 655066 (risankizumab) ver<br>fulticenter randomized doub<br>atients with Moderate to sev<br>soriasis evaluating the effica<br>andomized withdrawal and re<br>MMhance) | ple-blind study in<br>ere chronic plaque<br>acy and safety with |
| To be implemented only after | | | |
| approval of the IRB / IEC / | | | |
| Competent Authorities | | | |
| To be implemented immediately in order to eliminate hazard – IRB / IEC / Competent Authority to be notified of change with request for | | | |
| approval Can be implemented without | X | | |
| IRB / IEC / Competent Authority approval as changes involve logistical or administrative aspects only | A | | |
| Section To be changed | T | itle page and synopsis | |
| Description of change | | he compound name was revi<br>66" to BI 655066 (risankizu | |
| Rationale for change | In ag O tra ch of ce | February 2016, AbbVie engreement with BI related to a ctober 2016, the US IND for ansitioned from BI to AbbVie was reflects that AbbVie was study in the US, as well entain study conduct respons at license agreement are listelow. | tered into a license risankizumab, and in r risankizumab ie. This protocol vill now be the Sponsor ll as the modifications to ibilities as a result of |
| Section To be changed | Se | ection 3.1.1 | |
| Description of change | to | Changed sponsor from Boe AbbVie in the USA and BI articipating countries. | |
| Rationale for change | 2.<br>be | Changed text to specify State done by AbbVie according | |
| Section To be changed | Se | ection 3.3.4.2 | |

Rationale for change

Trial Protocol 

Refer to rational for first change listed

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies Updated text to "AbbVie/Boehringer Ingelheim **Description of change** reserves the right to discontinue the trial overall or at a particular trial site at any time for the following reasons". Refer to rational for first change listed Rationale for change Section 5.5.2.2 Section To be changed Changed DNA banking sample storage from **Description of change** Boehringer Ingelheim to "AbbVie or a third party delegate (e.g. Boehringer Ingelheim Pharma GmbH & Co. KG; Birkendorfer Str. 65, 88397 Biberach, Germany)". Refer to rational for first change listed Rationale for change Section 7.3.4 **Section To be changed** Changed text to specify that AbbVie summary tables **Description of change** and listings will be produced and analyses based on AbbVie standards.